#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title : | Reporting and Analysis Plan for A Phase III,<br>randomised, multicenter, parallel-group, non-inferiority<br>study evaluating the efficacy, safety, and tolerability of<br>switching to dolutegravir plus lamivudine in HIV 1<br>infected adults who are virologically suppressed |
|---|---|
| Compound Number | GSK1349572 + GR109714 (GSK3515864) |
| Effective Date | 25 May 2022 |

# Description:

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Reports for Protocol 204862.
- This RAP will be provided to the study team members to convey the content of the 204862 Statistical Analysis Complete (SAC) deliverables for the reporting effort up to Week 200, including any post-Week 200 follow-up visits for participants with on-going AE or clinically significant laboratory abnormality at Week 200 (Final End of Study (EOS) Analysis).
- This version of the RAP is amendment to previous amendment 3 RAP (Week 144) dated 04-May-2021.

#### RAP Author(s):

| | Date |
|----------------------------------|-------------|
| Lead PPD | 17-May-2022 |
| Lead Statistician, Biostatistics | |

Copyright 2022 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# RAP Team Approvals (Method: E-mail):

| Approver | Date |
|---|---|
| PPD | 18-May-2022 |
| , ViiV Healthcare | |
| PPD | 19-May-2022 |
| Medicines Development Lead, Research and Development/Global<br>Medical Strategy Team | |
| PPD | 19-May-2022 |
| Principal Clinical Data Manager, Infectious Disease, Clinical Data<br>Management | |
| PPD | 19-May-2022 |
| Study Delivery Lead, R&D GCSD | |
| PPD | 18-May-2022 |
| , Safety and Medical Governance | |
| PPD | 18-May-2022 |
| Clinical Development Lead, ViiV Healthcare | |
| PPD | 19-May-2022 |
| Clinical Development Manager, ViiV Healthcare | |

# Clinical Statistics and Clinical Programming Line Approvals (Method: Pharma TMF eSignature):

| Approver | Approval Method |
|---------------------------------------|-----------------|
| Principal Statistician, Biostatistics | e-Signature |
| PPD , Clinical Programming | e-Signature |

The main changes included in RAP Amendment are as follows (and pertain to analyses relevant to Week 196/200):

The following displays have been added:

#### **Study Population**

- Summary of Subject Disposition for the Subject Conclusion Record DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase)
  (Table 1.101)
- 2. Summary of Reasons for Withdrawal by Visit DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 1.601)
- 3. Summary of Important Protocol Deviations DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 1.701)
- 4. Summary of Demographic Characteristics TBR arm Late Switch Phase (Table 1.1102)
- 5. Summary of Race and Racial Combinations Details TBR arm Late Switch Phase (Table 1.1402)
- 6. Summary of Hepatitis Status at Entry TBR arm Late Switch Phase (Table 1.1502)
- 7. Summary of CDC Classification of HIV Infection at Baseline TBR arm Late Switch Phase (Table 1.1602)
- 8. Summary of HIV Risk Factors TBR arm Late Switch Phase (Table 1.1702)
- 9. Summary of Screening Cardiovascular Risk Assessments TBR arm Late Switch Phase (Table 1.1802)
- 10. Summary of Distribution of CD4+ Cell Count (cells/mm^3) Results at LS Baseline TBR arm Late Switch Phase (Table 1.1902)
- 11. Summary of Current Medical Conditions DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 1.2001)
- 12. Summary of Past Medical Conditions TBR arm Late Switch Phase (Table 1.2101)
- 13. Summary of Concomitant Medications by Ingredient ATC Level 1 DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 1.2201)
- 14. Summary of Concomitant Medication Ingredient Combinations DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 1.2301)
- 15. Summary of Concomitant Medications by Combination Term ATC Level 1 DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 1.2401)
- 16. Summary of Antiretroviral Therapy Received at Screening TBR arm Late Switch Phase (Table 1.2602)
- 17. Summary of Current Cardiac, Gastrointestinal, Metabolism and Nutrition, Psychiatric, Renal and Urinary, and Nervous System Conditions DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 1.2701)
- 18. Summary of Past Cardiac, Gastrointestinal, Metabolism and Nutrition, Psychiatric, Renal and Urinary, and Nervous System Conditions DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 1.2801)

- 19. Summary of Lipid Modifying Agent Use at LS Baseline TBR arm Late Switch Phase (Table 1.2902)
- 20. Summary of Lipid Modifying Agent Use Starting Post-Baseline DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 1.3001)
- 21. Summary of History of Depression and Anxiety at LS Baseline TBR arm Late Switch Phase (Table 1.3102)
- 22. Summary of Baseline Third Agent Class TBR arm Late Switch Phase (Table 1.3202)
- 23. Summary of Number of Subjects Enrolled by Country and Site ID TBR arm Late Switch Phase (Table 1.3302)
- 24. Summary of Antiretroviral Therapy at Screening by Regimen TBR arm Late Switch Phase (Table 1.3602)
- 25. Summary of Distribution of Quantitative Plasma HIV-1 RNA Results at LS Baseline TBR arm Late Switch Phase (Table 1.3702)
- 26. Summary of Time since First Antiretroviral Therapy until Day 1 TBR arm Late Switch Phase (Table 1.3802)
- 27. Summary of On-Treatment Antiretroviral Therapy Starting after Day 1 for DTG + 3TC arm (Early and Late Switch Phase) and Starting after switch for TBR arm (Late Switch Phase) (Table 1.4001)
- 28. Summary of Antiretroviral Therapy Starting after Treatment Discontinuation DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 1.4101)
- 29. Summary of On-Treatment Antiretroviral after Day 1 for DTG + 3TC arm (Early and Late Switch Phase) and after switch for TBR arm (Late Switch Phase) by Regimen (Table 1.4201)
- 30. Summary of Antiretroviral Therapy Starting after Treatment Discontinuation by Regimen DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 1.4301)
- 31. Summary of Important COVID-19 Protocol Deviations DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 1.4401)
- 32. Summary of COVID-19 Pandemic Visit Impacts DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 1.4601)

#### Efficacy

- 33. Summary of Study Outcomes (Plasma HIV-1 RNA <sup>3</sup> / < 50 c/mL) at Week X Snapshot Analysis DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 2.401)
- 34. Summary of Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL by Visit Snapshot Analysis DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 2.1201)
- 35. Summary of Change from Baseline in CD4+ count (cells/mm3) by Visit DTG + 3TC arm DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 2.1701)
- 36. Summary of Change from Baseline in in CD4+/CD8+ count ratio (cells/mm3) by Visit DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 2.1801)

- 37. Summary of Post-Baseline HIV-1 Associated Conditions Including and Excluding Recurrences DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 2.1901)
- 38. Summary of Post-Baseline HIV-1 Disease Progressions DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 2.2101)
- 39. Cumulative Proportion of Subjects Meeting Confirmed Virologic Withdrawal Criteria by Visit DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 2.2201)
- 40. Summary of Study Outcomes (<40 c/mL and Target Not Detected Status) at Week X Snapshot DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 2.3101)
- 41. Summary of Study Outcomes (<40 c/mL) at Week X Snapshot Analysis DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 2.3501)
- 42. Individual Plasma HIV-1 RNA and CD4+ Profiles by Visit for subjects with at least one viral load ≥50 c/Ml DTG + 3TC arm Early and Late Switch Phase (Figure 2.401)
- 43. Individual Plasma HIV-1 RNA and CD4+ Profiles by Visit for subjects with at least one viral load ≥50 c/Ml TBR arm Late Switch Phase (Figure 2.402)

#### Safety

- 44. Summary of All Adverse Events by System Organ Class and Preferred Term and by Maximum Grade DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.601)
- 45. Summary of Common (>=2%) Adverse Events by Overall Frequency DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.701)
- 46. Summary of Common (>=2%) Grade 2-5 Adverse Events by Overall Frequency DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.801)
- 47. Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Grade DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.1001)
- 48. Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Grade TBR Late Switch Phase (Table 3.1002)
- 49. Summary of Common (>=2%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subject and Occurrences) DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.1101)
- 50. Summary of Common (>=0.5%) Drug-Related Grade 2-5 Adverse Events by Overall Frequency DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.1201)
- 51. Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.1401)

- 52. Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by Maximum Grade DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.1601)
- 53. Summary of Serious Adverse Events by System Organ Class DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.1801)
- 54. Summary of Drug-Related Serious Adverse Events by System Organ Class DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.2001)
- 55. Summary of Chemistry Changes from Baseline by Visit DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.2201)
- 56. Summary of Maximum Post-Baseline Emergent Chemistry Toxicities DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.2301)
- 57. Summary of Fasting Lipids Percentage Changes from Baseline by Visit DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.2601)
- 58. Summary of Changes in NCEP Lipid Baseline Category to Week X Category DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.3001)
- 59. Summary of Changes in Total Cholesterol /HDL Ratio Baseline Category to Week 196 DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.3201)
- 60. Summary of Hematology Changes from Baseline DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.3401)
- 61. Summary of Maximum Post-Baseline Emergent Hematology Toxicities DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.3501)
- 62. Summary of Change from Baseline in Bone Biomarkers by Visit DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.3701)
- 63. Summary of Change from Baseline in Renal Biomarkers by Visit DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.3801)
- 64. Summary of Change from Baseline in Renal Biomarkers by Visit Loge Transformed Data DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.3901)
- 65. Summary of Liver Monitoring/Stopping Event Reporting DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.4501)
- 66. Summary of Subjects Meeting Hepatobiliary Abnormality Criteria All Post-Baseline Abnormalities DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.4601)
- 67. Summary of True Positive Suicidal Indication Alerts Based on eCSSRS by Visit DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.4701)
- 68. Summary of Subjects with Post Baseline C-SSRS Suicidal Ideation or Behaviour DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.4901)

- 69. Summary of Characteristics of Post Baseline Anxiety Adverse Events of Special Interest DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.5001)
- 70. Summary of Characteristics of Post Baseline Depression Adverse Events of Special Interest DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.5101)
- 71. Summary of Characteristics of Post Baseline Suicidality and Self Injury Adverse Events of Special Interest DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.5201)
- 72. Summary of Characteristics of Post Baseline Insomnia Adverse Events of Special Interest DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.5301)
- 73. Summary of Characteristics of Post Baseline Rash Adverse Events of Special Interest DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.5401)
- 74. Summary of Characteristics of Post Baseline Nightmare/Abnormal Dreams Adverse Events of Special Interest DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.5501)
- 75. Summary of Characteristics of Post Baseline Drug Hypersensitivity Adverse Events of Special Interest DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.5601)
- 76. Summary of Onset and Duration of the First Occurrence of Post Baseline Anxiety Adverse Events of Special Interest DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.5701)
- 77. Summary of Onset and Duration of the First Occurrence of Post Baseline Depression Adverse Events of Special Interest DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.5801)
- 78. Summary of Onset and Duration of the First Occurrence of Post Baseline Suicidality and Self Injury Adverse Events of Special Interest DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.5901)
- 79. Summary of Onset and Duration of the First Occurrence of Post Baseline Insomnia Adverse Events of Special Interest DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.6001)
- 80. Summary of Onset and Duration of the First Occurrence of Post Baseline Rash Adverse Events of Special Interest DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.6101)
- 81. Summary of Onset and Duration of the First Occurrence of Post Baseline Nightmare/Abnormal Dreams Adverse Events of Special Interest DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.6201)
- 82. Summary of Onset and Duration of the First Occurrence of Post Baseline Drug Hypersensitivity Adverse Events of Special Interest DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.6301)
- 83. Summary of Post Baseline Depression and Suicidal and Self-Injury Adverse Events by AE of Special Interest, Maximum DAIDS Toxicity Grade, and Prior History of Depression and Anxiety DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.7101)

- 84. Summary of Change from Baseline in Weight (kg) by Visit DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.7501)
- 85. Summary of Change from Baseline in BMI (kg/m2) by Visit DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.7601)
- 86. Summary of HOMA-IR Shifts from Baseline to Week X DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.8101)
- 87. Summary of Change from Baseline in Inflammatory Biomarkers Loge Transformed Data - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.9601)
- 88. Summary of Proportion of Subjects with Change from Baseline in Weight (>=3%, >=5% and >=10%) at Week X DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.9801)
- 89. Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term up to the End of the Week 196 Reporting Window (USPI) DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.9901)
- 90. Summary of Common (>=0.5%) Drug-Related Grade 2-5 Adverse Events by Overall Frequency up to the End of the Week X Reporting Window (USPI) DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.10001)
- 91. Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term /by Overall Frequency up to the End of the Week X Reporting Window (USPI) DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.10101)
- 92. Summary of Characteristics of Post Baseline Increase in Weight Adverse Events of Special Interest DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.10401)
- 93. Summary of Characteristics of Post Baseline Decrease in Weight Adverse Events of Special Interest DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.10501)
- 94. Summary of Maximum Post-Baseline Emergent Clinical Chemistry Toxicities to the End of the Week X Reporting Window (USPI) LOCF DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.10801)
- 95. Summary of Maximum Post-Baseline Emergent Hematology Toxicities to the End of the Week X Reporting Window (USPI) DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.11001)
- 96. Summary of COVID-19 Assessments DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.11101)
- 97. Summary of Waist to Height Ratio and Waist to Hip Ratio by Visit DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.11801)
- 98. Summary of Change from LS Baseline in Waist to Height Ratio and Waist to Hip Ratio at Week 196 TBR arm Late Switch Phase (Table 3.11803)
- 99. Proportion of Subjects with Metabolic Syndrome at Week 196 DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.11901)

- Summary of Change from Baseline in Framingham Risk Score at Week
   196 DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.12001)
- 101. Summary of Change from Baseline in Systolic Blood Pressure and Diastolic Blood Pressure at week 196 DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 3.12101)
- 102. Scatter Plot of Maximum ALT vs. Maximum Total Bilirubin DTG + 3TC arm Early and Late Switch Phase (Figure 3.301)
- 103. Scatter Plot of Maximum ALT vs. Maximum Total Bilirubin TBR arm Late Switch Phase (Figure 3.302)
- 104. Heatmap plot of Triglycerides, LDL Cholesterol, Total Cholesterol (mmol/L) NCEP Categories and Total Cholesterol/HDL Ratio at Week X vs. Baseline DTG + 3TC arm Early and Late Switch Phase (Figure 3.401)
- 105. Heatmap plot of Triglycerides, LDL Cholesterol, Total Cholesterol (mmol/L) NCEP Categories and Total Cholesterol/HDL Ratio at Week X vs. LS Baseline TBR arm Late Switch Phase (Figure 3.402)
- 106. Heatmap plot of BMI at Week X vs. Baseline DTG + 3TC arm Early and Late Switch Phase (Figure 3.2501)
- 107. Heatmap plot of BMI at Week X vs. LS Baseline TBR arm Late Switch Phase (Figure 3.2502)

#### Virology

- 108. Summary of INSTI Mutations and Major Mutations of NRTI, NNRTI and PI Classes by region at Baseline and Time of CVW at or prior to Week X DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 4.101)
- 109. Summary of Phenotype at Baseline and Time of CVW by Phenotypic Cutoff at or prior to Week X - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 4.401)
- 110. Summary of Phenotype at time of CVW by Number of Drugs to Which Subject are Resistant at or prior to Week X DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 4.501)
- 111. Summary of Fold Change to DTG, 3TC, TDF and FTC at Time of CVW at or prior to Week X DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 4.601)
- 112. Summary of Subject Accountability: Genotypes Available at or prior to Week X DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 4.701)
- 113. Summary of Subject Accountability: Phenotypes Available at or prior to Week X DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 4.801)

#### **Health Outcomes**

114. Summary of EQ-5D Utility and Thermometer Scores by visit – DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) (Table 6.201)

There are numerous displays that have been removed but these are not listed for reasons of brevity.

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| TAI | ABLE OF CONTENTS | | 10 |
| 1. | INTRODUCTION | | 13 |
| 2. | <ul><li>2.1. Changes to the Protocol I</li><li>2.2. Study Objective(s) and Er</li><li>2.3. Study Design</li></ul> | L INFORMATION Defined Statistical Analysis Plan ndpoint(s) Statistical Analyses | 13<br>13 |
| 3. | 3.1. Interim Analyses | | 19 |
| 4. | | | _ |
| 5. | CONVENTIONS | ANALYSES AND DATA HANDLING roup Display Descriptors e Switch Phase s, Other Strata and Subgroups Other Strata Subgroups d Multiplicity Data Analyses and Data Handling | 25<br>25<br>26<br>26<br>26<br>27 |
| 6. | | ESdy Population Analyses | |
| 7. | 7.1. Primary Efficacy Analysis 7.1.1. Summary Meas 7.1.2. Population of Intelligence 7.1.3. Strategy for Intelligence | ureterestrcurrent (Post-Randomisation) Events | 32<br>32<br>32 |
| | 7.2. Secondary Efficacy Analy 7.2.1. Endpoint / Varia 7.2.2. Summary Meas 7.2.3. Populations of Ir 7.2.4. Strategy for Inte 7.2.5. Statistical Analy | vses | 36<br>36<br>36<br>36 |
| 8 | ı , | bles | |

### **CONFIDENTIAL**

| | 8.1. | Adverse | Events Analyses | 42 |
|---|---|---|---|---|
| | 8.2. | | Events of Special Interest Analyses | |
| | 8.3. | Clinical I | Laboratory Analyses | 44 |
| | 8.4. | Other Sa | afety Analyses | 52 |
| 9. | OTHE | R STATIS | STICAL ANALYSES | 55 |
| Ο. | 9.1. | | Outcomes. | |
| | 0.1. | 9.1.1. | Overview of Planned Analyses | |
| | | 9.1.2. | Planned Health Outcomes Statistical Analysis | |
| | 9.2. | - | | 56 |
| | • | 9.2.1. | | 56 |
| | | 9.2.2. | | |
| 10 | PHARI | MACOKIN | NETIC ANALYSES | 58 |
| | | | cokinetic Analyses | |
| | 10.1. | 10.1.1. | Endpoint / Variables | |
| | | 10.1.2. | Summary Measure | |
| | | 10.1.3. | Population of Interest | |
| | | 10.1.4. | | |
| | | 10.1.5. | | |
| 11. | POPU | LATION F | PHARMACOKINETIC (POPPK) ANALYSES | 60 |
| 12 | REFE | RENCES | | 61 |
| 13. | | | | 62 |
| | 13.1. | | x 1: Protocol Deviation Management and Definitions for Per<br>Population | 63 |
| | | | Exclusions from Per Protocol Population | |
| | 13.2. | Appendi | x 2: Protocol Defined Schedule of Activities | 65 |
| | | 13.2.1. | Week 148) | 65 |
| | | 13.2.2. | Late Switch Phase Time and Events Table: TBR subjects | |
| | | | who switched to DTG + 3TC at Week 148 | 69 |
| | | 13.2.3. | Late Switch Phase Time and Events Table: DTG + 3TC | |
| | | | arm | |
| | 13.3. | | x 3: Assessment Windows | |
| | | 13.3.1. | Definitions of Assessment Windows for Analyses | 74 |
| | | 13.3.2. | | |
| | 40.4 | | Analysis | |
| | 13.4. | | x 4: Study Phases and Emergent Adverse Events | |
| | | 13.4.1. | | /8 |
| | | 13.4.2. | <b>.</b> | |
| | 40.5 | | Emergent Flag for Adverse Events | |
| | 13.5. | Appendi | x 5: Data Display Standards & Handling Conventions | 84 |
| | | 13.5.1. | Reporting Process. | |
| | | 13.5.2. | Reporting Standards for Pharmacking tip | |
| | 13.6. | 13.5.3. | Reporting Standards for Pharmacokineticx 6: Derived and Transformed Data | |
| | 13.0. | 13.6.1. | | |
| | | 13.6.1. | | |
| | | | Efficacy | |

#### **CONFIDENTIAL**

| | 13.6.4. | Safety | |
|---|---|---|---|
| | 13.6.5. | Pharmacokinetic | |
| | 13.6.6. | Population Pharmacokinetic (PopPK) | 100 |
| | 13.6.7. | Not applicable to analyses post Week 48. Viral Genotyping | |
| | | and Phenotyping | |
| | 13.6.8. | Health Outcomes | |
| | 13.6.9. | | |
| | 13.6.10. | PK DataeCRF Baseline Third Agent Class Determination | 107 |
| 13.7. | | | |
| 13.7. | | x 7: Reporting Standards for Missing Data<br>Premature Withdrawals | |
| | | Handling of Missing Data | |
| 13.8. | | x 8: Values of Potential Clinical Importance | |
| 13.9. | | x 9: Population Pharmacokinetic (PopPK) Analyses | |
| | Appendi | x 10: Time to Event Details | 113 |
| | | TRDF Detailed Steps | |
| | | TRDF Detailed Steps for the Kaplan-Meier plot | |
| | | ERDF Detailed Steps | |
| 13.11. | | x 11: Snapshot | |
| 13.12. | Appendi | x 12: Abbreviations & Trade Marks | 123 |
| | | Abbreviations | |
| | | Trademarks | 124 |
| 13.13. | | x 13: Model Checking and Diagnostics for Statistical | |
| | Analyses | S | 125 |
| 40.44 | | Statistical Analysis Assumptions | 125 |
| 13.14. | | x 14: COVID-19 Modified Analyses and Supportive | 400 |
| | | ty Analyses | |
| 10 15 | | Efficacy Analyses (Snapshot) | |
| 13.15. | | x 15: List of Data Displays | |
| | 13.15.1. | Data Display Numbering Mock Example Shell Referencing | 130 |
| | | Deliverables | |
| | | Study Population Tables | |
| | | Efficacy Tables. | |
| | | Efficacy Figures | |
| | 13.15.7. | Safety Tables | 149 |
| | | Safety Figures | |
| | 13.15.9. | Virology tables | 176 |
| | | ).Pharmacokinetic Tables | |
| | 13.15.11 | I.Pharmacokinetic Figures | 180 |
| | 13.15.12 | 2.Health Outcomes Tables | 181 |
| | 13.15.13 | B.Health Outcomes Figures | 182 |
| | | I.ICH Listings | |
| | | 5.Non-ICH Listings | |
| 13.16. | Appendi | x 16: Example Mock Shells for Data Displays | 195 |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There are no changes or deviations to the originally planned statistical analysis specified in the protocol amendment 7 (Dated: 27-APR-2020).

# 2.2. Study Objective(s) and Endpoint(s)

| Objective | Endpoint |
|---|---|
| | mary |
| To demonstrate the non-inferior antiviral activity of switching to DTG+3TC once daily compared to continuation of Tenofovir alafenamide (TAF) based regimen (TBR) over 48 weeks in HIV-1 infected, ART therapy (ART)-experienced, virologically suppressed subjects | Virologic failure (subjects with plasma HIV-1 RNA ≥50 copies c/mL) endpointas per FDA snapshot category at Week 48 |
| | ndary |
| To demonstrate the antiviral activity of switching to DTG + 3TC once daily compared to continuation of TBR over 48 weeks | Proportion of subjects with plasma HIV-1 RNA <50 copies c/mL at Week 48 using the Snapshot algorithm for the ITT-E population |
| To demonstrate the antiviral activity of switching to DTG + 3TC once daily compared to continuation of TBR over 24, 96 and 144 weeks | <ul> <li>Subjects with plasma HIV 1 RNA ≥50 copies c/mL endpoint as per FDA snapshot category at Weeks 24, 96 and 144</li> <li>Proportion of subjects with plasma HIV-1 RNA &lt;50 c/mL at Weeks 24, 96 and 144 using the Snapshot algorithm for the ITT-E population</li> </ul> |
| To evaluate the immune effects of DTG + 3TC once daily compared to continuation of TBR over 24, 48, 96 and 144 weeks | <ul> <li>Change from Baseline in CD4+ cell count and in CD4+/CD8+ cell count ratio at Weeks 24, 48, 96 and 144</li> <li>Incidence of disease progression (HIV-associated conditions, AIDS, and death) through Weeks 24, 48, 96 and 144</li> </ul> |

| Objective | Endpoint |
|---|---|
| To evaluate the safety and tolerability of DTG + 3TC once daily compared to TBR over time | <ul> <li>Incidence and severity of AEs and laboratory abnormalities through 144 weeks</li> <li>Proportion of subjects who discontinue treatment due to AEs through 144 weeks</li> </ul> |
| To evaluate the effects of DTG + 3TC once daily on fasting lipids over time compared to TBR | Change from Baseline in fasting lipids at Weeks 24,48, 96 and 144 |
| To assess viral resistance in subjects meeting Virologic Withdrawal Criteria | Incidence of observed genotypic and phenotypic resistance to ARVs for subjects meeting Virologic Withdrawal Criteria |
| To evaluate renal (in urine and blood) and bone (in blood) biomarkers in subjects treated with DTG + 3TC compared to TBR | Change from Baseline in renal and bone biomarkers at Weeks 24,48, 96 and 144 |
| To assess health related quality of life for subjects treated with DTG + 3TC compared to TBR | Change from Baseline in health status using EQ-5D-5L at Weeks 24, 48, 96 and 144 (or Withdrawal from the study) |
| Explo | pratory |
| To evaluate the effect of patient characteristics (e.g., demographic factors, Baseline CD4) on antiviral and immunological responses to DTG + 3TC compared to TBR | <ul> <li>Proportion of subjects by subgroup(s) (e.g., by age, gender, Baseline CD4) with plasma HIV-1 RNA &lt;50c/mL using the Snapshot algorithm at Weeks 24, 48, 96 and 144</li> <li>Change from Baseline in CD4+ cell counts at Weeks 24, 48, 96 and 144 by patient subgroups</li> </ul> |
| To assess willingness to switch for subjects treated with DTG + 3TC compared to TBR | Reasons for Willingness to Switch at Day 1 |
| To evaluate biomarkers of telomerase function in a subset of subjects treated with DTG + 3TC compared to TBR. | Change from baseline in biomarkers of telomerase function at Weeks 48, 96 and 144 |
| To evaluate inflammation biomarkers and insulin resistance in a subset of subjects treated with DTG+3TC compared to TBR | Change from Baseline in inflammation biomarkers and homeostasis model of assessment-insulin resistance (HOMA-IR) at Weeks 48, 96 and 144 |
| To describe body morphologyat Week 144 in subjects treated with DTG + 3TC and TBR | <ul> <li>Waist to height ratio at Week 144 in each arm</li> <li>Waist to hip ratio at Week 144 in each arm</li> </ul> |
| To assess metabolic health and Cardiovascular disease risk at Week 144 in | Proportions of subjects with Metabolic<br>Syndrome at Week 144 in each arm |
| subjects treated with DTG+3TC and TBR | Change from Baseline in Framingham risk<br>Score through Week 144 in each arm |

| Objective | Endpoint |
|---|---|
| | Change from Baseline in resting Blood<br>Pressure at Week 144 in each arm |
| To evaluate the longer term antiviral and immunological effects, safety and tolerability of DTC + 3TC area daily in subjects treated | For subjects in the DTG + 3TC arm since Early Switch Phase: |
| of DTG + 3TC once daily in subjects treated with DTG + 3TC since the Early Switch Phase | <ul> <li>Proportion of subjects with plasma HIV-1 RNA &lt;50 c/mL at Week 196 using the Snapshot algorithm for the ITT-E population</li> <li>Change from Baseline in CD4+ lymphocyte count and in CD4+/CD8+ cell count ratio at Week 196</li> <li>Incidence and severity of AEs and laboratory abnormalities over 196 weeks</li> <li>Proportion of subjects who discontinue treatment due to AEs over 196 weeks</li> <li>Incidence of disease progression (HIV associated conditions, AIDS and death) through Week 196</li> <li>Change from Baseline in renal and bone biomarkers at Week 196</li> <li>Change from baseline in biomarkers of inflammation, HOMA-IR and telomerase function at Week 196</li> </ul> |
| To describe body morphologyat Week 196 in subjects treated with DTG + 3TC since the Early Switch Phase | <ul><li>Waist to height ratio at Week 196</li><li>Waist to hip ratio at Week 196</li></ul> |
| To assess metabolic health and Cardiovascular disease risk at Week 196 in subjects treated with DTG + 3TC since the | Proportions of subjects with Metabolic<br>Syndrome at Week 196 |
| Early Switch Phase | Change from Baseline in Framingham risk |
| | Score through Week 196 |
| | Change from Baseline in resting Blood<br>Pressure at Week 196 |
| To evaluate the antiviral and immunological effects, safety and tolerability of DTG + 3TC | For subjects switching to DTG + 3TC in the Late Switch Phase: |
| for subjects switching in the Late Switch Phase | <ul> <li>Proportion of subjects with plasma HIV-1<br/>RNA &lt;50 c/mL at Week 196 using the<br/>Snapshot algorithm for the ITT-E<br/>population</li> <li>Change from Baseline in CD4+<br/>lymphocyte count and in CD4+/CD8+ cell<br/>count ratio at Week 196</li> </ul> |

| Objective | Endpoint |
|---|---|
| | <ul> <li>Incidence and severity of AEs and laboratory abnormalities during the Late Switch Phase</li> <li>Proportion of subjects who discontinue treatment due to AEs during the Late Switch Phase</li> <li>Incidence of disease progression (HIV associated conditions, AIDS and death) during the Late Switch Phase</li> <li>Change from Baseline in renal and bone biomarkers at Week 196</li> <li>Change from baseline in biomarkers of inflammation, HOMA-IR and telomerase function at Week 196</li> </ul> |
| To assess body morphologyat Week 196 in subjects switching to DTG + 3TC in the Late Switch Phase | <ul> <li>Change in waist to height ratio from Switch to Week 196</li> <li>Change in waist to hip ratio from Switch to Week 196</li> </ul> |
| To assess metabolic health and Cardiovascular disease risk at Week 196 in subjects treated with DTG + 3TC since the Late Switch Phase | <ul> <li>Proportions of subjects with and incidence of Metabolic Syndrome at Week 196</li> <li>Change from Baseline in Framingham risk Score through Week 196</li> <li>Change from Baseline in resting Blood Pressure at Week 196</li> </ul> |
| To assess the steady-state DTG and 3TC exposure in HIV-1 infected patients | Steady state plasma PK parameters of DTG and 3TC will be assessed using intensive PK collected at week 4 (not applicable to analyses post Week 48). |
| To characterize the DTG and 3TC steady-<br>state PK of the DTG/3TC FDC in HIV-1<br>infected patients | Population estimates of DTG and 3TCPK parameters (e.g. apparent clearance [CL/F], apparent volume of distribution [V/F]) using DTG and 3TC intensive and sparse plasma concentrations at Weeks, 4, 8, 12, 24, 36 and 48 (not applicable to analyses post Week 48). |

## 2.3. Study Design



See study protocol for further details

## 2.4. Statistical Hypotheses / Statistical Analyses

This study is designed to show that the antiviral effect of switching to a simplified two-drug regimen of DTG + 3TC once-daily is not inferior to continuation of their TBR at week 48 in HIV-1 infected ART-experienced subjects. Assuming a true 2% virologic failure rate in each arm, a non-inferiority margin of 4%, and a 2.5% one-sided significance level, this study requires 275 subjects per treatment arm. This would provide 92% power to show non-inferiority for the proportion of subjects with virologic failure according to the FDA snapshot algorithm at 48 weeks post-switch.

While the targeted study size was 550 randomised subjects (from a target of 800 screened subjects), the study was over-enrolled based on an unexpected surge in recruitment in the last week of screening ending with a final number of 743 subjects randomised. This will provide 97.3% power to show non-inferiority with the current assumptions, and non-inferiority can be declared if the actual observed treatment difference in the trial is less than or equal to 1.6%.

Non-inferiority can be concluded if the upper bound of a two-sided 95% confidence interval for the difference in virologic failure rates between the two treatment arms is smaller than 4%. If  $r_d$  is the virologic failure rate on DTG + 3TC and  $r_f$  is the virologic failure rate on the current ART regimen, then the hypotheses can be written as follows:

$$H_0: r_d - r_f \ge 4\%$$
  $H_1: r_d - r_f < 4\%$ 

#### 3. PLANNED ANALYSES

## 3.1. Interim Analyses

An interim analysis will be performed at Week 24. To minimise bias, the results of the Week 24 results will not be shared with subjects and investigators, or presented externally until after the last subject completes their Week 48 visit. Please refer to the Blinding Agreement for more details.

The planned analysis at Week 24 will be performed after the completion of the following sequential steps:

- Last subject has completed their visit at Week 24 as defined in the protocol, including any re-test if required.
- All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.
- All criteria for unblinding<sup>1</sup> the randomisation codes at Week 24 have been met.

No adjustment for multiplicity will be made as the Week 24 analyses will be secondary, however non-inferiority at Week 24 will be declared if the upper bound of a two-sided 95% confidence interval for the difference in virologic failure rates between the two treatment arms is less than 4%<sup>2</sup>.

An IDMC was instituted to ensure external objective medical and/or statistical review of efficacy and safety in order to protect the ethical interests and well-being of subjects and to protect the scientific validity of the study. An ad-hoc review of data by the IDMC will be triggered whenever the number of confirmed virologic withdrawals (CVWs) exceeds thresholds pre-specified in the IDMC charter. Full details of the methods, timing, decision criteria and operating characteristics are pre-specified in the IDMC Charter. Details of the analyses and outputs provided to the IDMC are detailed in an IDMC RAP.

# 3.2. Final Analyses

The primary analysis is at Week 48. Additional analyses will be performed at Weeks 96, 144 and 196 and at the end of the continuation phase, if applicable. Analyses performed after Week 48 are considered interim analyses beyond the primary analysis.

<sup>&</sup>lt;sup>1</sup> Although this is considered an open-label study, any data transfers/dry-runs prior to formal analyses will be based on blinded or dummy treatment allocation. Any references to unblinding the study in this analysis plan pertains to the process of unmasking the actual randomisation codes at formal data base locks.

<sup>&</sup>lt;sup>2</sup> Please refer to Section 7.1.4 for details and conditions for presentation of test for superiority.

The planned analyses at Weeks 48, 96, 144 and 196 and end of continuation phase (if applicable)<sup>3</sup> will be performed after the completion of the following sequential steps:

- Last subject has completed their relevant visit at week 48 (96, 144, 196 or end of continuation) as defined in the protocol (or surpassed the time point at which their visit was scheduled but not completed due to COVID-19 at time of Week 196 analysis), including any re-test if required
- All required database cleaning activities have been completed as specified in the monitoring plan and Data Validation Manual and final database release and database freeze has been declared by Data Management. Any impact of COVID-19 on data management activities will be documented in the DBF Memo.
- All criteria for unblinding the randomisation codes at Week 48 (96, 144, 196 or end of continuation) have been met.

Further data cuts and analyses may be conducted as necessary in order to support regulatory submissions and publications.

### 4. ANALYSIS POPULATIONS

| Population | Definition/Criteria | Analyses Evaluated |
|---|---|---|
| All subjects screened | <ul> <li>Comprises all subjects screened for inclusion in the study, including screen-failures.</li> <li>This population will be based on the treatment to which the subject was randomised. Screenfailures will be categorised as "Non-randomised".</li> </ul> | Study Population |
| Randomised | The Randomised population will consist of all subjects who are randomised in the study | Study Population |
| Intent-to-Treat<br>(ITT) | <ul> <li>Comprises all randomised subjects</li> <li>Subjects will be assessed according to the treatment to which the subject was randomised regardless of treatment actually received.</li> <li>Any subject receiving a treatment randomisation number will be considered to be randomised.</li> </ul> | Efficacy (sensitivity analyses) |
| Intent-To-Treat<br>Exposed (ITT-E) | <ul> <li>Comprises all randomised subjects who receive at least one dose of study treatment either DTG + 3TC or TBR.</li> <li>This population will be based on the treatment to which the subject was randomised.</li> </ul> | <ul> <li>Study Population,<br/>Efficacy and Health<br/>Outcomes</li> </ul> |

20

<sup>&</sup>lt;sup>3</sup> Note that analyses for time points will be performed when subjects complete visits relevant to that time point i.e. Week 48 analysis takes place when the last patient has completed their Week 48 visit, and not when they have completed their Week 48, Week 96, Week 144, Week 196 and end of continuation phase.

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| · | Any subject who receives a treatment randomisation number will be considered to have been randomised. | - |
| Late-Switch<br>Intent-to-Treat<br>(Exposed) (LS-<br>ITT-E) | <ul> <li>Comprised of all subjects randomised to TBR who receive at least one dose of study treatment at or after the Week 148 Switch visit.</li> <li>Subjects will be assessed according to the treatment intended regardless of treatment actually received (i.e., subjects not receiving TBR in the Early Switch Phase or failing to switch to DTG + 3TC at Week 148 will be included provided they progress to the Late Switch Phase).</li> <li>Any subject who receives a treatment randomisation number will be considered to have been randomised.</li> <li>Any subject receiving a treatment at or after Week 148 will be considered treated within the Late Switch Phase.</li> </ul> | |
| Per-Protocol (PP) | <ul> <li>This population will consist of subjects in the ITT-E Population with the exception of significant protocol violators.</li> <li>Protocol deviations that would exclude subjects from the PP population are defined in Section 4.1 (Protocol Deviations) and Section 13.1 (Protocol Deviation Management and Definition for Per-Protocol Population).</li> </ul> | Efficacy (Sensitivity<br>Analysis) (not<br>applicable to post<br>Week 144) |
| CVW | Comprises all subjects in the ITT-E population who have met the derived CVW criteria Note: For TBR arm, this only includes subjects who have met CVW criteria before the switch (both assessments in early switch phase). For DTG/3TC subjects, this includes subjects who have met CVW criteria in either early or late switch phases | <ul><li>Genotypic</li><li>Phenotypic</li><li>Efficacy</li></ul> |
| Late-Switch<br>CWW (LS-CWW) | Comprises all subjects in the LS-ITT-E population who have met the derived CWV criteria in the late switch phase | <ul><li>Genotypic</li><li>Phenotypic</li><li>Efficacy</li></ul> |
| potential<br>Precautionary<br>Virologic<br>Withdrawal<br>(pPVW) | Comprises subjects in the ITT-E population having 2 consecutive measurements between 50 and 200 c/mL Note: For TBR arm, this only includes subjects who have met pPWW criteria before the switch (both assessments in early switch phase). For DTG/3TC subjects, this includes subjects who have met pPWW criteria in either early or late switch phases | <ul><li>Genotypic</li><li>Phenotypic</li></ul> |

| Population | Definition/Criteria | Analyses Evaluated |
|---|---|---|
| Late-Switch potential Precautionary Virologic Withdrawal (LS-pPWW) | Comprises subjects in the LS-ITT-E population<br>having 2 consecutive measurements between<br>50 and 200 c/MI in late switch phase | Genotypic Phenotypic |
| Viral Genotypic | Comprises all subjects in the ITT-E population who have available on-treatment genotypic resistance data. Assessed according to the treatment they actually received Note: For TBR arm, this only includes subjects with available on-treatment genotypic resistance data based n a viral load assessed before the switch (early switch phase). For DTG/3TC subjects, this includes subjects with available on-treatment genotypic resistance data in either early or late switch phases | Genotypic |
| Late-Switch Viral<br>Genotypic | Comprises all subjects in the LS-ITT-E population who have available on-treatment genotypic resistance data based on a viral load assessed in the late switch phase. Assessed according to the treatment they actually received | Genotypic |
| Viral Phenotypic | Comprises all subjects in the ITT-E population who have available on-treatment phenotypic resistance data. Assessed according the treatment they actually received Note: For TBR arm, this only includes subjects with available on-treatment phenotypic resistance data based on a viral load assessed before the switch (early switch phase). For DTG/3TC subjects, this includes subjects with available on-treatment phenotypic resistance data in either early or late switch phases | Phenotypic |
| Late-Switch Viral<br>Phenotypic | Comprises all subjects in the LS-ITT-E population who have available on-treatment phenotypic resistance data based on a viral load assessed in the late switch phase. Assessed according the treatment they actually received | Phenotypic |
| Efficacy<br>Evaluable | Comprises all subjects who did not have missing Week 96 (and repeated at Week 144) HIV-1 RNA visit data as a result of the COVID-19 pandemic i.e. discontinuation due to COVID-19 or on-study but missed visit due to | Efficacy |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| | COVID-19 (see Section 13.14.1 for further details) | |
| Safety | <ul> <li>Comprises all subjects who receive at least one dose of study treatment either DTG + 3TC or TBR.</li> <li>This population will be based on the treatment the subject actually received<sup>4</sup>.</li> </ul> | Safety |
| Late-Switch<br>Safety (LS-<br>Safety) | Comprised of all subjects randomised to TBR who received at least one dose of DTG+3TC at or after the Week 148 Switch visit. | Safety Late-Switch Phase |
| Sparse<br>Pharmacokinetic<br>Population | All subjects who received at least 1 dose of DTG/3TCFDC and have evaluable sparse samples with drug concentrations reported, where samples are collected according to the sparse sampling schedule (through Week 48). | PK (not applicable to<br>analyses post Week<br>48) |
| Intensive Pharmacokinetic Concentration Population | The subset of subjects enrolled into intensive<br>PK sampling, who received at least 1 dose of<br>DTG/3TCFDC and have evaluable drug<br>concentrations reported, where samples are<br>collected according to the intensive sampling<br>schedule (Week 4 only). | PK (not applicable to<br>analyses post Week<br>48) |
| Intensive Pharmacokinetic Parameter Population | All subjects in the Intensive Pharmacokinetic<br>Concentration Population who provide at least<br>one evaluable PK parameter. | PK (not applicable to<br>analyses post Week<br>48) |

### NOTES:

# 4.1. Protocol Deviations

| Term | Definition |
|---|---|
| Study Deviation<br>Rules Document | The document describing study deviations (and associated coding/naming conventions) that may be identified during a study and the frequency of study deviation reviews. |
| Protocol Deviation (PD) | Any departure from study-specific requirements specified in a protocol. Subsets of protocol deviations are categorized as important or significant. |

\_

<sup>1.</sup> Please refer to Appendix 15: List of Data Displays which details the population to be used for each display being generated.

<sup>&</sup>lt;sup>4</sup> As recorded on IVRS. If the randomised treatment is incorrect, the actual treatment will only be recorded in IVRS through sponsor intervention.

| Term | Definition |
|---|---|
| Important Protocol<br>Deviations | A subset of protocol deviations that may significantly impact the completeness, accuracy, and/or reliability of the study data or that may significantly affect a subject's rights, safety, or well-being. All important deviations have a Violation Flag in CTMS and are associated with a Rule Number. |
| Significant<br>Protocol<br>Deviations | Considered a subset of important protocol deviations, typically impacting efficacy assessments, which lead to the exclusion from the per-protocol population. All significant deviations are captured in CTMS and are associated with a Rule Number. |
| COVID-19<br>Protocol<br>Deviations | Important protocol deviations relating to the COVID-19 pandemic will be documented in CTMS with their respective rule number followed by 'COVID-19' before text description. All other COVID-19 related protocol deviations not associated with a rule number will be documented with 'COVID-19' before the text description. |

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Important deviations which result in exclusion from the analysis population (Significant deviations) will also be summarised and listed (see Section 13.1).

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- Data will be reviewed prior to unblinding and freezing of the database with the aim of capturing and categorising all important deviations and deviations which may lead to exclusion from the analysis in the protocol deviations SDTM dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Subgroup Display Descriptors

| Treatment Group Description | Order <sup>[1]</sup> |
|-----------------------------|----------------------|
| DTG+3TC | 1 |
| TBR | 2 |
| Late Switch Phase | |
| ES DTG+3TC | 1 |
| LS DTG+3TC | 2 |

#### NOTES:

1. Order represents treatments being presented in TFL, as appropriate.

ES DTG+3TC - Early Switch DTG+3TC

LS DTG+3TC – Late Switch DTG+3TC

Treatment comparisons will be displayed as follows using the descriptors as specified:

1. DTG + 3TC vs TBR

#### 5.2. Baseline Definitions

For all endpoints/parameters (unless otherwise stated) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

Unless otherwise stated, if baseline data are missing no derivation will be performed and baseline will be set to missing.

Unless otherwise specified, the baseline definitions specified in the table below will be used for derivations for endpoints/parameters and indicated on summaries and listings.

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit Value – Baseline |
| % Change from Baseline | = 100 x [(Post-Dose Visit Value – Baseline) / Baseline] |

#### 5.2.1. Baseline for Late Switch Phase

For the Late Switch Phase for TBR subjects, the last pre-switch data will be used to represent 'baseline' for DTG+3TC assessment. In most cases, this will be Week 144 data and summaries will be labelled accordingly (e.g., 'LS Baseline'). In particular, for disease progressions, this will involve assessing the disease progression observed during the Early Switch Phase (up to Week 144) and using any known progressed status as 'baseline' for assessing disease progression in the Late Switch Phase of the study.

### 5.3. Multicentre Studies

Data will be summarised for all centres combined. Country will be treated as an exploratory subgroup for analyses of the primary efficacy endpoint.

# 5.4. Examination of Covariates, Other Strata and Subgroups

### 5.4.1. Covariates and Other Strata

- The following is a list of covariates that may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses
- Additional covariates of clinical interest may also be considered.

| Category | Details |
|---|---|
| Randomisation Strata | Randomisation is stratified by baseline third agent class: |
| | Baseline third agent class (PI, NNRTI, INI). |
| | For analysis purposes, randomisation strata will be derived using eCRF data, even if this differs from the strata captured in IVRS (details of how this is derived can be found in Section 13.6.11) |
| | All statistical analyses will adjust for the above randomisation |
| | strata, unless stated otherwise. Treatment-by-Strata interactions will be assessed as specified in the analysis |
| | sections. |
| Covariates | • Age (years): <35, 35 to <50, ≥50 (or continuous) |
| | Gender: Male & Female |
| | Baseline CD4+ cell count: |
| | <200, 200 to <350, ≥350 cells/mm³ (or continuous) |
| | Race (White, Black or African American, Asian, Other), or (White, Non-White) |
| | <ul> <li>BMI (<vs. (or="" 25="" continuous)<="" kg="" li="" m²)="" ≥=""> </vs.></li></ul> |
| | <ul> <li>Smoking status (Never vs. Former vs. Current Smoker),</li> </ul> |
| | Vitamin D use (Yes vs. No) |
| | Diabetes mellitus (Yes vs. No) |
| | Hypertension (Yes vs. No) |
| | HCV-coinfection (Yes vs. No) |
| | Prior TAF duration: (continuous) |
| | Region |
| | North America (USA, Canada) |
| | <ul> <li>Europe (Belgium, France, Germany, Netherlands,<br/>Spain, UK)</li> </ul> |
| | <ul> <li>Asia/Australia (Japan, Australia)</li> </ul> |

# 5.4.2. Examination of Subgroups

The list of subgroups may be used in descriptive summaries and statistical analyses. Additional subgroups of clinical interest may also be considered. No subgroup analysis planned for W196/W200.

• If the percentage of subjects is small within a particular subgroup, then the subgroup categories may be refined prior to unblinding the trial.

If the category cannot be refined further, then descriptive rather than statistical comparisons may be performed for the particular subgroup.

| Subgroup | Subgroups |
|---|---|
| Randomisation Strata | Randomisation is stratified by baseline third agent class: |
| | Baseline third agent class (PI, NNRTI, INI). |
| | For analysis purposes, randomisation strata will be derived using eCRF data, even if this differs from the strata captured in IVRS |
| | All statistical analyses will adjust for the above randomisation strata, unless stated otherwise. Treatment-by-Strata interactions will be assessed as specified in the analysis sections. |
| Demographic and Baseline<br>Characteristics | <ul> <li>Age (years): &lt;35, 35 to &lt;50, ≥50, and &lt;50 vs. &gt;=50</li> <li>An additional split of Age &lt;50 and ≥60, or &lt;60 and ≥60 may also be performed if specifically required for regulatory purposes)</li> <li>Gender: Male &amp; Female</li> <li>Baseline CD4+ cell count: <ul> <li>&lt;200, 200 to &lt;350, ≥350 cells/mm³</li> <li>&lt;500, ≥500 cells/mm³</li> <li>&lt;350, ≥350 cells/mm³</li> </ul> </li> <li>CDC HIV-1 classification</li> <li>Country</li> <li>Race: White, Black or African American, Asian, Other; and: White vs non-White</li> <li>The prior TAF duration (duration of TAF prior to study entry): &lt;1 year, &gt;=1 year</li> </ul> |

Subgroup analyses for endpoints will be presented as shown in the table below.

| | | Endpoint | | |
|---|---|---|---|---|
| Subgroup | Proportion of patients with plasma HIV-1 RNA <50 <sup>5</sup> copies c/mL <sup>6</sup> | Summary of<br>Study<br>Snapshot<br>outcomes<br>(Plasma HIV-<br>1 RNA >=/<<br>50 c/mL) | CD4+ Cell<br>Count and<br>CD4+/CD8+<br>Ratio Change<br>from Baseline | AEs <sup>7</sup> |
| Baseline third agent class (PI, NNRTI, INI) | Y | Y | Y | Y |
| Age (years): <35, 35 to <50, ≥50 | Y | Y | Y | Y |
| Age (years): <50, ≥50 | Y | Υ | | |
| Gender: Male & Female | Υ | Υ | Υ | Υ |
| Baseline CD4+ cell count: <200, 2<br>00 to <350, ≥350 cells/mm3 and<br><500, ≥500 cells/mm3 and <350,<br>≥350 cells/mm³ | Y | Y | Y | Y |
| CDC HIV-1 classification: Stage 0-3 | Y | Y | Y | Y |
| Country | Y | Y | | |
| Race: White, Black or African<br>American, Asian, Other | Y | Y | Y | Y |
| Race: White, non-white | Υ | Υ | Υ | |

# 5.5. Multiple Comparisons and Multiplicity

The primary comparison of interest is the comparison between DTG + 3TC and TBR for the primary endpoint in the ITT-E population. This analysis will be adjusted for by the actual stratification factor as determined from the eCRF data (not as recorded in IVRS) randomisation.

No adjustment for multiplicity is required as there is only one primary comparison of interest.

<sup>&</sup>lt;sup>5</sup> A sensitivity analysis will also be performed for the following endpoint: HIV-1 RNA <40 c/mL and Target Not Detected Status. See Section 7.2.5 for more details. This subgroup analysis is not applicable post Week 48.

<sup>&</sup>lt;sup>6</sup> Includes forest plot for unadjusted difference of patients with plasma HIV1 RNA <50 copies c/mL between treatment arms.

<sup>&</sup>lt;sup>7</sup> Subgroup analyses will be presented for the following analyses: Adverse Events by System Organ Class, Maximum Toxicity; and Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study (see Section 13.15 Full Data Displays for more information). Not applicable to analyses post Week 48.

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---|---|
| Section 13.1 | Appendix 1: Protocol Deviation Management |
| Section 13.2 | Appendix 2: Schedule of Activities |
| Section 13.3 | Appendix 3: Assessment Windows |
| Section 13.4 | Appendix 4: Study Phases and Emergent Adverse Events |
| Section 13.5 | Appendix 5: Data Display Standards & Handling Conventions |
| Section 13.6 | Appendix 6: Derived and Transformed Data |
| Section 13.7 | Appendix 7: Reporting Standards for Missing Data |
| Section 13.8 | Appendix 8: Values of Potential Clinical Importance |
| Section 13.9 | Appendix 9: Population Pharmacokinetic (PopPK) Analyses |
| Section 13.10 | Appendix 10: Time to Event Details |
| Section 13.11 | Appendix 11: Snapshot |
| Section 13.12 | Appendix 12: Abbreviations & Trade Marks |
| Section 13.13 | Appendix 13: Model Checking and Diagnostics for Statistical Analyses |
| Section 13.14 | Appendix 14: COVID-19 Modified Analysis and Supportive Sensitivity Analyses |
| Section 13.15 | Appendix 15: List of Data Displays |
| Section 13.16 | Appendix 16: Example Mock Shells for Data Displays |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Intent-To-Treat Exposed (ITT-E) population, unless otherwise specified.

Table 1 provides an overview of the planned study population analyses, with full details of data displays being presented in Section 13.15: List of Data Displays.

Table 1 Overview of Planned Study Population Analyses

| Display Type | Data Displays Generated | |
|---|---|---|
| | Table | Listing |
| Randomisation | | |
| Randomisation | | Υ [1] |
| Subject Disposition | | |
| Subjects Enrolled by Country and Site ID [2] | Y | Y |
| History of Rescreened Subjects[2] | | Υ |
| Reasons for Screen Failure [2] | Y | Υ |
| Subject Disposition | Υ[3,4, 11,12] | |
| Reasons for Withdrawal by Visit | Υ[11,12] | Υ |
| Study Visit Dates | | Υ |
| Populations Analysed | | |
| Study Populations [2] | Y | Υ |
| Protocol deviations | | |
| Important Protocol Deviations | Υ [11,12,13] | Y |
| Deviations leading to exclusion from PP | Y | Υ |
| Inclusion and Exclusion Criteria Deviations | | Y |
| Demography and baseline characteristics | | |
| Demographic Characteristics <sup>[5]</sup> | Υ <sup>[12]</sup> | Υ |
| Summary of Age Ranges | Y | |
| Race & Racial Combinations <sup>[6]</sup> | Υ <sup>[12]</sup> | Υ |
| Hepatitis C Status | Υ[12] | Υ |
| CDC Classification of HIV infection at Baseline | Υ[12] | Υ |
| HIV Risk Factor | Υ[12] | Υ |
| Cardiovascular Risk Assessments at Baseline | Υ <sup>[12]</sup> | Y |
| Distribution of Quantitative Plasma HIV-1 RNA | Υ[12] | Υ |
| Distribution of CD4+ Cell Counts | Υ[12] | Υ |
| History of Cardiac Therapeutic Procedures | | Υ |
| Medical Conditions, Concomitant Medications & A | Antiretroviral Therap | у |
| Medical Conditions (Current and Past) | Υ[11,12] | Y |
| Medical Conditions: Sub-conditions (Current/Past) | Υ[11,12] | |
| Concomitant Medications (non-ART) | <b>Y</b> [7,11,12] | <b>Y</b> [8] |
| Prior,Concomitant ART and post ART Medications | Υ[11,12] | <b>Y</b> [9] |
| Baseline third agent class (Strata) [10] | Υ[12] | Y |
| Lipid Modifying agents (Baseline and Post-Baseline) | Υ[11,12] | |

| Display Type | Data Displays Generated | |
|---|---|---|
| | Table | Listing |
| Other | | |
| History of Depression and Anxiety at Baseline | Υ[12] | |
| Summary of Past and Current Cardiac,<br>Gastrointestinal, Metabolism and Nutrition,<br>Psychiatric, Renal and Urinary, and Nervous<br>System Conditions | Υ[11,12,13] | |
| History of Cardiac Therapeutic Procedures | | Y |
| Investigational Product Accountability | | Y |
| Important COVID-19 Protocol Deviations | Υ [11,12,13] | |
| Important non-COVID-19 Protocol Deviations | Υ [11,12,13] | |
| Non-important COVID-19 Protocol Deviations | | Y |
| Summary of COVID-19 Pandemic Assessments and Visit Impacts | Υ[11,12,13] | Y |

#### NOTES:

- Y = Display Generated, T = Tables, L = Listings, IP = Investigational Product
- 1. ITT-E. One listing of subjects randomised but not treated, and one listing of planned and actual treatment strata.
- 2. ITT-E and All Subjects screened population.
- 3. Subject Accountability by Phase (Overall, Early Switch Phase, Late Switch Phase)
- 4. Subjects who have not been recorded as withdrawing from the study in the respective phase will be categorized as "Ongoing at time of the analysis" for summary purposes.
- 5. Age, sex, ethnicity, weight, height, BMI (kg/m^2) and child-bearing potential collected at screening.
- 6. The five high level FDA race categories and designated Asian subcategories will be summarised along with all combinations of high level categories which exist in the data. The nine race categories collected will be summarised along with categories for mixed race. A by-subject listing of race will also be produced.
- 7. Three separate tables, summarised by: 1) Ingredient ATC Level 1, 2) Ingredient combinations and 3) Combination term ATC Level 1 (EG Includes single-ingredient medications with multi-ingredient medications labelled according to the sum of their ingredients, e.g., "TYLENOL Cold and Flu" would appear as "CHLORPHENAMINE MALEATE + DEXTROMETHORPHAN HYDROBROMIDE + PARACETAMOL + PSEUDOEPHEDRINE HYDROCHLORIDE" under the ATC headings for "Nervous System" and "Respiratory System" (the combination's ATC classifications).)
- 8. One listing for concomitant non-ART medications, one listing showing the relationship between verbatim text, ingredient and ATC Level 1 and and one listing showing the relationship between verbatim text, ingredient, combination and ATC Level 4.
- 9. One listing for Prior ART, one listing for ART received at screening, one listing for concomitant ART starting after screening while still on-treatment and one listing for post ART.
- 10. Based on the actual third agent class that subjects were classified into according to data captured on the eCRF.
- 11. Repeat for the Early + Late Switch Phase for the DTG+3TC am
- 12. Repeat for the Late Phase for the TBR arm
- 13. Include Week 200 data

#### 7. EFFICACY ANALYSES

## 7.1. Primary Efficacy Analysis

## 7.1.1. Summary Measure

Proportion of subjects with plasma HIV-1 RNA ≥50 copies c/mL at Week 48 using the snapshot algorithm.

## 7.1.2. Population of Interest

The primary efficacy analyses will be based on the Intent-To-Treat Exposed (ITT-E) population unless otherwise specified.

## 7.1.3. Strategy for Intercurrent (Post-Randomisation) Events

Intercurrent events will be accounted for as per the FDA snapshot algorithm.

# 7.1.4. Statistical Analyses / Methods

Details of the planned displays are provided in Section 13.15: List of Data Displays and will be based on GSK data standards and statistical principles commonly applied in GSK HIV-1 trials.

Table 2 provides an overview of the planned efficacy analyses, with full details of data displays being presented in Section 13.15: List of Data Displays.

| Table 2 Overview of Planned Prin | nary Efficacy Analyses |
|----------------------------------|------------------------|
|----------------------------------|------------------------|

| | Absolute | | | | | | |
|---|---|---|---|---|---|---|---|
| Endpoint | Stats Analysis | | | Summary | | Individual | |
| | T | F | L | Т | F | F | L |
| Proportion of Subjects with plasma HIV 1 RNA ≥50 copies c/mL at week 48 – Snapshot | | | | | | | |
| Primary Analysis | <b>Y</b> [1] | | <b>Y</b> [4] | | | | |
| Study Outcome [2] | | | | Υ | | | Υ |
| based on the | | | | | | | |
| Snapshot | | | | | | | |
| Sparse Data | <b>Y</b> [5] | | | | | | |
| Analysis | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
  - [1] Generated using the 'Intent-to-Treat Exposed' (primary), 'Per-Protocol' and 'Intent-to-Treat' (sensitivity) populations.
  - [2] Study outcomes (i.e., virologic failure, virologic success (response below 50 c/mL) or no virologic data at Week X window) based on the snapshot algorithm.
  - [3] Line plots, with 95% confidence intervals, for the proportion of subjects with virologic failure by treatment group at each visit.
  - [4] Listing of Quantitative and Qualitative Plasma HIV-1 RNA Data based on the snapshot algorithm.
  - [5] See methodology section below for more information.

### 7.1.4.1. Statistical Methodology Specification

#### **Endpoint**

- Proportion of subjects with plasma HIV 1 RNA ≥50 copies c/mL at Week 48 using the Snapshot algorithm for the ITT-E population
- The Snapshot algorithm treats all subjects without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of IP prior to the visit window) as non-responders. The nature of this missing data will be further classified in Snapshot summaries as either 'Virologic Failure' or 'No Virologic Data at Week 48'. Subjects who change their ART regimen prior to the visit of interest will be considered virologic failures since changes in ART are not permitted in this protocol (with the exception of a change in the booster ART as detailed below).
- 'Virologic failure' includes subjects who changed any ART; subjects who discontinued study drug or study before Week 48 for lack or loss of efficacy, discontinued for other reason while not < 50 c/mL, and subjects who have HIV-1 RNA ≥ 50 c/mL at the visit of interest.</li>
- Virologic success includes subjects who have HIV-1 RNA <50 c/mL at the visit of interest.</li>
- The only protocol-permitted substitutions are as follows:
  - A switch from a PI boosted with RTV to the same PI boosted with cobicistatis allowed.
  - A switch from a PI boosted with cobicistat to the same PI boosted with RTV is allowed.

Virologic success or failure will be determined by the last available HIV-1 RNA assessment while the subject is On-treatment within the visit of interest analysis window see Section 13.3. Full details of the Snapshot algorithm are in Section 13.11. Note: for Week 96 reporting onwards, refer to Section 13.14.1 instead for Modified Snapshot algorithm in presence of COVID-19 missing data.

#### **Model Specification**

- The primary endpoint will be analysed using a stratified analysis with Cochran-Mantel-Haenszel (CMH) weights, adjusting for baseline third agent class (PI, NNRTI, INI).
- The CMH estimate of the adjusted treatment difference will be calculated as a weighted average of strata-specific estimates of the treatment difference calculated within each of the following three Baseline analysis strata:
  - o Baseline third agent: PI
  - Baseline third agent: NNRTI
  - Baseline third agent: INI
- If  $n_k$  is the number of DTG + 3TC treated subjects,  $m_k$  is the number of PI-, NNRTI- or INI-based ART treated subjects, and  $N_k = n_k + m_k$  is the total number of subjects in the kth stratum, then the CMH estimate is given by:

$$\hat{d}_{cmh} = \frac{\sum W_k \hat{d}_k}{\sum W_k}$$

where,

$$W_k = \frac{n_k m_k}{N_k}$$

are CMH weights and  $d_k$  are estimates of the differences in virologic failure proportions between the two treatment arms,  $r_d$ - $r_a$ , for the kth strata.

• The corresponding two-sided 95% CI will be calculated as

$$\hat{d}_{cmh} \pm 1.96 \times \sqrt{\hat{\text{var}}(\hat{d}_{cmh})}$$

using the variance estimator,  $var(d_{cmh})$ , given by [Sato ,1989], which is consistent in both sparse data and large strata.

$$\operatorname{var}(\hat{d}_{cmh}) = \frac{\hat{d}_{cmh}(\sum P_k) + \sum Q_k}{\left(\sum n_k m_k / N_k\right)^2} = \frac{\hat{d}_{cmh}(\sum P_k) + \sum Q_k}{\left(\sum W_k\right)^2}$$

where

$$P_k = \frac{n_k^2 y_k - m_k^2 x_k + n_k m_k (m_k - n_k)/2}{N_k^2}$$

$$Q_k = \frac{x_k (m_k - y_k) / N_k + y_k (n_k - x_k) / N_k}{2}$$

## **Model Checking & Diagnostics**

Not applicable

#### Model Results Presentation

- Adjusted CMH estimate of the difference in the proportion of virologic failure between each treatment group (DTG + 3TC – TBR) and corresponding 95% confidence interval.
- Non-inferiority will be concluded if the upper bound of the two-sided 95% confidence interval
  (CI) for the CMH adjusted difference in the proportion of patients with virologic failure in the
  DTG+3TC group minus the proportion of patients with virologic failure in the TBR group is
  less than 4%.
- If ITT-E and Per Protocol analyses show non-inferiority (see Sensitivity and Supportive Analyses section below), then a superiority hypothesis will be tested at the two-sided 5% level of significance. Superiority favouring DTG + 3TC will be declared if the upper bound of two-sided confidence interval is below 0%. If superiority is declared, the p-value for superiority will also be presented. Figures: Line plots, with 95% confidence intervals, for the proportion of subjects >= 50 c/mL as per the FDA snapshot by treatment group at each visit (not applicable to analyses post Week 48).

## Subgroup Analyses

Subgroup analyses will not be performed for this endpoint

## Sensitivity and Supportive Analyses

- 1. Per-Protocol population analysis:
  - To assess the impact of significant protocol deviations, statistical analysis will be repeated using the Per-protocol population and compared for consistency with the results from the primary ITT-E population analysis. If both analyses show non-inferiority then the hypothesis that the antiviral effect of treatment with DTG + 3TC is superior to treatment with TBR will be tested at the two-sided 5% level of significance (as described above).
- 2. Intent-to-Treat population analysis:
  - Statistical analysis will be repeated using the Intent-to-Treat population and compared for consistency with the results from the ITT-E and PP populations.
  - In this analysis, subjects randomised but not exposed to study treatment will be classified as non-responders.
- 3. A sensitivity analysis will be conducted to assess the impact of sparse data (Miettinen, 1985).
  - The estimate is computed from Miettinen-Nurminen (score) confidence limits for the stratum risk differences. The score confidence interval for the risk difference in stratum h can be expressed as  $\hat{d}_h' \pm z_{\alpha/2} s_h'$ , where  $\hat{d}_h'$  is the midpoint of the score confidence interval and  $s_h'$  is the width of the confidence interval divided by  $2z_{\alpha/2}$ . The summary score estimate of the common risk difference is computed as:

$$\hat{d}_S = \sum_h \hat{d}'_h w'_h$$

where

$$w'_h = (1/{s'_h}^2)/\sum_i (1/{s'_i}^2)$$

The variance of  $\hat{d}_S$  is computed as

$$\sigma^2(\hat{d}_S) = 1/\sum_h (1/s_h'^2)$$

The  $100(1-\alpha)\%$  summary score confidence limits for the common risk difference are:

$$\hat{d_S} \pm \left(z_{\alpha/2} \times \hat{\sigma}(\hat{d_S})\right)$$

## 7.2. Secondary Efficacy Analyses

## 7.2.1. Endpoint / Variables

- Patients with plasma HIV 1 RNA ≥50 copies c/mL at week 24, 96 and 144.
- Patients with plasma HIV 1 RNA <50 copies c/mL at weeks 24, 48, 96 and 144.
- CD4+ cell count at Weeks 24, 48, 96 and 144.
- CD4+/CD8+ cell count ratio at Weeks 24, 48, 96 and 144.
- Incidence of disease progression (HIV-associated conditions, AIDS, and death) through Weeks 24, 48, 96 and 144.

# 7.2.2. Summary Measures

- Proportion of subjects with plasma HIV 1 RNA ≥50 copies c/mL at weeks 24, 96 and 144 using the snapshot algorithm.
- Proportion of subjects with plasma HIV 1 RNA <50 copies c/mL at weeks 24, 48, 96 and 144 using the snapshot algorithm.
- Change from baseline in CD4+ cell count at Weeks 24, 48, 96 and 144.
- Change from baseline in CD4+/CD8+ cell count ratio at Weeks 24, 48, 96 and 144.
- Incidence of disease progression (HIV-associated conditions, AIDS, and death) through Weeks 24, 48, 96 and 144.

## 7.2.3. Populations of Interest

The secondary efficacy analyses will be based on the ITT-E population.

## 7.2.4. Strategy for Intercurrent (Post-Randomisation) Events

Intercurrent events will be accounted for as per the FDA snapshot algorithm for the analyses of secondary endpoints of plasma HIV 1 RNA <50 copies c/mL and plasma HIV 1 RNA ≥50 copies c/mL. Intercurrent events will not be controlled for in disease progression and CD4+ cell count analyses. Intercurrent events as a result of COVID-19 will be accounted for as per the Modified Snapshot algorithm (see Section 13.14.1) for analyses post-Week 48.

#### 7.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 15: List of Data Displays.

Table 3 provides an overview of the planned secondary efficacy analyses, with full details of data displays being presented in Appendix 15: List of Data Displays.
Table 3 Overview of Planned Secondary Efficacy Analyses

| Endpoints | | | Ak | solut | е | | | | С | han | ge froi | n Ba | selin | е |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats | s Analys | sis | Sum | mary | Indiv | idual | Stats<br>Analysis | | | Summ | nary | Indi | vidual |
| | T | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Proportion of Subje | ects wit | h Plası | na HI | V-1 RI | NA ≥5 | 0 сор | ies/ml | \$ | Snap | sho | ot | | | |
| Secondary<br>analysis at Weeks<br>24, 96 and 144 | <b>Y</b> [15] | | Υ | | | | | | | | | | | |
| Study Outcome<br>based on the<br>Snapshot at<br>Weeks 24, 96 and<br>144 | | | | <b>Y</b> [14] | | | Y | | | | | | | |
| By Visit | | | | Υ | | | | | | | | | | |
| Proportion of subjects without virologic or virologic/tolerability failure at Week | Υ | <b>Y</b> [11] | | | | | Υ | | | | | | | |
| Proportion of Subj | ects wit | h Plası | na HI | V-1 RI | NA <50 | ) сор | ies/mL | . – \$ | Sna | psh | ot | | | |
| Secondary<br>analysis at Week<br>X <sup>[6]</sup> | <b>Y</b> [12,1 3, 15] | | | | | | | | | | | | | |
| Secondary<br>analysis by Visit<br>through Week X <sup>[6]</sup> | | | | Y | Y | | | | | | | | | |
| Secondary<br>analysis by<br>subgroup at Week<br>X <sup>[6]</sup> | | | | Υ | <b>Y</b> [1] | | | | | | | | | |
| Study Outcomes at Week X <sup>[6]</sup> | | | | <b>Y</b> [12, 16] | | | | | | | | | | |
| Study Outcomes<br>by subgroup at<br>Week X <sup>[6]</sup> | | | | Υ | | | | | | | | | | |

| Endpoints | | | Al | osolut | е | | | | С | har | nge fror | n Ba | selin | е |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | s Analy | sis | Sum | mary | Indi | idual | | Stats | | Summ | nary | Indi | vidual |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Confirmed Virologi | ic With | drawal | (CW | () | | | | | | | | | | |
| CVW by Visit | Υ | | | | | | Υ | | | | | | | |
| HIV-1 RNA distribution at time of suspected and confirmed Virologic withdrawal | Y | | | | | | | | | | | | | |
| Potential Precaution | nary V | irologi | c With | ndrawa | al (pP\ | W) | | | | | | | | |
| pPWW by Visit | | | | | | | Υ | | | | | | | |
| Plasma HIV-1 RNA | over tii | ne – C | bser | ved | | | | | | | | | | |
| By Visit through<br>Week X <sup>[6]</sup> | | | | | | <b>Y</b> [2] | <b>Y</b> [2,9] | | | | <b>Y</b> [5,16] | | | |
| CD4+ Cell Counts <sup>[3</sup> | ] | | | | | | | | | | | | | |
| By Visit through<br>Week X <sup>[6]</sup> | | | | | | <b>Y</b> [2] | Υ | | | | <b>Y</b> [16] | | | Υ |
| By Subgroup at<br>Week X <sup>[6]</sup> | | | | | | | | | | | Υ | | | |
| CD4+/CD8+ Cell Co | unt Ra | tio <sup>[3]</sup> | | | - | | • | | | | | | | |
| By Visit through<br>Week X <sup>[6]</sup> | | | | | | <b>Y</b> [2] | Υ | | | | <b>Y</b> [16] | | | Υ |
| By Subgroup at<br>Week X <sup>[6]</sup> | | | | | | | | | | | Υ | | | |
| Post-baseline HIV- | l Disea | se Pro | gress | ion <sup>[4]</sup> | | | | | | | | | | |
| HIV Conditions including Recurrences at Week X <sup>[6,7]</sup> | | | | <b>Y</b> [16, | | | Y | | | | | | | |
| HIV Conditions<br>excluding<br>Recurrences at<br>Week X <sup>[6,7]</sup> | | | | <b>Y</b> [16, | | | | | | | | | | |
| HIV Disease<br>Progressions at<br>Week X <sup>[6,8]</sup> | | | | <b>Y</b> [16, | | | | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed rawdata.
- Individual = Represents FL related to any displays of individual subject observed raw data.
  - 1. Plot of 95% confidence intervals for unadjusted treatment difference in the proportion of subjects below 50 c/mL with overall and by subgroup.
  - 2. Individual plasma HIV-1 RNA and CD4+ profiles only for subjects with at least one HIV-1 RNA levels ≥ 50 c/mL observed including at Day 1 and through withdrawal visit.
  - 3. Using observed case (OC) data which contains the data that is available at a particular time point, with no imputation for missing values.
  - 4. HIV disease progressions categories: CDC Category Stage 1 at enrolment to Stage 3 event, CDC Category Stage 2 at enrolment to Stage 3 event, CDC Category Stage 3 at enrolment to New Stage 3 Event, CDC Category Stage 1, 2 or 3 at enrolment to Death.
  - 5. Descriptive summary of the log10 change from baseline HIV-1 RNA by visit presented.
  - 6. Week X refers to Week 96 and week 144.
  - 7. Stage 3 only.
  - 8. Progression to Stage 3 or death.
  - 9. Includes target detected/not detected flag see Section 13.6.3 for more information.
  - 10. Outputs will be produced for Efficacy related discontinuation = Failure (ERDF) and Treatment related discontinuation = Failure (TRDF).
  - 11. Kaplan-Meier Plot of Time to Failure ERDF/TRDF.
  - 12. Repeated on the following endpoints: <40 c/mL and <40 c/mL and TargetNotDetected Status. For Week 96 reporting onwards, analyses will be based on Modified Snapshotalgorithm relevant to 40 c/mL and <40 c/mL and TargetNotDetected Status endpoints (see Section 13.14.1 for more details)
  - 13. Repeated for the withdrawal bias sensitivity analysis
  - 14. To be based on Modified Snapshotalgorithm (see Section 13.14.1 for more details). Note this is only relevant to analyses performed at Week 96 onwards.
  - 15. Repeated as a sensitivity analysis based on Evaluable Efficacy Population (see Section 13.14.1 for more details), for endpoints HIV-1 RNA >=50 c/mL, <50 c/mL and <40 c/mL and TND. Note this is only relevant to analyses performed at Week 96 onwards.
  - 16. Repeat for the Early + Late Switch Phase for the DTG+3TC arm and for the Late Phase for the TBR arm
  - 17. Week 200 data to be included

## 7.2.5.1. Statistical Methodology Specification

#### Endpoint

- Proportion of subjects with plasma HIV 1 RNA ≥50 copies c/mL at Weeks 24, 96 and 144, and plasma HIV 1 RNA <50 copies c/mL at Week 24, Week 48, Week 96 and Week 144 using the Snapshot algorithm for the ITT-E population.
- The analysis approach will follow the methods as described for the primary endpoint.

### **Model Specification**

Specification will be same as described for the primary endpoint

#### **Model Checking & Diagnostics**

Same as described for the primary endpoint

#### Model Results Presentation

Model presentation will be the same as described for the primary endpoint.

- Proportion subjects with plasma HIV 1 RNA ≥50 copies c/mL will be analysed at Weeks 24, 96 and 144. Proportion subjects with plasma HIV 1 RNA <50 copies c/mL will be analysed at Week 24, Week 48, Week 96 and Week 144
- For virologic success (plasma HIV-1 RNA <50 c/mL) endpoint, non-inferiority of switching to DTG + 3TC compared to continuation of TBR (as per FDA snapshot algorithm) will be assessed using a -8% non-inferiority margin. Non-inferiority will be concluded if the lower bound of a 2-sided 95% confidence interval for the difference in success rates between the two treatment arms is greater than -8%. Figures: Line plots, with 95% confidence intervals (figures not applicable for analyses post Week 48).</li>

## Subgroup Analyses

 Subgroup analyses will be performed for the proportion of patients with plasma HIV 1 RNA <50 copies c/mL, study outcomes and unadjusted difference in proportion of patients with plasma HIV 1 RNA <50 copies c/mL between treatment arms forest plot at Week 24,Week 48, Week 96 and Week 144 endpoints only.

## **Sensitivity and Supportive Analyses**

- 1. A sensitivity analysis will be performed on the proportion of patients with plasma HIV-1 RNA <50 c/mL endpoint at Week 48, Week 96 and Week 144. For this analysis, patients who withdrew from the study due to the prolongation of the study as defined in the protocol amendment 6 (as captured on the study discontinuation CRF) before providing virologic data within the analysis window of interest will be removed from the denominator in both arms. The purpose of this analysis is to investigate the impact of snapshot categorisation bias that may be introduced in the event of a higher withdrawal rate in the TBR arm. The Cochran-Mantel-Haenzel approach will then be followed as described in the primary analysis section.</p>
- 2. A sensitivity analysis based on the <50 HIV-1 RNA endpoint will be performed based on the same analysis for the following endpoints:
- Proportion of Subjects with Plasma HIV-1 RNA <40 c/mL at Week X</li>
- Proportion of Subjects with Plasma HIV-1 RNA <40 c/mL and Target Not Detected Status at Week X
- Proportion of Subjects with Plasma HIV-1 RNA <40 c/mL and Target Not Detected Status at Week X by Baseline Third Agent Class (not applicable for analyses post Week 48)
- 3. Proportion of subjects without virologic (ERDF) or virologic/tolerability (TRDF) failure:
- Estimated using the Kaplan-Meier nonparametric method based on the time to Confirmed Virologic Withdrawal (CWW) criteria met or treatment-related (i.e. drug-related AE, protocol defined safety stopping criteria, or lack of efficacy)/efficacy related discontinuation (i.e. lack of efficacy).
- The detailed algorithm for TRDF (and ERDF) is listed in Section 13.10. The estimate of the standard error used to derive confidence intervals for the difference in proportions between treatment groups will be based on Greenwood's formula [Kalbfleisch, 1980]
- The estimated proportion of subjects without Confirmed Virologic Withdrawal and not discontinued due to treatment-related/efficacy-related reasons at Week X will be presented by treatment group, along with estimated difference in proportions between treatment groups and its associated two-sided 95% CI.

## 7.3. Exploratory Efficacy Analyses

## 7.3.1. Endpoint / Variables

Randomised Early Switch Phase analyses:

- Subjects with plasma HIV-1 RNA <50 c/mL using the Snapshot algorithm at Week 24, 48, 96 and 144 by subgroup, based on the ITT-E population.
- Change from baseline CD4+ and CD4+/CD8+ ratio cell counts at Week 24, 48, 96 and 144 by subgroup

For subjects in the DTG + 3TC arm since Early Switch Phase and for subjects (TBR arm) switching to DTG + 3TC in the Late Switch Phase:

- Proportion of subjects with plasma HIV-1 RNA <50 c/mL at Week 196 using the Snapshot algorithm for the ITT-E population for DTG+3TC arm and LS-ITT-E population for subjects in TBR arm switched to DTG+3TC in the Late Switch Phase
- Change from Baseline in CD4+ lymphocyte count and in CD4+/CD8+ cell count ratio at Week 196
- Incidence of disease progression (HIV associated conditions, AIDS and death) through Week 196

These analyses have been specified in previous sections.

## 8. SAFETY ANALYSES

The safety analyses will be based on the Safety population (and Late-Switch Safety Population, where applicable), unless otherwise specified.

For Week 24, 48 96 and 144 analyses, outputs will be presented for the Early Switch Phase unless otherwise specified.

For W196 analysis,\

- For subjects in the DTG + 3TC arm since Early Switch Phase, outputs will be presented for Early and Late Switch Phase [DTG + 3TC arm only]
- For subjects switching to DTG + 3TC in the Late Switch Phase, outputs will be presented for Late Switch Phase [TBR arm switching to DTG + 3TC]).

Safety data presented through weeks 24,48, 96, 144 and 196 will comprise all available safety data collected at that time point within the phase reported. The safety endpoints collected at Week 200 will be included in Week 196 outputs.

## 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 15: List of Data Displays.

Emergent AEs will be tabulated by treatment group and a total column. For AEs captured more than once, the most severe intensity will be included in summaries, and all events will be included in listings. For the purposes of summarising AE data, unless stated otherwise, the summaries will include post-baseline data.

In the event withdrawal rate due to PAM6 study design change is higher in the TBR arm, similar sensitivity analyses to that stated for the HIV-1 RNA <50 c/mL endpoint as detailed in Section 7.2.5.1 considered for some AE analyses at Weeks 96 and 144.

Table 4 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 15: List of Data Displays.

Table 4 Overview of Planned Safety Analyses

| Endpoint | Absolu | te | | |
|---|---|---|---|---|
| | Sum | mary | Indi | vidual |
| | T | F | F | L |
| Exposure | | | | |
| Extent of Exposure | <b>Y</b> [1] [9] | | | <b>Y</b> [2] |
| Adverse Events[3] | | | | |
| All AEs by SOC and PT | <b>Y</b> [1] [9] | | | Y |
| All AEs by Maximum Grade[3] | <b>Y</b> [9] | | | <b>Y</b> [4] |
| Common AEs by freq [5] | <b>Y</b> [9] | <b>Y</b> [6] | | |
| Common Grade 2-5 AEs [5]<br>by freq | <b>Y</b> [9] | | | |
| Drug-Related AEs by SOC and PT | <b>\</b> [9] | | | Y |
| All Drug-Related AEs by<br>SOC and Maximum Grade <sup>[3]</sup> | <b>Y</b> [1] [9] | | | |
| Common non-Serious AEs<br>by SOC and PT (subjects<br>and number of occurrences) | Υ | | | |
| Common Drug-related Grade 2-5 AEs [5] | <b>Y</b> [9] | | | |
| Common Non-Serious AEs<br>(FDAAA) | <b>Y</b> [9] | | | |
| Cumulative AEs by visit | Υ | | | |

| Endpoint | Absolu | ute | | |
|---|---|---|---|---|
| | Sum | nmary | Indiv | idual |
| | T | F | F | L |
| Drug-Related AE leading to withdrawal from study | <b>\</b> [9] | | | |
| AEs Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment <sup>[8]</sup> | <b>Y</b> [1] [9] | | | Y |
| Serious and Other Significa | nt AEs | | | |
| All SAEs by SOC | <b>Y</b> [1] [9] | | | |
| Fatal SAEs | | | | Y |
| Non-Fatal SAEs | | | | Y |
| All Drug-Related SAEs by SOC | <b>Y</b> [9] | | | |
| Drug-Related Non Fatal<br>Serious AEs | | | | Y |
| Drug-Related Fatal Serious<br>AEs | <b>Y</b> [9] | | | Y |
| Serious AEs by SOC and PT | <b>Y</b> [9] | | | |
| Reason for Considering as a Serious Adverse Event | | | | Y |
| Possible Suicidality-Related<br>Adverse Event (PSRAE) | | | | <b>Y</b> [7] |
| Cardiovascular events | | | | Y |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Repeat for the Early + Late Switch Phase for the DTG+3TC arm and for the Late Phase for the TBR arm (Late Phase outputs to be included in an amendment of the RAP).
- 2. Includes reason for any dose change/interruption in both arms.
- 3. For AEs reported more than once by a subject, the most severe intensity will be included.
- 4. One listing of all AEs including verbatim text and preferred term, one showing the relationship between verbatim text, preferred term and SOC and another giving subject numbers for individual all treatment emergent AEs.
- 5. Common AEs are those with >=2% (or 0.5% for drug-related grade 2-5 AEs) incidence in either treatment group summarised by frequency.
- 6. Plots of incidence rates and relative risk with 95% CI for DTG+3TG vs. TBR.
- 7. Four PSRAE listings: Event and Description (Section 1 to Section 2), Possible Cause (Section 3), Section 4 and Section 5 to Section 8 (see ICH Listings Section 13.15.14).
- 8. Repeated by maximum grade as well.
- 9. Repeat for the Early + Late Switch Phase for the DTG+3TC arm and for the Late Phase for the TBR arm at Week 196 and including Week 200 datag

## 8.2. Adverse Events of Special Interest Analyses

A comprehensive list of MedDRA terms based on clinical review will be used to identify each type of event. Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting and/or emerging data from on-going studies may highlight additional adverse events of special interest, therefore the list of terms to be used for each event of interest and the specific events of interest will be based on the safety review team (SRT) agreements in place at the time of reporting. An overview of the planned adverse events of special interest analyses are presented in Table 5 and full details of the planned displays are provided in Appendix 15: List of Data Displays.

Table 5 Overview of Planned Adverse Events of Special Interest Analyses

| Endpoint | Absolu | te | | |
|---|---|---|---|---|
| | Sum | mary | Indiv | idual |
| | T | F | F | L |
| Adverse Events of Special Interest | | | | |
| Characteristics of Post<br>Baseline AESI | <b>Y</b> [1] | | | |
| Onset and Duration of the First Occurrence of Post Baseline AESI | <b>Y</b> [1] | | | |
| Post Baseline Depression, Suicidal and Self-Injury Adverse Events by AE of Special Interest, Maximum DAIDS ToxicityGrade, and Prior History of Depression and Anxiety | <b>Y</b> [1] | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Repeat for the Early + Late Switch Phase for the DTG+3TC arm and for the Late Phase for the TBR arm at Week 196 and including Week 200 data

## 8.3. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and Liver Function tests will be based on GSK Core Data Standards. Table 6 provides an overview of the planned laboratory analyses, with full details of data displays being presented in Appendix 15: List of Data Displays.

Table 6 Overview of Planned Laboratory Analyses

| Endpoint | | Α | bsol | ute | C | Change from Baseline | | | | | | Max Post BL | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sum | mary | Indi | vidual | Summary | | Indiv | idual | Sta<br>Ana | | Sum | mary | Indiv | idual |
| | Т | F | F | L | Т | F | F | L | Т | F | T | F | F | L |
| Laboratory Values | Ove | r Time | е | | | | | | | | | | | |
| Clinical Chemistry | Υ | | | <b>Y</b> [1] | <b>Y</b> [9,10] | | | | | | | | | |
| Lipids (%) | | | | | <b>Y</b> [4,9] | | | | | | | | | |
| Fasted Lipid<br>(Triglycerides,<br>LDL, HDL and TC<br>and TC/HDL) | <b>Y</b> [4] | | | | <b>Y</b> [4] | | | | Υ | Υ | | | | |
| Hematology | Υ | | | <b>Y</b> [1] | <b>Y</b> [9,10] | | | | | | | | | |
| Urine Dipstick | | | | <b>Y</b> [1] | | | | | | | | | | |
| Urine<br>Concentration | | | | <b>Y</b> [1] | | | | | | | | | | |
| Liver Chemistries | | | | | | | | | | | | <b>Y</b> [2] | | |
| NCEP shifts in lipids | | | | | <b>Y</b> [4] [9] | <b>Y</b> [3,4] | | | | | <b>Y</b> [4] | <b>Y</b> [3,4] | | |
| Total<br>Cholesterol/HDL<br>ratio | | | | | <b>Y</b> [4] [9] | <b>Y</b> [3,4] | | | | | <b>Y</b> [4] | <b>Y</b> [3,4] | | |
| Biomarkers | | • | | | • | | • | • | | | | | • | |
| Bone biomarkers | | | | Υ | <b>Y</b> [9] | | | Υ | Υ | Υ | | | | |
| Bone biomarkers (%) | | | | | | | | Υ | | | | | | |
| Renal biomarkers | | | | Υ | <b>Y</b> [9] | | | Υ | Υ | Υ | | | | |
| Renal biomarkers (%) | | | | | | | | Υ | | | | | | |
| Inflammation<br>Biomarkers | | | | Υ | <b>Y</b> [9] | | | Υ | Υ | Υ | | | | |
| Telomere length <sup>[8]</sup> | | | | Υ | <b>Y</b> [9] | | | Υ | | | | | | |
| Change from<br>baseline in HOMA-<br>IR at Week 24, 48,<br>96 and 144 | | | | Υ | <b>Y</b> [9] | | | Y | <b>Y</b> [5] | Y | | | | |
| HOMA-IR vs<br>weight scatter plot | | | | | | | <b>Y</b> [6] | | | | | | | |
| HOMA-IR shift table <sup>[7]</sup> | | | | | <b>Y</b> [9] | | | | | | Υ | | | |

| Endpoint | Absolute | | | | C | hang | e froi | m Bas | eline | ) | N | Max Post BL | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sum | mary | Indi | vidual | Sumi | mary | Indiv | idual | | ats<br>Iysis | Sum | mary | Indiv | idual |
| | Т | F | F | L | Т | F | F | L | T | F | Т | F | F | L |
| Emergent Laboratory Toxicities | | | | | | | | | | | | | | |
| Clinical Chemistry | | | | | | | | | | | <b>Y</b> [9,<br>10] | | | |
| Hematology | | | | | | | | | | | <b>Y</b> [9, 10] | | | |
| Fasting LDL<br>Cholesterol<br>Abnormalities of<br>Grade 2 or<br>Greater | | | | | | | | | | | <b>Y</b> [4]<br>[9] | | | |
| AST, ALT and<br>Total Bilirubin<br>Maximum Post-<br>Baseline<br>Emergent Toxicity<br>By Baseline<br>Hepatitis C Status | | | | | | | | | | | <b>Y</b> [9, 10] | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed rawdata.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Listings for subjects with abnormalities for potential clinical concern/importance, defined as any Grade1-5 toxicity.
- 2. Scatter plot of baseline vs. maximum post-baseline for ALT. Scatter plot of maximum ALT vs. maximum Bilirubin.
- 3. Bar chartfor LDL, HDL, TC, Trig and TC/HDL ratio.
- Subjects on lipid-lowering agents at baseline are not included in summaries, see Lipids. Section 13.7.2 for more details.
- 5. Not performed at Week 24. Also repeated on HOMA-IR >=2 endpoint (logistic regression) at Week 96 and Week 144 (dependent on degree of missing data resulting from COVID-19 see below for further details).
- 6. A scatter plot of change in HOMA-IR (y-axis) vs change in weight (x-axis) at Weeks 24, 48.
- 7. See Section 13.6.4 for more details.
- 8. Presented at Week 196 only.
- 9. Repeatfor the Early + Late Switch Phase for the DTG + 3TC arm and for the Late Phase for the TBR arm at Week 196
- 10. Week 200 data to be included

#### **Endpoints**

 Change from baseline in bone biomarkers marker (bone specific alkaline phosphatase, procollagen type I N-terminal propeptide, type I collagen cross-linked C-telopeptide, osteocalcin, 25-hydroxyvitamin D) at Weeks 24, 48, 96 and 144

#### **Covariates & Factors**

- Baseline 3<sup>rd</sup> Line Agent
- CD4+ cell count (continuous)
- Age (continuous)
- Sex (Female vs. Male)
- Race (White, Black or African American, Asian, Other)
- BMI (continuous)
- Smoking status (Never vs. Former vs. Current Smoker)
- Vitamin D use (Yes vs. No)

## **Data Handling**

No multiple imputation techniques will be used to deal with the missing data.

## **Model Specification**

- It is anticipated that at least some biomarkers will not be normally distributed and for those, the data will be log transformed and geometric means will replace arithmetic means, a 95% CI will replace the standard deviations and mean changes from baseline will be presented as geometric mean ratios.
- Change from baseline will be analysed for each bone biomarker for the comparison between DTG + 3TC and TBR.
- Mixed Model Repeated Measures (MMRM), using the observed margins (OM) option, will
  adjust for treatment, covariates (listed above) and biomarker value at baseline as a
  covariate, with visit as the repeated factor. The OC dataset will be used for MMRM model.
- The model will make no further assumptions about the correlations between a subject's value (the correlation matrix for within-subject errors will be unstructured).
- The repeated measures analysis will assume that the treatment difference can vary between visits (ie. a treatment\*visit interaction will be included in the model), and separates estimates and 95% confidence intervals will be produced at each visit. The model will also assume that the effect of baseline value for the endpoint can vary between visits (i.e. baseline value\*visit interaction will be included in the model).
- Interactions between treatment and each of the covariates will not be assessed.

## **Model Checking & Diagnostics**

• Refer to Section 13.13: Model Checking and Diagnostics for Statistical Analyses.

#### Model Results Presentation

- Adjusted least squares means and corresponding standard errors (SEs) of adjusted least squares means will be presented for each treatment, together with estimated treatment difference (DTG+3TC-TBR) and corresponding 95% confidence interval and p-value.
- Note: For biomarkers that are not normally distributed, the geometric mean and a 95% CI of geometric mean will be presented for each treatment, as well as geometric mean ratios and corresponding 95% CI and a p-value.

## **Sensitivity Analyses**

 Line plots of LS means with 95% confidence intervals for Adjusted Mean Change from Baseline will be generated for each treatment group by visit

## Subgroup Analyses

Not applicable

## Statistical Analyses

#### **Endpoints**

Change from baseline in renal biomarkers (serum Cystatin C, Urine Beta-2 Microglobulin /Urine Creatinine ratio (mg/mmol), urine albumin/creatinine ratio, urine protein/creatinine ratio, urine phosphate, eGFR (based on CKD-EPI-creatinine and CKD-EPI-cystatin C), serum creatinine and Urine Retinol Binding Protein 4/Urine Creatinine ratio (ug/mmol)) at Weeks 24, 48, 96 and 144

#### **Covariates & Factors**

- Baseline 3<sup>rd</sup> Line Agent
- CD4+ cell count (continuous)
- Age (continuous)
- Sex (Female vs. Male)
- Race (White, Black or African American, Asian, Other)
- BMI (continuous)
- Presence of diabetes mellitus (DM) (Yes vs no)
- Presence of Hypertension (Yes v no)

#### Data Handling

No multiple imputation techniques will be used to deal with the missing data.

- It is anticipated that at least some biomarkers will not be normally distributed and for those, the data will be log transformed and geometric means will replace arithmetic means, a 95% CI will replace the standard deviations and mean changes from baseline will be presented as geometric mean ratios.
- Change from baseline will be analysed for each renal biomarker for the comparison between DTG + 3TC and TBR.
- Using OC dataset, the Mixed Model Repeated Measures (MMRM), using the observed margins (OM) option, will adjust for treatment, covariates (listed above) and baseline renal biomarker value at baseline as a covariate, with visit as the repeated factor.
- The model will make no further assumptions about the correlations between a subject's value (the correlation matrix for within-subject errors will be unstructured).
- The repeated measures analysis will assume that the treatment difference can vary between visits (ie. a treatment\*visit interaction will be included in the model), and separate estimates and 95% confidence intervals will be produced at each visit. The model will also assume that the effect of baseline value for the endpoint can vary between visits (ie. baseline value\*visit interaction will be included in the model).
- Interactions between treatment and each of the covariates will not be assessed.

## **Model Checking & Diagnostics**

Refer to Section 13.13: Model Checking and Diagnostics for Statistical Analyses.

#### Model Results Presentation

- Adjusted least squares means and corresponding standard errors (SEs) of adjusted least squares means will be presented for each treatment, together with estimated treatment difference (DTG + 3TC – TBR) and corresponding 95% confidence interval and p-value.
- Note: For biomarkers that are not normally distributed, the geometric mean and a 95% CI of geometric mean will be presented for each treatment, as well as geometric mean ratios and corresponding 95% CI and a p-value.

## Sensitivity Analyses

 Line plots of LS means with 95% confidence intervals for Adjusted Mean Change from Baseline will be generated for each treatment group by visit

## Subgroup Analyses

Not applicable

## **Statistical Analyses**

## **Endpoints**

Change from baseline in inflammatory biomarkers (Interleukin-6 (IL-6), High-sensitivity C reactive protein (hs-CRP), D-dimer, Soluble CD14 (sCD14), Soluble CD163 (sCD163)) at Weeks 48, 96 and 144

#### Covariates & Factors

- Baseline 3<sup>rd</sup> Line Agent
- CD4+ cell count (continuous)
- Age (continuous)
- Sex (Female vs. Male)
- Race (White, Black or African American, Asian, Other)
- BMI (continuous)
- Smoking status (Never vs. Former vs. Current Smoker)
- HCV-coinfection (Yes vs. No)

#### **Data Handling**

No multiple imputation techniques will be used to deal with the missing data.

- It is anticipated that at least some biomarkers will not be normally distributed and for those, the data will be log transformed and geometric means will replace arithmetic means, a 95% CI will replace the standard deviations and mean changes from baseline will be presented as geometric mean ratios.
- Change from baseline will be analysed for each inflammatory biomarker for the comparison between DTG + 3TC and TBR.
- Using OC dataset, the Mixed Model Repeated Measures (MMRM), using the observed margins (OM) option, will adjust for treatment, covariates (listed above) and baseline inflammatory biomarker value at as a covariate, with visit as the repeated factor.

- The model will make no further assumptions about the correlations between a subject's value (the correlation matrix for within-subject errors will be unstructured).
- The repeated measures analysis will assume that the treatment difference can vary between visits (ie. a treatment\*visit interaction will be included in the model), and separate estimates and 95% confidence intervals will be produced at each visit. The model will also assume that the effect of baseline value for the endpoint can vary between visits (i.e. baseline value\*visit interaction will be included in the model).
- Interactions between treatment and each of the covariates will not be assessed.

## **Model Checking & Diagnostics**

Refer to Section 13.13: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- Adjusted least squares means and corresponding standard errors (SEs) of adjusted least squares means will be presented for each treatment, together with estimated treatment difference (DTG + 3TC – TBR) and corresponding 95% confidence interval and p-value.
- Note: For biomarkers that are not normally distributed, the geometric mean and a 95% CI of geometric mean will be presented for each treatment, as well as geometric mean ratios and corresponding 95% CI and a p-value.

## Sensitivity Analyses

 Not applicable Line plots of LS means with 95% confidence intervals for Adjusted Mean Change from Baseline will be generated for each treatment group by visit

## Subgroup Analyses

Not applicable

#### **Statistical Analyses**

#### **Endpoints**

 Change from baseline in HOMA-IR at Weeks 48, 96 and 144 (refer to Section 13.6.4 for details of derivation)

#### **Covariates & Factors**

- Baseline 3<sup>rd</sup> Line Agent
- CD4+ cell count (continuous)
- Age (continuous)
- Sex (Female vs. Male)
- Race (White, Black or African American, Asian, Other)
- BMI (continuous)
- Hypertension (Yes vs no)

#### Data Handling

• No multiple imputation techniques will be used to deal with the missing data.

- If change in HOMA-IR is not normally distributed the data will be log transformed and geometric means will replace arithmetic means, a 95% CI will replace the standard deviations and mean changes from baseline will be presented as geometric mean ratios.
- Change from baseline will be analysed for HOMA-IR for the comparison between DTG + 3TC and TBR.

- Using OC dataset, the Mixed Model Repeated Measures (MMRM), using the observed margins (OM) option, will adjust for treatment, covariates (listed above) and baseline HOMA-IR value at as a covariate, with visit as the repeated factor.
- The model will make no further assumptions about the correlations between a subject's value (the correlation matrix for within-subject errors will be unstructured).
- The repeated measures analysis will assume that the treatment difference can vary between visits (ie. a treatment\*visit interaction will be included in the model), and separate estimates and 95% confidence intervals will be produced at each visit. The model will also assume that the effect of baseline value for the endpoint can vary between visits (i.e. baseline value\*visit interaction will be included in the model).
- Interactions between treatment and each of the covariates will not be assessed.

## **Model Checking & Diagnostics**

Refer to Section 13.13: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- Adjusted least squares means and corresponding standard errors (SEs) of adjusted least squares means will be presented for each treatment, together with estimated treatment difference (DTG + 3TC-TBR) and corresponding 95% confidence interval and p-value.
- Note: If change from baseline in HOMA-IR data are not normally distributed, the geometric mean and a 95% CI of geometric mean will be presented for each treatment, as well as geometric mean ratios and corresponding 95% CI and a p-value.

## Sensitivity and Supportive Analyses

- Line plots of LS means with 95% confidence intervals for Adjusted Mean Change from Baseline will be generated for each treatment group by visit
- A logistic regression model will be performed on the proportion of subjects with HOMA-IR >= 2 at Week 96 adjusting for the same covariates as specified in the MMRM analysis (without visit or interaction terms). Odds ratios, standard errors, confidence intervals and p-values will be presented for all covariates specified in the model. Odds ratios for CD4+, age and BMI will be presented on the 100 cells,10-years and unit incremental scale respectively. This analysis will be repeated on the proportion of subjects with HOMA-IR>=2 at Week 144. Upon delivery of data, an assessment regarding the amount of missing data will be made. If it's considered the amount of missing HOMA-IR outcome data at Week 96 as a result of COVID-19 is substantial, the logistic regression analysis may not be performed.

## Subgroup Analyses

Not applicable

#### **Statistical Analyses**

### **Endpoints**

 Change from baseline in fasting lipids (Total Cholesterol, HDL, LDL, Triglycerides and Total Cholesterol/HDL ratio) at Week 96 and 144

#### **Covariates & Factors**

- Baseline 3<sup>rd</sup> Line Agent
- CD4+ cell count (continuous)
- Age (continuous)
- Race (White, Black or African American, Asian, Other)

BMI (continuous)

## **Data Handling**

• No multiple imputation techniques will be used to deal with the missing data.

## **Model Specification**

- Provided assumptions are satisfied, lipid data will be log transformed and geometric mean ratios with 95% Cls will be presented. Mean changes from baseline will be presented as geometric mean ratios.
- Change from baseline will be analysed for each lipid for the comparison between DTG + 3TC and TBR.
- Using OC dataset, the Mixed Model Repeated Measures (MMRM), using the observed margins (OM) option, will adjust for treatment, covariates (listed above) and baseline fasted lipid value at as a covariate, with visit as the repeated factor.
- The model will make no further assumptions about the correlations between a subject's value (the correlation matrix for within-subject errors will be unstructured).
- The repeated measures analysis will assume that the treatment difference can vary between visits (ie. a treatment\*visit interaction will be included in the model), and separate estimates and 95% confidence intervals will be produced at each visit. The model will also assume that the effect of baseline value for the endpoint can vary between visits (i.e. baseline value\*visit interaction will be included in the model).
- Interactions between treatment and each of the covariates will not be assessed.
- Lipid parameters only summarised on fasting data. Lipid parameter data collected after the
  introduction of a lipid-modifying agent are censored and an LOCF method applied such that
  the last available fasted, on-treatment lipid value prior to the initiation of a lipid-lowering
  agent is used in place of future, observed values. Subjects on lipid-lowering agents at
  baseline are excluded.

## **Model Checking & Diagnostics**

• Refer to Section 13.13: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

• The geometric mean and a 95% CI of geometric mean will be presented for each treatment, as well as geometric mean ratios and corresponding 95% CI and a p-value.

#### Sensitivity Analyses

• Line plots of geometric means with 95% confidence intervals for geometric mean ratio from Baseline will be generated for each treatment group by visit

#### Subgroup Analyses

Not applicable

## 8.4. Other Safety Analyses

The analyses of non-laboratory safety test results will be based on GSK Core Data Standards, unless otherwise specified. An overview of other safety analyses is presented in Table 7 and full details of the planned displays are presented in Appendix 12 Section 13.15: List of Data Displays. Note that ECGs and vital signs are only collected at screening, so will only be listed.

Table 7 Overview of Other Safety Analyses

| Endpoint | | Abso | olute | | Change from Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Sumi | mary | Indi | vidual | Sum | mary | Indiv | idual | | ats<br>Iysis |
| | T | F | F | L | T | F | F | L | T | F |
| Other | | | | | | | | | | |
| ECG at screening | | | | Υ | | | | | | |
| Vital Signs | | | | Υ | | | | | | |
| Liver Assessment | <b>Y</b> [7] | | | Υ | | | | | | |
| Hepatobiliary<br>Abnormality criteria | <b>Y</b> [3, 4]<br>[7] | | | <b>Y</b> [3, 4] | | | | | | |
| eC-SSRS | <b>Y</b> [7] | | | <b>Y</b> [1] | | | | | | |
| Subjects who became<br>Pregnant | | | | Υ | | | | | | |
| Patient Profiles | | | | <b>Y</b> [2] | | | | | | |
| Weight, by visit | Υ | | | | <b>Y</b> [7,8] | | | | Υ | Υ |
| BMI, by visit | Υ | | | | <b>Y</b> [7,8] | | | | Υ | Υ |
| BMI category shifts from baseline | | | | | Y | | | | | |
| Waist to height ratio at Week 144 | <b>Y</b> [7] | | | | <b>Y</b> [9] | | | | | |
| Waist to hip ratio at<br>Week 144 | <b>Y</b> [7] | | | | <b>Y</b> [9] | | | | | |
| Proportion of subjects with Metabolic syndrome at Week 144 <sup>[5]</sup> | <b>Y</b> [7] | | | | | | | | | |
| Framingham Risk Score at Week 144 <sup>[6]</sup> | | | | | Υ[7] | | | | | |
| SBP and DBP at week<br>144 | | | | | <b>Y</b> [7,8] | | | | | |

- 1. Includes Baseline and lists all visits for a subject who reports any ideation or behaviour at any visit.
- 2. Patient profiles for subjects meeting protocol defined liver stopping criteria and for patients with virologic failure. Patient profiles can also be provided for any other subjects.
- 3. All post-baseline abnormalities meeting Hepatobiliary Abnormality Criteria.
- 4. Repeat for the Early + Late Switch Phase for the DTG+3TC arm and for the Late Phase for the TBR arm (Late Phase outputs to be included in an amendment of the RAP).
- 5. See Section 13.6.4 for more details on Metabolic syndrome derivation.
- 6. See Section 13.6.2 for more details on Framingham Risk Score
- 7. Repeat for the Early + Late Switch Phase for the DTG + 3TC armand for the Late Phase for the TBR armat Week 196
- 8. Week 200 data to be included
- 9. For Late Switch Phase only

#### **Endpoints**

• Change from baseline in weight (kg) and BMI (kg/m2) at Weeks 24, 48, 96 and 144

#### **Covariates & Factors**

- Baseline 3<sup>rd</sup> Line Agent
- CD4+ cell count (continuous)
- Age (continuous)
- Sex (Female vs. Male)
- Race (White, Black or African American, Asian, Other)
- Prior TAF duration (Continuous)
- Region (North America, Europe, Asia/Australia)

## Data Handling

• No multiple imputation techniques will be used to deal with the missing data.

## **Model Specification**

- If the change from baseline in weight (BMI for BMI analysis) is not normally distributed, the
  data will be log transformed and geometric means will replace arithmetic means, a 95% CI
  will replace the standard deviations and mean changes from baseline will be presented as
  geometric mean ratios.
- Change from baseline will be analysed for the comparison between DTG + 3TC and TBR.
- Using OC dataset, the Mixed Model Repeated Measures (MMRM), using the observed margins (OM) option, will adjust for treatment, covariates (listed above) and baseline weight (BMI for BMI analysis) value as a covariate, with visit as the repeated factor.
- The model will make no further assumptions about the correlations between a subject's weight (BMI for BMI analysis) (the correlation matrix for within-subject errors will be unstructured).
- The repeated measures analysis will assume that the treatment difference can vary between visits (i.e. a treatment\*visit interaction will be included in the model), and separate estimates and 95% confidence intervals will be produced at each visit. The model will also assume that the effect of baseline weight (BMI for BMI analysis) can vary between visits (i.e. baseline value\*visit interaction will be included in the model).
- Interactions between treatment and each of the covariates will not be assessed.

#### Model Checking & Diagnostics

Refer to Section 13.13: Model Checking and Diagnostics for Statistical Analyses.

#### Model Results Presentation

- Adjusted least squares means and corresponding standard errors (SEs) of adjusted least squares means will be presented for each treatment, together with estimated treatment difference (DTG + 3TC – TBR) and corresponding 95% confidence interval.
- Note: If change in weight is not normally distributed, the geometric mean and a 95% CI of geometric mean will be presented for each treatment, as well as geometric mean ratios and corresponding 95% CI and p-values.

## **Sensitivity Analyses**

 Line plots of LS means with 95% confidence intervals for Adjusted Mean Change from Baseline will be generated for each treatment group by visit.

## **Subgroup Analyses**

Subgroup analysis (including summarytable and figure) will be performed for change from baseline in weight by BMI category(underweight/normal, overweight, obese).
 Analysis will be performed as described above and will adjust for the covariates listed above, treatment, visit, BMI subgroup category, treatment\*visit interaction, treatment\*subgroup, subgroup\*visit, treatment\*subgroup\*visit interaction terms with visit as the repeated factor regardless of their significance. Exclude Baseline Weight (continuous) from the model to avoid collinearity with Baseline BMI Category.

## 9. OTHER STATISTICAL ANALYSES

#### 9.1. Health Outcomes

## 9.1.1. Overview of Planned Analyses

The Health Outcomes analyses will be based on the Intent-To-Treat (Exposed) population, unless otherwise specified.

Full details of data displays being presented in Section 13.15: List of Data Displays.

## 9.1.2. Planned Health Outcomes Statistical Analysis

#### Statistical Analyses

#### Endpoint(s)

- Change from baseline in EQ-5D-5L Utility Score at Weeks 24, 48, 96 and 144
- Change from baseline in EQ Visual Analogue Scale (VAS) at Weeks 24, 48, 96 and 144

#### **Covariates & Factors**

Baseline 3<sup>rd</sup> Line Agent

#### Data Handling

LOCF dataset will be used.

- If HO endpoints will not be normally distributed then, the data will be log transformed and geometric means will replace arithmetic means, a 95% CI will replace the standard deviations and mean changes from baseline will be presented as geometric mean ratios.
- Any missing values should be imputed using LOCF. In the last observation carried forward (LOCF) dataset missing values will be carried forward from the previous, non-missing available On-treatment assessment from the same dimension. This technique will be applied for all missing values, regardless if the subject discontinued the treatment. Missing total values can then be calculated using a combination of present and carried forward individual items.
- With LOCF dataset, Mixed Model Repeated Measures (MMRM), using the observed margins (OM) option, will adjust for treatment, covariates (listed above) and baseline EQ-5D-5L value as a covariate, with visit as the repeated factor.
- The repeated measures analysis will assume that the treatment difference can vary between visits (ie. a treatment\*visit interaction will be included in the model), and separates estimates and 95% confidence intervals will be produced at each visit. The model will also assume that the effect of baseline score for the endpoint can vary between visits (ie. baseline score\*visit interaction will be included in the model).

• The model will make no further assumptions about the correlations between a subject's score (the correlation matrix for within-subject errors will be unstructured).

#### **Model Results Presentation**

- Adjusted means and corresponding standard errors (SEs) of adjusted means will be presented for each treatment by visit, together with estimated treatment difference (DTG + 3TC – TBR) and corresponding 95% confidence interval and p-value.
- Figures showing the adjusted mean change from baseline with 95% Cls for each treatment group across visits in EQ-5D-5L Utility Score and EQ Visual Analogue scale.
- Figures to show the differences for subjects treated with DTG + 3TC compared to TBR in adjusted mean change from baseline with 95% Cls in Utility Score and Visual Analog Scale at each visit.

## 9.2. Virology

## 9.2.1. Overview of Planned Analyses

## 9.2.2. Planned Virology Statistical Analysis

The virology analyses of genotype and phenotype data will be based on the CVW and pPVW resistance populations (and LS-CVW, LS-pPVW, LS-populations, LS-Virologic Genotypic and LS-Virologic Phenotypic populations where applicable). Please see Section 13.6.3 for details of the derivation of CVW. Please see Section 4 for details of the derivation of pPVW.

The CVW population will be based on subjects who have experienced a CVW at any point. Summary tables will present CVWs at the time point of the SVW (or first elevation if this was >=50 c/mL and <200 c/mL). Listings will present CVWs occurring at any point, and within the analysis visit in which the CVW date occurred. CVWs must be confirmed within the phase in which they are reported. Full details of data displays being presented in Appendix 15: List of Data Displays.

Table 8 provides an overview of the planned virology analyses, with full details of data displays being presented in Section 13.15: List of Data Displays.

Reisistance testing will also be performed on any participant with a last on-treatment plasma HIV-1 RNA >=400 c/mL.

Table 8 Overview of Planned Virology Analyses

| Endpoint | | Abso | olute | |
|---|---|---|---|---|
| | Sumr | mary | Indivi | dual |
| | Т | F | F | L |
| Genotypic resistance | | | | |
| Incidence of genotype at time of CW[1] | <b>Y</b> [2,6] | | | <b>Y</b> [4] |
| Phenotypic resistance <sup>[5]</sup> | | | | |
| Incidence of phenotype at time of CWI1] | <b>Y</b> [3,6] | | | <b>Y</b> [4] |
| INI replication capacity at time of CWI1] | | | | <b>Y</b> [4] |
| Fold Change at CVW | <b>Y</b> [6] | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- Sample used for resistance testing is taken at the time suspected virologic withdrawal criteria are met, and only
  tested once a subject confirms virologic failure at a subsequent visit. Occasionally, if the viral load sample of
  SVW timepoint is below the assay cut-off (<400 c/mL), resistance testing using CVW timepoint sample may be
  attemped.</li>
- 2. Separate outputs for INI and NRTI/NNRTI/PI mutations
- 3. Separate outputs by phenotypic cut-off and by number of drugs to which subjects are resistant.
- 4. Produce for CVW and pPVW resistance population (athough not for pPVW populations for Week 96 or Week 144).
- 5. Phenotypic data are not generated for Baseline using proviral -DNA GenoSure Archive assay
- 6. Repeatfor the Early + Late Switch Phase for the DTG+3TC arm and for the Late Phase for the TBR arm at Week 196

## 10. PHARMACOKINETIC ANALYSES

Pharmacokinetic analyses are not applicable to analyses post Week 48.

Steady state plasma PK parameters of DTG and 3TC will be assessed using intensive PK collected at week 4 in a sub-set of subjects. PK concentrations summaries for intense and Sparse PK will be performed.

## 10.1. Pharmacokinetic Analyses

## 10.1.1. Endpoint / Variables

#### 10.1.1.1. Drug Concentration Measures

All PK concentration listing displays will be based on the Intensive and Sparse Pharmacokinetic populations. Concentrations of DTG and 3TC in plasma will be listed and summarized according to GSK standards, where applicable (Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 13.5.3 Reporting Standards for Pharmacokinetic)).

DTG and 3TC concentration listings for the intensive PK population will be sorted by subject and time relative to dose, noting the study visit; summaries will be presented by study visit and time relative to dose.

DTG and 3TC concentration listings for the sparse PK population will be sorted by subject, study visit and time (or sampling window) relative to dose; summaries will be presented by study visit and time (or sampling window) for weeks 4, 24, 36, and 48 and by sampling window for weeks 8 and 12. Patient profiles refer to a collection samples collected sequentially with regard to the dosing schedule for the intensive PK population. Please refer to Section 13.3.2 for definitions of assessment windows for inclusion of PK concentrations in summary statistics. Please refer to Section 13.6.10 for rules around data derivation and imputation. Please refer to Section 13.6.5 for rules regarding exclusions for the intensive and sparse PK populations. Please refer to the protocol for more information regarding the sparse and intensive populations and dosing schedules.

# 10.1.1.2. Derived Pharmacokinetic Parameters for subjects participating in the intense PK sub-study

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin 5.3 or higher. All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| Cmax | 3TC and DTG maximum observed plasma concentration, determined directly from the concentration-time data |
| tmax | 3T C and DTG time to reach Cmax, determined directly from the concentration-time data |
| Сτ | 3TC and DTG observed plasma concentration at the end of the dosing interval, determined directly from the concentration-time data |

| Parameter | Parameter Description |
|---|---|
| C0 | 3TC and DTG observed pre-dose plasma concentration, determined directly from the concentration-time data |
| AUC(0-τ) | 3TC and DTG area under the concentration-time curve in one dosing interval |

## 10.1.2. Summary Measure

Not applicable.

## 10.1.3. Population of Interest

The primary pharmacokinetic analyses will be based on the Sparse and Intensive Pharmacokinetic Populations population, unless otherwise specified.

## 10.1.4. Strategy for Intercurrent (Post-Randomisation) Events

Not applicable.

## 10.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 15: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 10.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

Table 9 provides an overview of the planned analyses, with full details being presented in Appendix 15: List of Data Displays.

Table 9 Overview of Planned Pharmacokinetic Analyses

| | | | Untr | ansfor | med | | | Lo | g-Tran | sforme | d |
|---|---|---|---|---|---|---|---|---|---|---|---|
| End Point | Sta | ts Anal | ysis | Sum | Summary | | Individual | | Summary | | Individual |
| | T | F | L | T | F | F | L | Т | F | F | L |
| Intensive PK Cor | ncentra | ations | | | | | | | | | |
| Plasma 3TC | | | | Υ | Υ | Υ | Υ | Υ | Υ | | |
| Concentrations | | | | ı | ı | ı | ı | | | | |
| Plasma DT G | | | | Υ | Υ | Υ | Υ | Υ | Υ | | |
| Concentrations | | | | ı | ı | • | ı | • | ' | | |
| Sparse PK Conc | Sparse PK Concentrations | | | | | | | | | | |
| Plasma 3T C | | | | | | | | | | | |
| Concentrations | | | | | | | | | | | |
| by Visit and | | | | Υ | Υ | | Υ | | | | |
| sampling | | | | | | | | | | | |
| window | | | | | | | | | | | |
| Plasma DTG | | | | | | | | | | | |
| Concentrations | | | | Υ | Υ | | Υ | | | | |
| by Visit and | | | | | | | | | | | |

| | | | Untr | ansfor | med | | | Lo | g-Tran | sforme | d |
|---|---|---|---|---|---|---|---|---|---|---|---|
| End Point | Stats Analysis T F L | | | Sum | mary | Indivi | dual | Sum | mary | Indivi | dual |
| | T | F | L | T | F | F | L | T | F | F | L |
| sampling<br>window | | | | | | | | | | | |
| Intensive PK Para | ameter | 'S | | | | | | | | | |
| Plasma 3T C<br>Parameters | | | | Y | | | Y | Y | | | |
| Plasma DT G<br>Parameters | | | | Y | | | Y | Y | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- 1. Individual = Represents FL related to any displays of individual subject observed raw data.

# 11. POPULATION PHARMACOKINETIC (POPPK) ANALYSES

Population PK analyses are not applicable to analyses post Week 48.

If data permits, the sparse concentrations of 3TC and DTG collected at weeks 4, 8, 12, 24, 36 and 48 will be pooled with the intensive PK concentrations and potentially data from other studies to perform integrated PK analyses for DTG and 3TC. The primary goal of this analysis is to characterize the population pharmacokinetics of 3TC and DTG administered as a dual regimen maintenance treatment for HIV in participants who are virologically suppressed. The influence of subject demographics, baseline characteristics, including disease activity, and co-medication on the pharmacokinetics of 3TC and DTG in this population will be investigated. The individual subject PK parameters will be estimated and documented for the purposes of any subsequent exposure response (PK/PD) analyses. The PopPK analyses for DTG and 3TC will be performed under a separate RAP and will be reported separately.

Further details to be included in a separate RAP.

## 12. REFERENCES

D'Agostino R.B., Vasan R.S., Pencina M.J., Wolf P.A., Cobain M., Massaro J.M. Kannel W.B. General Cardiovascular Risk Profile for Use in Primary Care: The Framingham Heart Study. Epidemiology. 2008; 117:743-753.

Devlin N., Shah K., Feng Y., Mulhern B, Hout VB. Valuing Health-Related Quality of Life: An EQ-5D-5L Value Set for England. Office of Health Economics, 2016

Fleiss J.L. Statistical Methods for Rates and Proportions. 2nd ed. New York: John Wiley; 1981.

Grundy S.M., et al. Executive summary of the third report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). JAMA. 2001;285

Johnson VA, Calvez V, Gunthard HF, et. al. Special Contribution. Update of the Drug Resistance Mutations in HIV-1: March 2013. IAS-USA Topics in Antiviral Medicine. Available at: https://www.iasusa.org/sites/default/files/tam/21-1-6.pdf. Accessed Octover 24, 2016.

Kalbfleisch J.D., Prentice R.L. The Statistical Analysis of Failure Time Data. 1st ed. New York: John Wiley & Sons; 1980.

Klingenberg. A new and improved confidence interval for the Mantel-Haenszel risk difference. *Statistics in Medicine*. 2014; 2968-2983.

Levey A.S., Stevens L.A., Schmid C.H., Zhang Y.L., Castro A.F. 3rd, Feldman H.I., Kusek J.W., Eggers P., Van Lente F., Greene T., Coresh J. CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration). A New Equation to Estimate Glomerular Filtration Rate. *Ann Intern Med* 2009;150(9):604-612.

Liu TF, Shafer RW. Web Resources for HIV type 1 Genotypic-Resistance Test Interpretation. Clin Infect Dis. 2006;42 (11):1608-1618.

Lui K.J., Kelly C. A Revisit on Tests for Homogeneity of the Risk Difference, *Biometrics*, 2000;56:309-315.

Miettinen O, Nurminen M. Comparative Analysis of two rates. *Statistics in Medicine*. 1985; 4:213-226.

Ralph B. D'Agostino, Ramachandran S. Vasan, Michael J. Pencina, Philip A. Wolf, Mark Cobain, Joseph M. Massaro, William B. Kannel. 2008. General Cardiovascular Risk Profile for Use in Primary Care (The Framingham Heart Study). *Circulation* 2008; 117: 743-753.

Sato T. On the variance estimator for the Mantel-Haenszel risk difference. *Biometrics*. 1989;42:311-323.

# 13. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 4 : Ar | nalysis Populations |
| Section 13.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| RAP Section 5 : Go | eneral Considerations for Data Analyses & Data Handling Conventions |
| Section 13.2 | Appendix 2: Schedule of Activities |
| Section 13.3 | Appendix 3: Assessment Windows |
| Section 13.4 | Appendix 4: Study Phases and Emergent Adverse Events |
| Section 13.5 | <ul> <li>Appendix 5: Data Display Standards &amp; Handling Conventions</li> <li>Study Treatment &amp; Sub-group Display Descriptors</li> <li>Baseline Definitions &amp; Derivations</li> <li>Reporting Process &amp; Standards</li> </ul> |
| Section 13.6 | Appendix 6: Derived and Transformed Data |
| Section 13.7 | Appendix 7: Reporting Standards for Missing Data Premature Withdrawals Handling of Missing Data Handling of Missing and Partial Dates |
| Section 13.8 | Appendix 8: Values of Potential Clinical Importance |
| Section 13.9 | Appendix 9: Population Pharmacokinetic (PopPK) Analyses |
| Section 13.10 | Appendix 10: Time to Event Details |
| Section 13.11 | Appendix 11: Snapshot |
| Other RAP Appen | dices |
| Section 13.12 | Appendix 12: Abbreviations & Trade Marks |
| Section 13.13 | Appendix 13: Model Checking and Diagnostics for Statistical Analyses |
| Section 13.14 | Appendix 14: COVID-19 Modified Analyses and Supportive Sensitivity Analyses |
| Section 13.15 | Appendix 15: List of Data Displays |
| Section 13.16 | Appendix 16: Example Mock Shells for Data Displays |

# 13.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

## 13.1.1. Exclusions from Per Protocol Population

A subject meeting any of the following criteria (Significant Protocol Deviations) will be excluded from the Per Protocol population:

| Number | Exclusion Description |
|---|---|
| | Subject deviates from any inclusion or |
| 01 | exclusion criteria, as recorded in the eCRF |
| 02* | Subject took/received incorrect IP, i.e., other than the one to which they were randomised for greater than 10% of the total time On-treatment |
| 03* | Interruption of IP for greater than 10% of the total time On-treatment, for reasons other than treatment-related adverse events/laboratory abnormalities, based on eCRF IP exposure forms or eCRF CONART forms in case commercial supply is used before study completion. |
| 04 | HIV immunotherapeutic vaccines used |
| 05 | Concurrent use of drugs that may decrease DTG concentration for >7 days: (Carbamazepine, Oxcarbazepine, Phenobarbital, Phenytoin, St. John's wort (Hypericum perforatum), rifampin |
| 06 | Concomitant use of rifapentine |
| 07 | Other experimental agents, antiretroviral drugs not otherwise specified in the protocol, cytotoxic chemotherapy, or radiation therapy used |
| 08 | Systemically administered immunomodulators used through Week 144 visit |
| 09 | HCV therapy based on interferon or any other medications that have a potential for adverse drug-drug interactions with study treatment |
| 10 | Concomitant use of acetaminophen in subjects with acute viral hepatitis |

| Number | Exclusion Description |
|---|---|
| 11 | Dofetilide or pilsicainide used concurrently with DTG |
| 12 | Subject's change (i.e., substitution or dose modification) of DTG, 3TC or component of TBR (except protocol allowed switches, e.g. switch of booster) but was not withdrawn from the study |
| 13 | Subject became pregnant while on study |
| 14 | Permanent discontinuation of IP/withdrawal due to a reason of "Protocol Deviation" (as recorded in the eCRF) |

<sup>\*</sup>Programmatically derived protocol deviations, which are defined in a separate protocol deviations specification document.

Please refer to Section 13.6.9 regarding cut-off dates regarding protocol deviations leading to exclusion from the per protocol set.

# 13.2. Appendix 2: Protocol Defined Schedule of Activities

# 13.2.1. Early Switch Phase Time and Events Table (Screening to Week 148)

| Procedures | /isita | | | | | | Ор | en-lal | el Rai | ndomi | sed Ea | rly Sw | vitch Phase | | | | Switch<br>Visit | al | p <sub>d</sub> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | _<br>V gι | e/ | | | | | | | | | | Wee | k | | | | | Iraw | ln-w |
| | Screening Visita | Baseline/<br>Day 1 | 4 | 8 | 12 | 24 | 36 | 48 | 60 | 72 | 84 | 96 | 108<br>(optional) <sup>b</sup> | 120 | 132<br>(optional) <sup>b</sup> | 144 | 148° | Withdrawal | Follow-up <sup>d</sup> |
| Clinical and Other Asse | essmen | ts | | | | | | | | | | | | | | | | | |
| Written informed consent | Х | | | | | | | | | | | | | | | | | | |
| Inclusion/Exclusion criteriae | Х | Х | | | | | | | | | | | | | | | | | |
| Demography | Χ | | | | | | | | | | | | | | | | | | |
| Prior ART history | Χ | | | | | | | | | | | | | | | | | | |
| Medical history <sup>f</sup> | Χ | | | | | | | | | | | | | | | | | | |
| Currentmedical conditions | Х | | | | | | | | | | | | | | | | | | |
| Cardiovascularrisk<br>assessment, including<br>vital signs | Х | | | | | | | | | | | | | | | | | | |
| Vital Signs: Resting<br>Blood pressure (see<br>Section 7.4.4 and<br>Appendix 10 of<br>Protocol) | | | | | | | | | | | | | | | | Х | Х | Х | |
| Body Weight (BMI will<br>be calculated within the<br>eCRF) | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |

| Procedures | isita | | | | | | Ор | en-lal | bel Ra | ndomi | sed Ea | rly S w | vitch Phase | | | | Switch<br>Visit | al | P0 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | νgι | / e | | | | | | | | | | Wee | k | | | | | raw | h-v |
| | Screening Visit | Baseline/<br>Day 1 | 4 | 8 | 12 | 24 | 36 | 48 | 60 | 72 | 84 | 96 | 108<br>(optional)♭ | 120 | 132<br>(optional) <sup>b</sup> | 144 | 148° | Withdrawal | Follow-up <sup>d</sup> |
| Vital Signs: Hip and<br>waist circumference<br>(see Section 7.4.4 and<br>Appendix 10 of<br>Protocol) | | | | | | | | | | | | | | | | Х | | | |
| HIV risk factors and mode of transmission | | Х | | | | | | | | | | | | | | | | | |
| CDC HIV-1 classification | Χ | Х | | | | | | | | | | | | | | | | | |
| HIV associated conditions | | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Χ | Х | Χ | |
| Columbia Suicidality<br>Severity Rating Scale | | Xh | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Χ | Х | Χ | Х | Χ | | Χ | |
| Concomitant medication | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Χ | Х | Χ | Х |
| Symptom Directed<br>Physical Exam | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Χ | | Χ | Х |
| 12-lead ECG | Χ | | | | | | | | | | | | | | | | | | |
| Adverse events | | Х | Χ | Χ | Χ | Х | Х | Χ | Х | Х | Х | Χ | Х | Χ | Х | Χ | Х | Χ | Х |
| Serious adverse events | Xk | Х | Χ | Χ | Χ | Х | Х | Χ | Х | Х | Х | Χ | Χ | Х | Х | Χ | Х | Χ | Χ |
| Willingness to Switch <sup>i</sup> | | ΧI | | | | | | | | | | | | | | | | | |
| EQ-5D-5 <sup>m</sup> | | Х | Χ | | | Х | | Χ | | | | Χ | | | | Χ | | Χ | |
| Laboratory Assessmen | ts | | | | | | | | | | | | | | | | | | |
| Quantitative plasma<br>HIV-1 RNA <sup>n</sup> | Χ | Х | Х | Х | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Χ | Х | Χ | | Χ | |

| Procedures | isita | | | | | | Ор | en-lal | oel Ra | ndomi | sed Ea | rly Sw | ritch Phase | | | | Switch<br>Visit | a | p <b>o</b> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | ν g r | <i>)</i> 6 | | | | | | | | | | Wee | k | | | | | raw | yu-√ |
| | Screening Visit | Baseline /<br>Day 1 | 4 | 8 | 12 | 24 | 36 | 48 | 60 | 72 | 84 | 96 | 108<br>(optional)♭ | 120 | 132<br>(optional) <sup>b</sup> | 144 | 148° | Withdrawal | Follow-up⁴ |
| Lymphocyte subset<br>(CD4+ at all visits and<br>CD8+ at Baseline, and<br>Weeks 24, 48, 96, 144<br>and 196 only) | X | Х | Х | Х | X | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | х | | Х | |
| Plasma for storage <sup>o</sup> | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | X | Χ | X | Χ | | Χ | |
| Clinical chemistry | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | X | Χ | X | Χ | | Χ | Χ |
| Hematology | Χ | Χ | Χ | Х | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Χ | X | Χ | | Χ | Χ |
| PT/INR | Χ | | | | | | | | | | | | | | | | | | |
| Fasting lipids and glucose <sup>p</sup> | | Χ | | | | Х | | Х | | | | Х | | | | Х | | Χq | |
| Urinalysis and spot<br>urine for protein<br>analysis <sup>r</sup> | | Х | | | | Х | | Χ | | | | Х | | | | Х | | Χ | Х |
| Pregnancy tests,t,u | S | U/S <sup>v</sup> | S | S | S | S | S | S | S | S | S | S | S | S | S | S | U | S | |
| HbsAg, anti-HBc, anti-<br>HBs, and HBV DNA <sup>w</sup> | Х | | | | | | | | | | | | | | | | | | |
| HCV antibody | Χ | | | | | | | | | | | | | | | | | | |
| RPR | Χ | | | | | | | | | | | | | | | | | | |
| Insulin, HbA1c and renal, and bone marker analytes (blood/urine)x | | Х | | | | Х | | Х | | | | Х | | | | Х | | Хq | |
| Whole Blood (Virology)y | | Х | | | | | | Χ | | | | Χ | | | | Χ | | Χ | |
| Whole Blood (Telomere length) <sup>z</sup> | | Χ | | | | | | Χ | | | | Χ | | | | Х | | Хаа | |
| Cryopreserved<br>PBMCsbb | | Χ | | | | | | Χ | | | | Х | | | | Х | | Xaa | |

| Procedures | /isita | | | | | | Ор | en-lal | oel Ra | ndomi | sed Ea | rly Sw | ritch Phase | | | | Switch<br>Visit | al | ρ <b>d</b> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | J g ( | ) e | | | | | | | | | | Wee | k | | | | | raw | n-v |
| | Screening Visit | Baseline /<br>Day 1 | 4 | 8 | 12 | 24 | 36 | 48 | 60 | 72 | 84 | 96 | 108<br>(optional) <sup>b</sup> | 120 | 132<br>(optional) <sup>b</sup> | 144 | 148° | Withdrawal | Follow-up <sup>d</sup> |
| Inflammation<br>biomarkers (Blood)∞ | | Χ | | | | | | Χ | | | | Х | | | | Χ | | Xaa | |
| Study Treatment | | | | | | | | | | | | | | | | | | | |
| IVRS/IWRS <sup>dd</sup> | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Χ | Х | Χ | Χ | Χ | Χ |
| Dispense study treatment | | Χ | Χ | Х | Χ | Χ | Χ | Χ | Χ | Х | Χ | Х | | Х | | Χ | Х | | |
| Study treatment accountability (pill counts) | | | Х | Х | Х | Х | Χ | Χ | Х | Х | Χ | Х | | Х | | Х | | Х | |
| Pharmacokineticee | | | | | | | | | | | | | | | | | | | |
| Intensive PK sample collection at selected sites for subset of ~30 subjects (Fasting)ee | | | Xff | | | | | | | | | | | | | | | | |
| Dispense PK Diary<br>Card to intensive PK<br>sub-set | | Х | | | | | | | | | | | | | | | | | |
| Sparse PK sample collectionee | | | <b>X</b> 99 | Χ | Χ | Χ | Χ | Χ | | | | | | | | | | | |
| Dispense PK Diary Card to Sparse PK subjects anti-HRc = antibody to be | | Χ | Χ | Х | Χ | Χ | Χ | | | | | | | | | | | | |

anti-HBc = antibody to hepatitis B core antigen, anti-HBs = hepatitis B surface antibody, ART = antiretroviral therapy, CDC = Centers for Disease Control and Prevention, DNA = deoxyribonucleic acid, HbA1c = Glycated hemoglobin, HBsAg = hepatitis B surface antigen, HCV = hepatitis C virus, HIV-1 = human immunodeficiency virus type 1, IVRS = interactive voice recognition system, IWRS = interactive web recognition system, PBMC = peripheral blood mononuclear cell, RNA = ribonucleic acid, RPR = rapid plasma reagin

## 13.2.2. Late Switch Phase Time and Events Table: TBR subjects who switched to DTG + 3TC at Week 148

TBR subjects switching at Week 148 are followed up at 4, 12 and 24 weeks post-switch after which 24 weekly visits are resumed.

| Procedures | | Late | Switch Pha | se through End o<br>Week | ofStudy | | Continuation Phase | wal | 효 |
|---|---|---|---|---|---|---|---|---|---|
| | 152 | 160 | 172 | 184<br>(optional) <sup>b</sup> | 196 | 200 <sup>hh</sup> | Every 24 weeks after Week 200bj | Withdrawal | Follow-up |
| Clinical and Other Assessments | | | | <u> </u> | | l | | | |
| Vital Signs: Resting Blood pressure (see Section 7.4.4 and Appendix 10 of Protocol) | | | Х | | Х | Х | | Х | |
| Body Weight (BMI will be calculated within the eCRF) | Х | Х | Х | Х | Χ | Х | X | Х | Х |
| Vital Signs: Hip and waist circumference (see Section 7.4.4 and Appendix 10 of Protocol) | | | Х | | Х | | | Х | |
| HIV associated conditions | Χ | Х | Χ | Х | Χ | Х | X | Χ | |
| Columbia Suicidality Severity Rating Scale | Χ | Х | Χ | Х | Х | | X | Χ | |
| Concomitant medication | Χ | Х | Х | Х | Χ | Х | X | Χ | Х |
| Symptom Directed Physical Exam | Χ | Х | Х | Х | Х | Х | | Х | Х |
| Adverse events | Χ | Χ | Χ | Х | Χ | Х | X | Χ | Χ |
| Serious adverse events | Χ | Χ | Χ | Х | Χ | Х | X | Χ | Χ |
| EQ-5D-5L <sup>m</sup> | | | | | Χ | | | Χ | |
| Laboratory Assessments | | | | | | | | | |
| Quantitative plasma HIV-1 RNAn | Χ | X | Х | X | Х | | X | Χ | |
| Lymphocyte subset (CD4+ at all visits and CD8+ at Baseline, and Weeks 24, 48, 96, 144 and 196 only) | Х | Х | X | Х | Х | | | Х | |
| Plasma for storage∘ | Χ | Χ | Χ | Х | Χ | | X | Χ | |

| Procedures | | Late | Switch Pha | se through End<br>Week | ofStudy | | Continuation Phase | wal | d- |
|---|---|---|---|---|---|---|---|---|---|
| | 152 | 160 | 172 | 184<br>(optional) <sup>b</sup> | 196 | 200 <sup>hh</sup> | Every 24 weeks after Week 200bj | Withdrawal | Follow-up |
| Clinical chemistry | Χ | Х | Х | Х | Х | Х | | Х | Х |
| Hematology | Χ | Х | Х | Х | Χ | Х | | Χ | Х |
| Fasting lipids and glucose <sup>p</sup> | | | | | Х | | | Χq | |
| Urinalysis and spoturine for protein analysis <sup>r</sup> | | | | | Χ | | | Χ | Х |
| Pregnancy test <sup>s,t,u</sup> | S | S | S | S | S | S | S | S | |
| Insulin, HbA1c and renal, and<br>bone marker analytes<br>(blood/urine)× | | | | | Х | | | Χq | |
| Whole Blood (Virology) <sup>y</sup> | | | | | X | | | Χ | |
| Whole Blood (Telomere length)z | | | | | Х | | | Xaa | |
| Cryopreserved PBMCsbb | | | | | Х | | | Хаа | |
| Inflammation biomarkers<br>(Blood)∞ | | | | | Χ | | | Xaa | |
| StudyTreatment | | | | | | | | | |
| IVRS/IWRS <sup>dd</sup> | Χ | Χ | Χ | Χ | Χ | Х | X | Χ | Χ |
| Dispense study treatment | Χ | Х | Х | | Χ | | X | | |
| Study treatment accountability (pill counts) | Χ | X | Х | | Χ | Х | X | Χ | |

## 13.2.3. Late Switch Phase Time and Events Table: DTG + 3TC arm

| Procedures | | _ate Switcl | h Phase through I | End of Stud | ly | Continuation Phase | | |
|---|---|---|---|---|---|---|---|---|
| | | | Week | | T | 1 | awa | 핰 |
| | 160<br>(optional) <sup>b</sup> | 172 | 184<br>(optional) <sup>b</sup> | 196 | 200 <sup>hh</sup> | Every 24 weeks after Week 200 <sup>b,j</sup> | Withdrawal | Follow-up |
| Clinical and Other Assessments | LL | | L | | | 1 | | |
| Vital Signs: Resting Blood pressure (see<br>Section 7.4.4 and Appendix 10 of Protocol) | | Х | | Х | Х | | Х | |
| Body Weight (BMI will be calculated within the eCRF) | Х | Х | Х | Х | Х | X | Х | Х |
| Vital Signs: Hip and waist circumference (see Section 7.4.4 and Appendix 10 of Protocol) | | Х | | Х | | | Х | |
| HIV associated conditions | Х | Χ | Х | Χ | Х | X | Χ | |
| Columbia Suicidality Severity Rating Scale | Х | Χ | Х | Χ | | X | Χ | |
| Concomitant medication | Х | Χ | X | Χ | Х | X | Х | Х |
| Symptom Directed Physical Exam | Х | Χ | X | Χ | Х | | Χ | Х |
| Adverse events | Х | Χ | Х | Χ | Х | X | Χ | Х |
| Serious adverse events | Х | Χ | Х | Χ | Х | X | Χ | Х |
| EQ-5D-5L <sup>m</sup> | | | | Χ | | | Χ | |
| Laboratory Assessments | | | | | | | | |
| Quantitative plasma HIV-1 RNAn | Х | Χ | X | Χ | | X | Χ | |
| Lymphocyte subset (CD4+ at all visits and CD8+ at Baseline, and Weeks 24, 48, 96, 144 and 196 only) | Х | Χ | X | Χ | | | Χ | |
| Plasma for storage <sup>o</sup> | X | Χ | X | Χ | | X | Χ | |
| Clinical chemistry | Х | Χ | X | Χ | Х | | Χ | Х |
| Hematology | Х | Χ | X | Χ | Х | | Χ | Х |
| Fasting lipids and glucose <sup>p</sup> | | | | Χ | | | Χq | |
| Urinalysis and spoturine for protein analysis | | | | Χ | | | Χ | Х |
| Pregnancy tests,t,u | S | S | S | S | S | S | S | |
| Insulin, HbA1c and renal, and bone marker analytes (blood/urine) <sup>x</sup> | | | | Х | | | Χq | |
| Whole Blood (Virology) <sup>y</sup> | | | | Χ | | | Χ | |

| Procedures | | Late Switch | Phase through<br>Week | End of Stud | у | Continuation Phase | la | dn |
|---|---|---|---|---|---|---|---|---|
| | 160<br>(optional) <sup>b</sup> | 172 | 184<br>(optional) <sup>b</sup> | 196 | 200 <sup>hh</sup> | Every 24 weeks after Week 200 <sup>b,j</sup> | Withdrawal | Follow-u |
| Whole Blood (Telomere length)z | | | | Χ | | | Xaa | |
| Cryopreserved PBMCsbb | | | | Χ | | | Xaa | |
| Inflammation biomarkers (Blood)∞ | | | | Χ | | | Xaa | |
| StudyTreatment | | | | | | | | • |
| IVRS/IWRS <sup>dd</sup> | X | Χ | X | Χ | X | X | Χ | Х |
| Dispense study treatment | | Χ | | Χ | | X | | |
| Study treatment accountability (pill counts) | | Χ | | Χ | X | X | Χ | |

- a. As soon as all Screening results are available, randomization may occur.
- b. This optional study visit is ONLY to be conducted in countries that require visits every 3 months per standard of care.
- c. Subjects with plasma HIV-1 RNA ≥50 c/mL at Week 144 must have HIV-1 RNA level re-assessed by a second measurement performed 2-4 weeks later. Subjects should have received full doses of study treatment for at least 2 weeks at the time of HIV-1 RNA re-assessment. Subjects randomized to DTG + 3TC do not attend a Week 148 switch visit.
- d. An in-clinic Follow-Up visit will be conducted 4 weeks after the last dose of study medication for subjects with the following conditions at the last on-study visit ongoing AEs, serious adverse events (SAEs) regardless of attributability, any laboratory abnormalities considered to be AEs or potentially harmful to the subject. Only the laboratory tests necessary to evaluate the AE/SAE/laboratory abnormality should be collected.
- e. Inclusion/exclusion criteria will be assessed fully at the Screening visit. Changes between the Screening visit and the Day 1 visit should be considered to ensure eligibility, including review of additional assessments performed at Day 1. Genotypic resistance testing results MUST be provided to ViiV after screening and before randomization.
- f. Full medical history will be conducted prior to randomization and include assessments of cardiovascular, metabolic (e.g., Type I or II diabetes mellitus), psychiatric (e.g., depression), renal (e.g., nephropathy, renal failure), and bone disorders.
- g. Assessment for cardiovascular risk will include height, weight, blood pressure, smoking status and history, pertinent medical conditions (e.g., hypertension, diabetes mellitus), and family history of premature cardiovascular disease. BMI will be calculated within the eCRF.
- h. On Day 1, the electronic Columbia Suicidality Severity Rating Scale eC-SSRS, patient completed questionnaire) is to be administered prior to randomization.
- i. Limited physical examination to include blood pressure at Day 1 (recorded in eCRF) for Framingham score assessment. Blood pressure to be measured after resting in a semi-supine position for at least 5 minutes.
- j. A 12-lead ECG will be performed after resting in a semi-supine position for at least 5 minutes.
- k. Only SAEs related to study participation or to a concomitantly administered ViiV/GSK product will be collected between obtaining informed consent and administration of study drug at Day 1.
- I. Willingness to Switch Survey must be done prior to randomization.
- m. Questionnaire/Surveys are recommended to be administered at the beginning of the visit before any other assessments are conducted. Only conduct questionnaires/surveys at Withdrawal if occurring prior to Week 196.
- n. See Virologic Withdrawal and Stopping Criteria Section of protocol (Section 5.4 of Protocol).
- o. Plasma samples for storage will be collected at each visit starting at Screening, including unscheduled visits (e.g. for HIV-1 RNA levels and immunological parameters). These samples will be used when needed such as when samples are lost, arrive at the laboratory unevaluable, or for genotypic and/or phenotypic analyses when subjects meet Suspected and Confirmed Virologic Withdrawal criteria.
- p. An overnight fast is preferred; however, a minimum of a 6-hour fast is acceptable.
- g. Collect sample for these assessments ONLY if the Withdrawal visit occurs at Week 24, 48, 96, 144 or 196.
- r. A morning specimen is preferred. To assess renal biomarkers: urine albumin/creatinine ratio; urine protein/creatinine ratio; and urine phosphate.
- s. Women of childbearing potential only. S=serum, U=urine. Pregnancy events will be captured starting at Day 1 following exposure to study drug.
- t. Remind females of reproductive potential of the need to avoid pregnancy while in study and adherence to the study's contraception requirements.
- u. Beginning after Week 96, if study visits are every 24 weeks, participants who are women of child bearing potential must also do a home-based urine pregnancy test approximately every 12 weeks between study visits at approximately Weeks 108, 132, 160 and 184 and during the Continuation Phase. Site staff must contact the participants who are women of child bearing potential to remind them to complete the test and to verify and record pregnancy test results in the source documents. The site must also complete the pregnancy status eCRF if a pregnancy occurs and report the pregnancy to ViiV/GSK per Section 13.3.2 of Protocol.
- v. Local serum pregnancy test on Day 1 is allowed if it can be done, and results obtained, within 24 hours prior to randomization
- w. HBV DNA testing will be performed for subjects with positive anti-HBc and negative HBsAg and negative anti-HBs (past and/or current evidence). Subjects will have to return to the clinic to provide a sample for HBV DNA testing prior to randomisation.
- x. Blood sample for insulin, HbA1c, and renal and bone biomarker assessments: **Renal:** Cystatin C; Beta-2-Microglobulin; Retinol Binding Protein (RBP); **Bone:** bone specific alkaline phosphatase, procollagen type 1-N-propeptide, type 1 collagen cross-linked C-telopeptide, osteocalcin, 25 hydroxy-Vitamin D.
- y. Whole blood (Virology) may be used for virologic analyses as described in the protocol.
- z. Whole blood will be used for telomere length evaluation at Day 1, Week 48, Week 96, Week 144, Week 196 and at the Withdrawal visit.
- aa. Collect sample for these assessments ONLY if the Withdrawal visit occurs at Week 48, 96, 144 or 196
- bb. PBMCs will be collected, cryopreserved and stored in a subset of sites. These samples will be used for the measurement of telomerase activity.
- cc. Blood sample for inflammation biomarker assessments: IL-6, hs-CRP, d dimer, sCD14, sCD163.
- dd. At Screening, a subject number will be generated.
- ee. PK sampling in subjects from the DTG/3TC FDC armonly, as detailed in Section11 of Protocol.
- ff. Intensive PK sampling in a subset of subjects from the DTG/3TC FDC arm at select sites at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 10 and 24 hours post-dose. On the intensive PK day, patients are required to fast from 8 hours prior to dosing and then through 4 hours post-dose. Detailed in Section 11 of Protocol.
- gg. At Week 4, subjects who performed intensive PK do not perform Sparse PK sampling.
- hh. Subjects must return to the clinic for a Week 200 End of Study visit when transitioning to commercial supplies or to an alternate ART regimen, if appropriate. Do not dispense study treatment at this study completion visit unless the participant is entering the Continuation Phase.
- ii. Only in case of non-availability of DTG + 3TC FDC. Subjects completing the Continuation Phase must return to the clinic for an End of Continuation Phase visit when transitioning to commercial supplies or to an alternate ART regimen, if appropriate. At this visit, conduct study assessments as specified for all Continuation Phase visits with the exception of dispensing study treatment.

## 13.3. Appendix 3: Assessment Windows

Laboratory data, health outcomes, vital signs and genotypic and phenotypic data will be assigned to assessment windows according to actual dates rather than the nominal visit labels as recorded on the eCRF or in the laboratory database.

A window around a target Study Day will typically include all days from the midpoints between it and the target Study Days of the previous and the proceeding visits. In general, the nominal target study day for week w is (7\*w)+1.

## 13.3.1. Definitions of Assessment Windows for Analyses

| Early Switch Phase | Early Switch Phase | | | | |
|---|---|---|---|---|---|
| Analysis Set / Domain | Parameter | Target | Analy | Analysis | |
| | (if applicable) | | Beginning<br>Timepoint | Ending<br>Timepoint | Timepoint |
| All | All | -35 | ≤-4 | ≤-4 | Screening |
| | | 1 | -3 | 1 | Day 1 |
| | | 29 | 2 | 42 | Week 4 |
| | | 57 | 43 | 70 | Week 8 |
| | | 85 | 71 | 126 | Week 12 |
| | | 169 | 127 | 210 | Week 24 |
| | | 253 | 211 | 294 | Week 36 |
| | | 337 | 295 | 378 | Week 48 |
| | | 421 | 379 | 462 | Week 60 |
| | | 7*w+1 | 7*w-41 | 7*w+42 | Week w, w=72,<br>84, 96, 120 |
| | | 757 | 715 | 798 | Week 108<br>(Optional<br>Visits) * |
| | | 925 | 883 | 966 | Week 132<br>(Optional<br>Visits) * |
| | | 1009 | 967 | 1036, but can be extended up to latest day of scheduled Week 144 visit or unscheduled visit that occurs between Day 1037 and Day 1050 (inclusive). | Week 144 |

<sup>1.</sup> For parameters which are not scheduled to be assessed at particular visits, the all-inclusive windows defined will still be used.

<sup>2.</sup> Assessments at unscheduled visits will be included for 'any time On-treatment' time points and in data listings, as well as algorithms that make use of additional data (e.g., Snapshot). In the event a baseline value is missing, the latest pre-dose value prior to baseline will be used, notwithstanding this date occurring more than 3 days prior to baseline.

<sup>\*</sup> Optional study visit is conducted as per a site and/or participant decision. Data from these visits will be listed but not summarized

| Analysis Set / | Parameter | Arm | Target | Analysis | Window | Analysis |
|---|---|---|---|---|---|---|
| Domain | (if applicable) | | | Beginning<br>Timepoint | Ending<br>Timepoint | Timepoint |
| Efficacy/HO/Safety | Snapshot endpoints, CD8+,lipids, | DTG+3TC<br>(Visit Not<br>Applicable) | Not<br>Applicable | Not<br>Applicable | Not<br>Applicable | Week 148 |
| | glucose, Insulin,<br>HbA1c<br>biomarkers<br>telomere,<br>urinalysis,<br>EQ5D &<br>CSSRS | TBR | 1037 | 1037 | 1037 | |
| | | DTG+3TC<br>(Visit Not<br>Applicable) | Not<br>Applicable | Not<br>Applicable | Not<br>Applicable | Week 152 |
| | | TBR | 1065 | 1038 | 1092 | |
| | | DTG+3TC<br>(Optional<br>visit)* | 1121 | 1093 | 1162 | Week 160 |
| | | TBR | 1121 | 1093 | 1162 | 1 |
| | | DTG+3TC | 1205 | 1163 | 1246 | Week 172 |
| | | TBR | 1205 | 1163 | 1246 | 1 |
| | | DTG+3TC<br>(Optional<br>visit)* | 1289 | 1247 | 1330 | Week 184 |
| | | TBR<br>(Optional<br>visit)* | 1289 | 1247 | 1330 | |
| | | DTG+3TC | 1373 | 1331 | 1414 | Week 196 |
| | | TBR | 1373 | 1331 | 1414 | (7*w-41d,<br>7*w+42d) |
| | | | | be -/+6 weeks, V<br>alysis window for | | al visit will be |
| | | | Study Day<br>of last<br>dose + 28 | >Study Day<br>of last dose<br>+1 | >Study Day<br>of last dose<br>+1 | Follow-up |

- 1. For parameters which are not scheduled to be assessed at particular visits, the all-inclusive windows defined will still be used.
- 2. Assessments at unscheduled visits will be included for 'any time On-treatment' time points and in data listings, as well as algorithms that make use of additional data (e.g., Snapshot).
- 3. In the event a baseline value is missing, the latest pre-dose value prior to baseline will be used, notwithstanding this date occurring more than 3 days prior to baseline.
- 4. This assessment windows applies to the endpoints collected at Week 196, but not at Week 200 visit.

<sup>\*</sup> Optional study visit is conducted as per a site and/or participant decision. Data from these visits will be listed but not summarized

| Late Switch Pha | ase | | | | | |
|---|---|---|---|---|---|---|
| Analysis Set / | Parameter | Arm | Target | Analysis | Analysis | |
| Domain | (if<br>applicable) | | | Beginning<br>Timepoint | Ending<br>Timepoint | Timepoint |
| Efficacy/Safety | Vital Signs,<br>BMI, clinical<br>chemistry, | DTG+3TC<br>(Visit Not<br>Applicable) | Not<br>Applicable | Not<br>Applicable | Not<br>Applicable | Week 148 |
| | Haematology,<br>HIV<br>associated<br>conditions,<br>AEs,<br>concomitant<br>medications | TBR | 1037 | 1037 | 1037 | |
| | | DTG+3TC<br>(Visit Not<br>Applicable) | Not<br>Applicable | Not<br>Applicable | Not<br>Applicable | Week 152 |
| | | TBR | 1065 | 1038 | 1092 | |
| | | DTG+3TC<br>(Optional<br>visit)* | 1121 | 1093 | 1162 | Week 160 |
| | | TBR | 1121 | 1093 | 1162 | |
| | | DTG+3TC | 1205 | 1163 | 1246 | Week 172 |
| | | TBR | 1205 | 1163 | 1246 | |
| | | DTG+3TC<br>(Optional<br>visit)* | 1289 | 1247 | 1330 | Week 184 |
| | | TBR<br>(Optional<br>visit)* | 1289 | 1247 | 1330 | |
| | | DTG+3TC | 1373 | 1331 | 1386 | Week 196 |
| | TBR 1373 1331 1386 | 1386 | (7*w-41d,<br>7*w+14d) | | | |
| | | DTG+3TC | 1401 | 1387 | 1414 | Week 200 (7*w- |
| | | TBR | 1401 | 1387 | 1414 | 13d, 7*w+14d) |
| | | | Study Day<br>of last<br>dose + 28 | >Study Day<br>of last dose<br>+1 | >Study Day<br>of last dose<br>+1 | Follow-up |

- 1. For parameters which are not scheduled to be assessed at particular visits, the all-inclusive windows defined will still be used.
- 2. Assessments at unscheduled visits will be included for 'any time On-treatment' time points and in data listings, as well as algorithms that make use of additional data (e.g., Snapshot).
- 3. In the eventa baseline value is missing, the latest pre-dose value prior to baseline will be used, notwithstanding this date occurring more than 3 days prior to baseline.
- 4. This assessment windows applies to the endpoints collected at both W196 and W200 visit.

<sup>\*</sup> Optional study visit is conducted as per a site and/or participant decision. Data from these visits will be listed but not summarized

# 13.3.2. Definitions of Assessment Windows for Inclusion in the PK Analysis

Not applicable to analyses post Week 48.

The windows for inclusion of PK samples in summary statistics will be as follows:

- For intensive PK population (Week 4 only):
  - Samples collected 1 hour prior to dose for pre-dose sample
  - Samples collected within ±15 min of the 0.5, 1, 1.5, 2 H time points
  - o Samples collected within ± 30 min of the 3h, 4h, 6h time points
  - Samples collected within ± 1h for the 10h time point
  - Samples collected within ± 2h for the 24 h time point
- For sparse PK population (Weeks, 4, 8, 12, 24, 36 and 48):
  - Samples collected within 1 hour prior to dose for pre-dose sample, within ±15 min
    of the 1H time point, within ±30 min window for 1-4hr post dose sample (i.e.
    between 0.5-4.5hr) and within ±60 min window for 4-12hr post dose sample (i.e.
    between 3-13hr).

Outside these allowed windows, concentration results will be flagged and NOT included in the calculations for the summaries, but will be used in listings.

Given steady state will be reached by Day 5, sparse PK analyses will use nominal visit windows for all sparse PK analyses.

# 13.4. Appendix 4: Study Phases and Emergent Adverse Events13.4.1. Study Phases

Data collected from both arms up to and including the date of the Week 148 visit will be considered to be during the Early Switch Phase of the study. For subjects randomised to TBR, this will be the date of their Week 148 switch visit. For subjects randomised to DTG + 3TC, this will be calculated as 1035 (=[148x7] - 1)) days after exposure start date or if the latest of scheduled or unscheduled W144 visit takes place between Day 1037 and Day 1050 (inclusive) then the day of W144 visit.

For subjects randomised to DTG + 3TC, data collected from 1036 days after IP start day to Week 200 will be considered to be during the Late Switch Phase. Data collected after Week 200 will be considered to be during the Continuation Phase of the study (if applicable).

For subjects randomised to the TBR arm, data collected from the date of the Week 148 switch visit to Week 200 will be considered to be during the Late Switch Phase of the study. Data collected after Week 200 will be considered to be during the Continuation Phase of the study (if applicable).

| Phase | Randomised | Start | End |
|---|---|---|---|
| Early Switch Phase | DTG+3TC | IP start date | IP start date + 1035 (=[148x7 - 1). If the latest of scheduled or unscheduled W144 visit takes place between Day 1037 and Day 1050 (inclusive) then the day of W144 visit or Withdrawal date on or before study day 1036 |
| | TBR | Day 1 DOV | IP start date for switch to DTG + 3TC -1 or Withdrawal date before Week 148 |
| Late Switch Phase | DTG+3TC* | IP start date +1036 Or the day after the latest of scheduled or unscheduled W144 visit if this visit takes place between Day 1037 and Day 1050 (inclusive) | Week 200 DOV -1<br>or<br>Withdrawal date before Week 200 |
| | TBR** | IP start date for DTG+3TC | Week 200 DOV -1<br>or<br>Withdrawal date before week 200 |

| Phase | Randomised | Start | End |
|---|---|---|---|
| | Arm | | |
| Continuation Phase(if applicable) | DTG+3TC | Week 200 DOV | IP end date or Withdrawal date |
| | TBR | Week 200 DOV | IP end date or Withdrawal date |

<sup>\*</sup> For subjects randomised to DTG + 3TC, data collected from day1037(or the day after scheduled W144 visit if scheduled W144 visit takes place between Day 1037 and Day 1050 (inclusive)) to Week 200 will be considered to be during the Late Switch Phase. There will not be a visit at week 148 in DTG+ 3TC arm, so this needs to be derived programmatically.

13.4.1.1. Study Phases for Laboratory, HIV Associated Conditions, Vital Signs, Health Outcomes and Genotypic and Phenotypic Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | Date ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date < Date ≤ Study Treatment Stop Date + 1 |
| Post-Treatment | Date > Study Treatment Stop Date +1 |

#### NOTES:

## 13.4.1.2. Study Phases for Adverse Events

For adverse events, partial AE start date will use imputation as described in Section 13.7.2.1. In the case of a completely missing start date, the event will be considered to have started On-treatment unless an end date for the AE is provided which is before start of study treatment; in such a case the AE is assigned as Pre-treatment.

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE Start Date < Study Treatment Start Date |
| On-Treatment | If AE onset date is on or after treatment start date & on or before treatment stop date. |
| | Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date |
| Post-Treatment | If AE onset date is after the treatment stop date. |
| | AE Start Date > Study Treatment Stop Date |
| Onset Time Since 1st Dose | If Treatment Start Date > AE Onset Date = AE Onset Date - |
| (Days) | Treatment Start Date |
| | If Treatment Start Date ≤ AE Onset Date = AE Onset Date - |
| | Treatment Start Date +1 |
| | Missing otherwise. |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on CRF. |

<sup>\*\*</sup> For subjects randomised to the TBR arm, IP start date as collected on the late switch eCRF at the Week 148 switch visit will be used to define the beginning of the Late Switch Phase of the study.

<sup>1.</sup> If the study treatment stop date is missing then the assessment will be considered to be On-Treatment

#### NOTES:

- Partial AE start date will use imputation as described in Section 13.7.2.1
- In the case of a completely missing start date, the eventwill be considered to have started On-treatment unless
  an end date for the AE is provided which is before start of investigational product; in such a case the AE is
  assigned as Pre-treatment.
- If the IP Stop Date is missing, then any event with a start date on or after IP Start Date will be considered to be
  On-treatment.
- If the start date of the AE is after IP Stop Date but has been recorded as potentially related to IP, then it will be
  classified as On-treatment.

## 13.4.1.3. Study Phases for Concomitant Medication

- Prior medications: Those taken (i.e., started) before the start date of investigational product.
- Concomitant medications: Those taken (i.e., started or continued) at any time between the start date and stop date of study treatment, inclusive. Prior medications that were continued during this period are also considered as concomitant medications.
- Post treatment medications: Those started after the stop date of study treatment. Concomitant medications that were continued during this period are also considered as post-treatment medications.

It will be assumed that medication has been taken on the date in which it is reported as started or stopped. For any medication starting on the same date as study treatment, it will be assumed that the medication was taken after the subject started taking study treatment.

Duration of episodes of concomitant medication will be calculated as medication stop date – medication start date, so long as the medication is defined as concomitant according to the rules above (and presented below in the scenario matrix). Durations will be left blank if stop date is missing.

ART medications will also be classified as prior to screening, concomitant to screening and/or post-treatment according with the following modifications:

- ART starting on or after study treatment stop date will be considered as only posttreatment and not concomitant. It is expected that after discontinuation of study treatment, a subject may immediately begin taking another ART.
- ART stopping on study treatment start date will only be considered as prior and not concomitant.
- Any ART entered on the Prior ART eCRF with partial end date will be assumed to have finished before Screening.
- ART stopped prior to screening includes all ART that has stopped prior to screening. All ingredients from any regimen that is switched to another regimen prior to the screening visit e.g. from TDF-based to TAF-based ART will be presented as having stopped.
- ART Medications received at or after Day 1 while still on study treatment includes all ART that started after Day 1 and before study treatment discontinuation. Note this will be recorded as ConART
- ART Medications Received at Screening includes all ART that is ongoing at the screening visit only.

| | Pre-treatment | | On-treatment | | | Post-treatment | Prior | Conco-<br>mitant | Post |
|---|---|---|---|---|---|---|---|---|---|
| (a) | ХХ | | | | | | Υ | N | N |
| (b) | X | | ———Х | | | | Υ | Y | N |
| (c) | X <u>-</u> | | | | | ———х | Υ | Y | Υ |
| (d) | | | ХХ | | | | N | Y | N |
| (e) | | بو | Χ | يو | + | ———х | N | Y | Υ |
| (f) | | Daf | | Daí | ate | хх | N | N | Υ |
| (g) | ?x | IP Start Date | | IP Stop Date | IP Stop Date+1 | | Υ | N | N |
| (h) | ? | St | ———Х | Š | Sto | | <b>Y</b> * | Y | N |
| (i) | ? | _ ₾ | <del></del> | <u> </u> | <u> </u> | x | Υ* | Y* | Υ |
| (j) | X | | | | | ? | Υ | Y** | Y** |
| (k) | _ | | X | | | ? | N | Y | Y** |
| (I) | | | | | | x? | N | N | Υ |
| (m) | ? | | <del></del> | | | ? | Y*** | γ*** | Y*** |
| (n) | X | х | | | | | Υ | Υ | N |
| (o) | ? | Х | | | | | <b>Y</b> * | Υ | N |
| (p) | | Х | ———Х | | | | N | Y | N |
| (p) | | Х | <del></del> | Х | | | N | Y | N |
| (r) | | | | х | | ———х | N | Y | Υ |
| (s) | | | | х | | ? | N | Y | Y** |
| (t) | | | | | Χ | ———х | N | N | Υ |
| (u) | | | | | Χ | ? | N | N | Υ |
| (v) | | | X | | Χ | | N | Y | Υ |

#### CONFIDENTIAL

204862

- 1. x = start/stop date of medication
- ? = missing start/stop date of medication
   \* If a medication is stopped On-treatment or Post-treatment and no start date is recorded it will be assumed that the medication was ongoing from the Pretreatment phase
- 4. \*\* If a medication is started Pre-treatment or On-treatment and no stop date is recorded then usage will be assumed to be ongoing for the remainder of the study
  5. \*\*\* If a medication has no start or stop date it will be assumed that the medication was ongoing from the Pre-treatment phase to the Post-treatment phase

## 13.4.2. Combining Treatment Phases and States

On-treatment and Post-treatment assessments and events will be classified as occurring during the Early Switch, Late Switch or Continuation Phase of the study (if applicable) as follow:

- If a subject did not enter the Late Switch Phase, then any Post-treatment data will be assigned to the Early Switch Phase.
- For subjects who did enter the Late Switch Phase, If a subject did not enter the Continuation Phase, then any Post-treatment data will be assigned to the Late Switch Phase (provided this was after the Early Switch Phase).
- For subjects who did enter the Continuation Phase, any Post-treatment data will be assigned to the Continuation Phase.

For concomitant medication, if there is a duration overlapping any period then this should be reflected such that a concomitant medication (at time of the data cut):

- Starting and ending before treatment start then phase is set to missing
- Is taken at any point during the early switch phase only then phase is set to "Early Switch Phase"
- Is taken at any point during the late switch phase only then phase is set to "Late Switch Phase"
- Is taken at any point during the continuation phase only then phase is set to "Continuation Phase"
- Is taken at any point across the early and late switch phases only then phase is set to "Early and Late Switch Phase"
- Is taken at any point across the late and continuation phases only then phase is set to "Late Switch and Continuation Phase"
- Is taken at any point across all three phases then phase is set to "Early Switch and Late Switch and Continuation Phase".

## 13.4.3. Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Emergent | Emergent refers to AE Severity/ Lab toxicity that develops or increases in intensity after baseline |

For adverse events, partial AE start date will use imputation as described in Section 13.7.2. In the case of a completely missing start date, the event will be considered to have started On-treatment unless an end date for the AE is provided which is before start of investigational product; in such a case the AE is assigned as Pre-treatment.

For laboratory data, there will be no imputation of dates, which are expected to be fully complete and available in SDTM transfers. Any laboratory dates that are partially missing will be queried.

# 13.5. Appendix 5: Data Display Standards & Handling Conventions

## 13.5.1. Reporting Process

| <ul> <li>The currently supported versions of SAS software and any other statistical reporting<br/>software required for the analysis and reporting will be used.</li> </ul> |
|---|
| Reporting Area |
| HARP Server uk1salx00175 |
| HARP Compound :\ARPROD\GSK3515864\mid204862\reporting_effort_number |

#### **Analysis Datasets**

Software

- Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 & ADaM IG Version 1.0).
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented as SDTM.

#### **Generation of RTF Files**

RTF files will be generated for all reporting efforts.

## 13.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location:
  - https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings
- All data displays will use the term "subjects" rather than "participants".

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.
  - For [Insert Endpoint / Parameter] the following DP's places will be applied:
  - Summary Statistics:
  - Listings:

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Actual time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

- Unscheduled visits will be assigned to a study visit using the all-inclusive windows defined in Section 13.3.
- However, data summaries will only report visits that are planned assessment time points for each parameter (according to the Time and Events table).
- Assessments at unscheduled visits will be included for 'any time On-treatment' time points and in data listings, as well any algorithms that make use of additional data (e.g., Snapshot).

#### **Optional Visits**

 For optional visits (DTG+3TC-Week 108, 132, 160 & 184, TBR-Week 108, 132 &184), data will be listed but will not be summarized

## Listings

Listings will include all data, regardless of treatment phase or state.

#### Treatment Phases and States

- Study population, efficacy, virology and health outcome tables will not include post-treatment data according to the phase, unless otherwise stated. The data will be presented up to the visit window of interest.
- Safety tables will present on-treatment and post-treatment data according to the phase, unless otherwise stated.

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7 01 to 7 13 | |

## 13.5.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Concentration Data | |
|---|---|
| PC Windows Non-Linear<br>(WNL) File | PC WNL file (CSV format) for the non-compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to PK One document (Standards for the Transfer and Reporting of PK Data using HARP). Note: Concentration values will be imputed as per GUI_51487 |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| NONMEM/Pop PK File | Pop-PK file (CSV format) for the POP-PK analysis by Clinical PharmacologyModelling and Simulation function will be created according to the data specification detailed in a separate RAP |
| NONMEM/PK/PD File | Pop-PKPD file (CSV format) for the POP-PK analysis by Clinical PharmacologyModelling and Simulation function will be created according to the data specification detailed in a separate RAP. |
| Pharmacokinetic Param | eter Derivation |
| PK Parameter to be<br>Derived by Programmer | The PK parameters will be calculated by standard non-<br>compartmental analysis according to current working practices and<br>using WinNonLin v 5.2 or above. All calculations of non-<br>compartmental parameters will be based on actual sampling times. |
| Pharmacokinetic Param | eter Data |
| Is NQ impacted PK Parameters Rule Being Followed | If any PK parameter is not calculable because of NQs, it will be noted as NC (non-calculable) for the PKPar file and excluded (set to missing) from the PK parameter summary statistics. Refer to PK One document (Standards for the Transfer and Reporting of PK Data using HARP) for handling of non-numeric values in the parameter data. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. |

Not applicable to analyses post Week 48.

## 13.6. Appendix 6: Derived and Transformed Data

#### 13.6.1. General

## Multiple Measurements at One Time Point

- If there are multiple assessments within Screening window, the last assessment before Day 1 will be used
- If there are multiple assessments within Day 1 window, the latest pre-dose assessment will be used
- With the exception of the Snapshot endpoints, if after window assignment (see Section 13.3), there are multiple valid assessments of a parameter within the same window, then the following hierarchy will be used to determine the value to be used for summary statistics of observed values:
  - the assessment closest to the window target Study Day;
  - o if there are multiple assessments equidistant from the target Study Day, then the mean of these values will be used. For HIV-1 RNA, the geometric mean of the number of copies will be used as opposed to the arithmetic mean
- Assessments not chosen for use in summary statistics by this algorithm will still appear in
  the associated listings. Also, such valid assessments will be used when determining values
  of potential clinical concern for the 'any time On-treatment' time point, and for any algorithm
  that has specific rules for which observation to use (e.g., SNAPSHOT or LOCF).
- In the event of laboratory re-tests being performed the last re-test in the visit window will be used. For example:
- If a subject had a week 24 viral load and then two re-tests (i.e. three viral loads labeled as week 24, unscheduled 1 unscheduled 2). and the first two viral loads were within the upper bound of the week 24 visit (Day 210) but the last re-test was slotted to week 36 then the last re-test would not be used for the week 24 snapshot.
- If a subject had a week 24 viral load but the re-test was performed on Day 220 (week 36) then the re-test viral load would not be used for the week 24 snapshot.

#### Study Day

- Calculated as the number of days from initial study treatment start date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Treatment Start Date → Study Day = Ref Date -Treatment Start Date</li>
  - Ref Data ≥ Treatment Start Date → Study Day = Ref Date (Treatment Start Date) + 1

Note that Treatment Start Date is considered to be on Study Day 1 and the day before this is Study Day -1; i.e., there is no Study Day 0.

#### Post-baseline

Post-baseline refers to the combined time periods of On-treatment and Post-treatment.
 Post-baseline may be further specified according to phase of the study. Randomised Early Switch, Late Switch and Continuation Phase.

#### Study Drug

• Study Drug refers to either Investigational Product DTG + 3TC or TBR.

## 13.6.2. Study Population

#### **Demographics**

#### Age

- Age, in whole years, will be calculated with respect to the subject's Screening visit where year
  of birth is collected.
- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing date and month will have this imputed as '30th June'.
  - For analysis purposes, if a subject did not fail to meet inclusion criteria #1 (aged 18 years or older), then set any age imputed as <18 by the standard IDSL algorithm to 18. If the subject failed to meet inclusion criteria #1 then the imputed age will not be reset.</li>
- Birth date will be presented in listings as 'YYYY'.
- Completely missing dates of birth will remain as missing, with no imputation applied.
   Consequently, the age of the subject will not be calculated and will remain missing.

## Framingham Risk Equation

The predicted probability, , of having a cardiovascular disease (CVD) within the next 10-years according to the Framingham formula [D'Agostino, 2008] is

for females:

$$F = 1 - S_0(t) \exp\{2.32888 \times \log(\text{age}) + 1.20904 \times \log(TC) - 0.70833 \times \log(HDL) + 2.76157 \times \log(SBPu) + 2.82263 \times \log(SBPt) + 0.52873 \times I_S + 0.69154 \times I_d - 26.1931\}$$

for males:

$$M = 1 - S_0(t) \exp\{3.06117 \times \log(\text{age}) + 1.12370 \times \log(TC) - 0.93263 \times \log(HDL) + 1.93303 \times \log(SBPu) + 1.99881 \times \log(SBPt) + 0.65451 \times I_S + 0.57367 \times I_d - 23.9802\}.$$

where

 $S_0(t) =$ 

TC = total serum cholesterol (mg/dL),

HDL = serum HDL cholesterol (mg/dL),

SBPu = systolic blood pressure (mmHg) if subject is not treated for high blood pressure (note that if a subject is treated for high blood pressure then log(SBPu) = 0)

SBPt = systolic blood pressure (mmHg) if subject is treated for high blood pressure (note that if a subject is not treated for high blood pressure then log(SBPt) = 0)

$$I_{s} = \begin{cases} 1, \ current \ smo \ \ker \\ 0, \ otherwise \end{cases}$$
 
$$I_{d} = \begin{cases} 1, \ diabetic \\ 0, \ otherwise \end{cases}$$

 Smoking status is collected in the eCRF on Day 1. A current smoker is defined as currently smoking/using tobacco or has smoked/used tobacco within the previous 6 months; a former smoker is defined as previously smoked/used tobacco products and has not smoked/used tobacco products within the previous 6 months.

## **Demographics**

- Risk score needs to be calculated at baseline week 144 and Week 196. For deriving
  week 144 and Week 196 risk score, use the lab and vital signs values of the respective
  visits and target age at that visit needs to be derived
- This calculation will not be performed for subjects who have indicated current or past
  myocardial infarction conditions on the eCRF. These subjects will not be included in
  summary statistics of risk and change from baseline in risk, but will be counted in the
  highest category of risk in the summary by category

#### Extent of Exposure

- Exposure to DTG + 3TC will be calculated from the IP eCRF pages. Exposure to TBR will be calculated from the CONART eCRF pages.
- Subjects who were randomised to DTG + 3TC but did not report a IP start date will be categorised as having zero days of exposure.
- Subjects who were randomised to TBR but withdrew on Day1 will be categorised as having zero days of exposure
- Missing Treatment Stop Date will be imputed, for purposes of calculating exposure, as the date
  of last visit or the recorded date of withdrawal/completion, whichever is earlier.
- Actual exposure will be calculated where the duration of any dosing interruptions based on eCRF data will be subtracted from the result above.
- The ratio (percentage) of the actual exposure to the overall exposure (i.e. study treatment stop date study treatment start date+1) will be used to define protocol deviation leading to exclusion from PP Population due to study treatment interruption (i.e. >10%).
- Further clarifications on extent of exposure during the early and late switch phases is provided in the Section 13.6.4.

#### Strata

- For analysis purposes, randomisation strata will be used from that derived using eCRF data, even if this differs from the strata captured in IVRS.
- For patients randomised to DTG + 3TC, baseline third agent class is collected on the prior ART history form. For patients randomised to current TBR, baseline third agent class is collected on the concomitant ART form.
- Third agent class is identified using terms from the GSK Drug Dictionary

## 13.6.3. Efficacy

#### **HIV-1 RNA**

#### Snapshot

- It is intended to be primarily a virologic assessment of the endpoint, and as such follows a "virology first" hierarchy.
- Virologic Success (e.g., <50 c/mL) or Virologic Failure within an analysis window (see Section 13.3) is typically determined by the last available HIV-1 RNA measurement in that window while the subject is On-treatment.
- When no HIV-1 RNA data is available within a window, a subject cannot be a Virologic Success. Depending on the reason for lack of data, the subject will be classified as a Virologic Failure or reported as 'No Virologic Data at Week X'; in the latter case, the algorithm further classifies the nature of the missing data. Typically, a subject withdrawn (i) due to AE or, (ii) for another reason yet was suppressed at the time, will be counted as 'No Virologic Data at Week X'. Should a subject withdraw for reasons other than AE and was not suppressed at the time, they will be a Virologic Failure.
- For each scheduled assessment time, the snapshot response rate for a given threshold (e.g.,
   <50 c/mL) is defined as:</li>

Snapshot Rate =  $\frac{\text{Number of responders in that analysis window}}{\text{Number of subjects in the analysis population}}$ 

 Full details of the algorithm, including the handling of special cases, are included in Section 13.11 of note, the date at which the subject 'discontinue/withdrawn from the study' in the Snapshot algorithm is the date of treatment discontinuation, rather than the date of study withdrawal,

#### Plasma HIV-1 RNA

- For summaries and analyses which use HIV-1 RNA level as a continuous measure, the logarithm to base 10 of the value will be used.
- HIV-1 RNA results may be provided as censored values, such as <40 or >9,999,999 c/mL. For
  the purposes of summary statistics, such values will be replaced by the next value beyond the
  limit of detection, e.g., 39 or 10,000,000 c/mL, respectively, for the given examples. Data
  listings will show the censored values as provided.
- Qualitive measures (i.e. "target detected" and "target non-detected") may also be provided by
  the laboratory vendor for values <40 c/ml. When a measurement of plasma HIV-1 RNA is below
  the limit of quantification (i.e. 40 c/mL) and is qualitatively observable that will be denoted as a
  "Target Detected" measure, while HIV-1 RNA below the limit of quantification that is not
  qualitatively observable that will be denoted as "Target Not Detected". Any measurements <40
  c/mL characterised as "Target Non-Detected" or "Target Detected" will be captured in the
  database.</li>

Confirmed Virologic Withdrawal (CVW), Suspected Virologic Withdrawal (SVW) and Precautionary Virologic Withdrawal (PVW) and potential Precautionary Virologic Withdrawal (pPWW)

Please refer to the protocol, Section 5.4.1 for more details of the derivation of CVW, PVW, pPVW and SVWs.

#### HIV-1 RNA

PVW (leading to discontinuation – this definition will not be used in statistical analysis or reporting)

May be met after two consecutive assessments with HIV-1 RNA >=50 and <200 c/mL without an identifiable, non-virologic cause (immunization, illness, nonadherence) and after discussion with Medical Monitor, ORWill be met with three consecutive assessments with HIV-1 RNA >=50 and <200 c/mL</li>

#### <u>pPVW</u>

 Will be met after two consecutive assessments with HIV-1 RNA >=50 and <200 c/mL (instances where a first elevation of HIV-1 RNA >=200 c/mL followed by HIV-1 RNA >=50 and <200 c/mL will also be considered pPVW</li>

## <u>SVW</u>

 One assessment with HIV-1 RNA >= 200 c/mL after Day 1 with an immediatelyprior HIV-1 RNA <50 c/mL.</li>

#### **CVW**

 One assessment with HIV-1 RNA >= 200 c/mL after Day 1 with an immediately prior HIV-1 RNA >=50 c/mL.

#### **General Considerations**

- The subsequent HIV-1 RNA sample taken after SWW will be used for the determination of CVW.
- Based on the protocol specific conditions outlined in the protocol, derivation of SWW and CWW will use nominal visits and unscheduled visits.
- Visit windowing will not be applied.
- The condition of 2-4 weeks between the suspected and confirmatory re-test (as described in protocol Section 5.4) will not be used when programmatically identifying CVW.
- A patient can only be classified as CVW for the analyses if the patient has not withdrawn IP at the time of the HIV-RNA re-test value (at CVW value), where Treatment Start < HIV-1 RNA sample date <= Treatment Stop Date + 1 (if Treatment Stop date exists). Note: study drug interruptions will not be taken into account when programmatically identifying CVW.</li>
- Similarly, viral loads above criteria cut-offs resulting in SWW, CWW, PWW and pPWW need
  to have occurred post-Day 1 in order for the criteria to be met. For example an SWW can
  occur at Week 4 if Week 4 HIV-1 RNA >=200 i.e. the viral load above SWW criterion
  occurred post-Day 1.
- Additional guidelines specified in the protocol related to patient management only and will
  not be taken into account when programmatically identifying CWW.
- Please refer to Section 5.4.1 of the protocol for details of the derivation.

#### HIV-1 RNA

#### CDC HIV-1 Classification and HIV-associated conditions

- HIV associated conditions will be assessed according to the 2014 CDC Revised Classification System for HIV Infection in Adults (see protocol Section 13.7).
- Any 'other' conditions reported in the CRFs will be identified programmatically before being sent for clinical review to determine whether they should be classed as stage 3 associated conditions. Review will be ongoing and as a minimum will take place prior to each reporting effort.

## 13.6.4. Safety

## **Extent of Exposure**

 Exposure to DTG + 3TC will be calculated from the IP eCRF pages. Exposure to TBR will be calculated from the CONART eCRF pages. Number of days of exposure to study drug will be calculated as:

Duration of Exposure in Days = Treatment Stop Date – (Treatment Start Date) + 1

For subjects randomised to DTG + 3TC at Day 1:

- For Early Switch Phase:
  - For subjects completing the early switch phase Exposure = IP Start Date + 1035 (=[7\*148] -1) or if the latest of scheduled or unscheduled W144 visit takes place between Day 1037 and Day 1050 (inclusive) then the day of W144 visit
  - If a subject discontinues prior to Week 144 (Day 1036), the IP Stop Date recorded in the eCRF will be used. A partial or missing IP stop date is handled as described in Section 13.7.2.1.
- A Day 1 Date of Visit will be used for partial or missing IP start date. For Late switch phase:
  - Start date of late switch phase is IP start date +1036 or the day after the latest of scheduled or unscheduled W144 visit if this visit takes place between Day 1037 and Day 1050 (inclusive)
- The overall exposure is calculated as
  - Exposure = IP Stop Date IP Start Date + 1

For subjects randomised to TBR at Day 1:

- For Early Switch Phase:
  - Exposure = (IP Start Date 1) Day 1 DOV + 1
  - If a subject discontinues prior to Week 148, the Withdrawal Date (earliest of date recorded in disposition, study visit page and TBR stop date) recorded in the eCRF will be used in the following way:
    - Exposure = (earliest of date recorded in disposition, study visit page and TBR stop date) Day 1 DOV + 1
- After the Week 148 switch visit, the exposure to DTG + 3TC is calculated as
  - Exposure = IP Stop Date IP Start Date + 1.

## Extent of Exposure

- Duration of dosing in subject years will be calculated as the sum of subject duration of dosing in days (across all subjects)/365.25
- Subjects who were randomised to DTG + 3TC but did not report a IP start date will be categorised as having zero days of exposure.
- Subjects who were randomised to TBR but withdrew on Day1 will be categorised as having zero days of exposure.
- Missing Treatment Stop Date will be imputed, for purposes of calculating exposure, as the date
  of last visit or the recorded date of withdrawal/completion, whichever is earlier.
- An alternative calculation of exposure will be performed where the duration of any dosing interruptions based on eCRF data will be subtracted from the result above.
- The ratio (percentage) of the actual exposure to the overall exposure (i.e. study treatment stop date – study treatment start date+1) will be used to define protocol deviation leading to exclusion from PP Population due to study treatment interruption (i.e. >10%).

#### Adverse Events

## AE Severity - DAIDS Grading

- The DAIDS grading (VERSION 2.1, March 2017) for severity of clinical adverse events will be performed.
- See protocol for DAIDS grading criteria.

## Adverse Events of Special Interest (AESI)

The preferred terms for each AESI will be updated on an ongoing effort before each formal analysis in a separate document. The following table below shows the AESI categories.

| AESI |
|-----------------------------|
| Anxiety |
| Depression |
| Drug Hypersensitivity |
| Insomnia |
| Nightmare/Abnormal Dreams |
| Rash |
| Suicidality and self-injury |
| Weight increased |
| Weight decreased |

## **Laboratory Parameters**

- Additional non-protocol specified laboratory assessments performed at the institution's local laboratory that are databased will not be included in the listings or analyses/summaries. All analyses will be based on central laboratory assessments only. If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01</li>
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - $\circ$  Example 3: 0 Significant Digits = '< x' becomes x 1

## Lab Toxicities - DAIDS Grading

- Toxicities will be based on the Division of AIDS (DAIDS) grading system, as specified in the protocol.
- Toxicity grades provided by the central laboratory do not distinguish between abnormally high or low criteria, when both are relevant for a particular parameter.
- When summarising toxicity grades for such parameters, they will be categorised as to whether they are above or below the midpoint of normal range.

| Parameter | Below Midpoint | Above Midpoint |
|----------------|----------------|----------------|
| Calcium | Hypocalcaemia | Hypercalcaemia |
| Fasted glucose | Hypoglycaemia | Hyperglycaemia |
| Sodium | Hyponatremia | Hypernatremia |
| Potassium | Hypokalemia | Hyperkalemia |

## National Cholesterol Education Program (NCEP) Lipid Categories

 In addition to DAIDS toxicity scales (see protocol), lipid values will be categorized according to the 2001 NCEP Adult Lipid Guidelines [Grundy, 2001].

| Parameter | Value Range (mmol/L) | Value Range (mg/dL) | Category |
|---|---|---|---|
| Triglycerides | <1.70 | <150 | Normal |
| | 1.70 to <2.26 | 150 to <200 | Borderline High |
| | 2.26 to <5.65 | 200 to <500 | High |
| | ≥5.65 | ≥500 | Very High |
| Total Cholesterol | <5.18 | <200 | Desirable |
| | 5.18 to <6.21 | 200 to <240 | Borderline High |
| | ≥6.21 | ≥240 | High |
| HDL Cholesterol | <1.04 | <40 | Low |
| | 1.04 to <1.56 | 40 to <60 | Normal |
| | ≥1.56 | ≥60 | High |
| LDL Cholesterol | <2.59 | <100 | Optimal |
| | 2.59 to <3.37 | 100 to <130 | Near/Above Optimal |
| | 3.37 to <4.14 | 130 to <160 | Borderline High |
| | 4.14 to <4.92 | 160 to <190 | High |
| | ≥4.92 | ≥190 | Very High |

## **Laboratory Parameters**

## Glomerular Filtration Rate (GFR)

Chronic Kidney Disease EpidemiologyCollaboration (CKD-EPI) equation [Levey, 2009] will be
used by the central laboratory to provide an estimate of GFR, in mL/min per 1.73 m2, as follows
for the CKD-EPI creatinine equation:

$$GFR = 141 \times min \left(\frac{CRT_{mg/dL}}{\kappa}, 1\right)^{\alpha} \times max \left(\frac{CRT_{mg/dL}}{\kappa}, 1\right)^{-1.209} \times 0.993^{Age} \times [1.018 \text{ if Female}] \times [1.159 \text{ if Black}]$$

where age (in years) is at time of assessment,  $\kappa = 0.7$  if female or 0.9 if male,  $\alpha = -0.329$  if female and -0.411 if male, min() indicates the minimum of CRT/ $\kappa$  or 1, max() indicates the maximum of CRT/ $\kappa$  or 1, and CRT mg/dL is serum creatinine concentration in mg/dL. The serum creatinine concentration in mg/dL is obtained from GSK standard units of  $\mu$ mol/L as CRT mg/dL =0.0113x CRT  $\mu$ mol/L.

## **CKD-EPI Cystatin C Equation (2012)**

The following will be used for the CKD-EPI Cystatin C Equation:

eGFR =  $133 \times \min(\text{Scys/0.8}, 1)^{-0.499} \times \max(\text{Scys/0.8}, 1)^{-1.328} \times 0.996^{\text{Age}} \times 0.932$  [if female]

Abbreviations / Units

eGFR (estimated glomerular filtration rate) = mL/min/1.73 m2

Scys (standardized serum cystatin C) = mg/l

min = indicates the minimum of Scys/0.8 or 1

max = indicates the maximum of Scys/0.8 or 1

age = years

Assays

#### Total Cholesterol / HDL Cholesterol Ratio

 When both total cholesterol and HDL cholesterol results are available from the same date for a subject, then the ratio will be calculated by dividing the total cholesterol result by the HDL cholesterol result. The ratio can be classified as follows:

| Parameter | Value Range |
|-------------------|--------------|
| Total Cholesterol | < 3.5 |
| / HDL Ratio | 3.5 to < 4.4 |
| | 4.4 to < 5 |
| | ≥5 |

#### **Hepatitis Status**

- Hepatitis C status will be determined using antibody (IgM or IgG) and/or hepatitis C virus (HCV) RNA assessments performed during screening.
- If both antibody and virus RNA assessments are available, then the latter will take precedence and positive/negative status will be based on whether HCV RNA is detectable (i.e., ≥43 IU/mL [≥1.63 log IU/mL]) or not
- Antibody (IgM or IgG) status with 'BORDERLINE' or 'REACTIVE' will be considered Positive
- A subject will be considered positive for hepatitis B virus (HBV) if they have a positive surface antigen or detectable HBV DNA result during screening. Subjects positive for HBV are not allowed to enter the study.

#### **BMI**

BMI classification is based on standard categories adopted by the WHO and FDA:

Underweight = BMI of < 18.5 kg/m2

Normal = BMI of 18.5 - 24.99 kg/m2

Overweight = BMI of 25 - 29.99 kg/m2

Obese = BMI of > =30 kg/m2

Note: Any shift to a higher BMI category counts as a shift to a 'worse category'.

## Other Safety Endpoints

## Columbia Suicide Severity Rating Scale (C-SSRS)

- Missing data will not have any imputation performed.
- A positive alert is triggered if a subject has reported suicidal ideation/behaviour in categories 4-
- Questions in categories 3-5 will be triggered if suicidal ideation is reported in categories 1 or/and
- Incomplete calls:
  - when no complete call is databased on the same day, the data from the incomplete call will be used
  - o if a subject has only an incomplete call, and it resulted in a positive alert, the relevant pages in the CRF should be completed, even though the call was incomplete
  - when a complete call is databased on the same day, the data from the complete call will be used in the summaries.
- Duplicate calls, if they occur on the same day.
  - Both calls will be reported in the listings.
  - o For summary tables, the entry with latest time record will be used.
  - o For summary tables at baseline, unscheduled repeat visits will not be summarised.
  - Relevant CRF pages will be completed based on the latest entry (if it was a positive alert).
- Late Day 1 assessments
  - Late DAY 1 assessments will be summarised as representing baseline status (i.e., treated as true DAY 1 assessments). Where this leads to multiple DAY 1 assessments, 'complete' assessments will be used over 'incomplete' assessments to represent baseline status. Such assessments will be considered DAY 1 if they occur by Day 14.
- Day 1 assessments performed at later visits
  - DAY 1 assessments on (or close to) study day 1 will be accepted as DAY 1
    assessments (as above). For DAY 1 assessments performed at later visits, the
    'Lifetime' assessment observation will not be summarised but the 'Within the past 2
    months' assessment will be used as a surrogate for the later post-baseline visit
    assessment.

## Homeostatic model assessment-Insulin Resistance (HOMA-IR)

- HOMA-IR = (fasting plasma insulin (mU/L) \* fasting plasma glucose (mmol/L)) / 22.5.
- HOMA-IR categories will be categorised as follows for the HOMA-IR shift table analysis:
  - 0 <2
  - o 2 to <3
  - o 3 to <4
  - o >=4

HOMA-IR shift tables will be presented for baseline vs maximum value post-baseline and Week X, for Weeks 24, 48 and only for baseline vs Week X for Weeks 96 and 144. HOMA-IR categories will be broken down into: <2, 2 to <3, 3 to <4 and >=4.

All HOMA-IR analyses will be based on fasting values and only patients with post-baseline values will be included in analyses (i.e. patients with missing post-baseline HOMA-IR will not be included in summary tables or figures). Additionally, patients who are diabetic as captured on the medical history form at screening will be excluded from all HOMA-IR analyses. Finally, patients with anti-diabetic medication starting at or prior to screening are excluded.

## Metabolic Syndrome per IDF definition

Metabolic syndrome (required at Baseline, Week 144 and Week 196) is defined as a subject having:

Central obesity (defined as the last value within the visit window of interest as BMI>=30kg/m2)

plus any two of the following four factors:

| Raised<br>triglycerides | The last fasted value within visit window of interest >=150 mg/dL (1.7 mmol/L) or specific treatment for this lipid* abnormality at any time prior the end of the visit window of interest |
|---|---|
| Reduced HDL | The last fasted value within visit window of interest: |
| cholesterol | < 40 mg/dL (1.03 mmol/L) in males < 50 mg/dL (1.29 mmol/L) in females or specific treatment for this lipid* abnormality at any time prior the end of the visit window of interest |
| Raised blood pressure | Systolic BP $\geq$ 130 or diastolic BP $\geq$ 85 mm Hg or treatment* of previously diagnosed hypertension at any time prior the end of the visit window of interest |

| | or any AE with preferred term "Hypertension", "Essential hypertension", "Blood pressure increased" or "Blood pressure diastolic increased" experienced at any time prior to the end of the visit window of interest |
|---|---|
| Raised fasting plasma glucose | The last value within visit window of interest (FPG) >= 100 mg/dL (5.6 mmol/L), |
| | <i>or</i> previously diagnosed type 2 diabetes at any time prior the end of the visit window of interest |

<sup>\*</sup> List of the unique medications identified by the clinical review of the Week 196 data for determination of Metabolic Syndrome (for lipid abnormalities i.e. triglyceride elevations and HDL reductions, and hypertension-related medications) will be provided.

#### 13.6.5. Pharmacokinetic

#### General

 Data at specific timepoints of subjects who had major PK protocol deviations that could impact DTG or 3TC exposure will be removed, as detailed below:

| PK Protocol Deviation | Populations Affected | Analysis Consideration |
|---|---|---|
| Non-fasting 8 hours pre-dose | - Intensive Concentration and Parameter Populations | Pre-dose and subsequent samples that day (not including 24 hours) will be excluded from summaries and figures but will be included in listings and flagged |
| Use of prohibited medications* at time of sample | <ul><li>Intensive Concentration and<br/>Parameter Populations</li><li>Sparse Population</li></ul> | Samples will be excluded from summaries and figures but will be included in listings and flagged |

- The Intensive pharmacokinetic population will be used for listing PK concentrations, calculating PK parameters, summaries of concentration-time data and plotting of individual concentration-time files for the intensive PK population.
- The Intensive Pharmacokinetic Parameter Population will be used for intensive PK parameter analyses
- If during clinical phase, 3 consecutive samples in any phase i.e.(Absorption, Distribution and Metabolism / Excretion) are found to be missing then data for that subject will not be included in PK and only the concentration data of that subject(s) will be presented
- The sparse pharmacokinetic population will be used for summarising PK concentrations.
- Listings will be based on the safety population, and only patients with a sample from the relevant dosing schedule will be presented in these listings.
- \* Prohibited medications that could decrease DTG or 3TC exposure will be identified as leading to exclusion from PK summaries and figures if they are ongoing at the visit at which the analysis is taking place. If a prohibited medication has a non-missing start and stop date before, say Week 24, then there will be no exclusion from PK analyses at the Week 24 analysis. Prohibited medications are defined as follows:
  - Carbamazepine
  - Oxcarbazepine
  - Phenobarbital
  - Phenytoin
  - Rifampin
  - Rifapentine
  - St. John's wort

Not applicable to analyses post Week 48.

## 13.6.6. Population Pharmacokinetic (PopPK)

# 13.6.7. Not applicable to analyses post Week 48. Viral Genotyping and Phenotyping

## Genotype

#### **Amino Acid Changes**

- A mutation is considered present whenever the encoded amino acid residue differs from the amino acid that would have been encoded by the wild-type (e.g., HXB2, NL43) comparator gene; e.g., Q148K.
- If the encoded amino acid is seen as a mixture of wild-type and mutant amino acid, e.g., Q148Q/K, the mutated amino acid is considered present at the codon of interest.
- If the encoded amino acid is seen as a mixture of two or more amino acids, which may or may
  not include wild type, e.g., Q184K/H or Q184K/H/Q, etc., for the purposes of calculating the
  number of mutated amino acids, only one mutation is considered to be present at the codon of
  interest.

## Representation of Amino Acid Changes

| Mutations | Amino acid change |
|---|---|
| T69S | Single mutation from amino acid 'T' (vendor reference) to 'S' (sample) at codon '69' |
| Q148H/K/R | Mixture of amino acid mutations 'H', 'K' and 'R' (sample) from amino acid 'Q' |
| | (vendor reference) at codon '148' |
| _69_1T | First insertion of amino acid 'T' (sample) at codon '69' |
| _69_2S | Second insertion of amino acid 'S' (sample) at codon '69' |
| _69_3S/A | Third insertion of a mixture of amino acids 'S' and 'A' (sample) at codon '69' |
| L74L/- | Mixture of amino acid 'L' (sample) and a deletion at codon '74' |
| V75- | Single deletion of amino acid (sample) at codon '75' |

#### **Resistance Associated Mutations**

• Known INI mutations associated with the development of resistance to RAL, EVG, BIC or DTG:

| Amino Acids in | H51Y, <b>T66A/I/K</b> ,L74M, <b>E92Q/V</b> /G, Q95K, T97A, G118R, <b>F121Y</b> , |
|---|---|
| HIV Integrase for | E138A/K, G140A/C/S, <b>Y143C/H/R/K/S/G/A, P145S</b> , <b>Q146P</b> , <b>S147G</b> , |
| Analysis | <b>Q148</b> N/ <b>H/K/R</b> , <b>V151</b> I/ <b>L</b> /A, S153F/Y, <b>N155H</b> /S/T, E157Q, G163R/K, |
| | S230R, R263K, L68V/I*, L74I*, E138T*, G193E* |

- Current listing includes INSTI mutations identified via the Stanford HIV Resistance database, or identified during in vitro passage of DTG, or as seen in a previous DTG studies in INI-experienced subjects (i.e. ING112574) and may be modified in case of additional substantive data availability.
- 2. INSTI mutations underlined and in bold have a maximum score of 60 for any INSTI drug in the Stanford database v8.9 (http://hiv.db.stanford.edu/DR/cgi-bin/rules\_scores\_hiv.db.cgi?class=INI last updated on 25 OCT 2019 and accessed on 17 FEB 2020); the rest have a maximum score <60.
- 3. This table is updated only by Virologists.
- Major resistance mutations to other classes (i.e., NRTI, NNRTI, PI) as defined by the International Antiviral Society-USA (IAS-USA). The most up to date IAS-USA guidelines available at the time of DBF will be used in the analysis.

## Genotype

## **Amino Acid Changes**

| Class | Mutations |
|---|---|
| NRTIs | M41L, K65R/E/N, D67N, 69 insert, K70E/R, L74V, Y115F, M184V/I, L210W, T215Y/F, K219Q/E; [A62V, V75I, F77L, F116Y, Q151M]* |
| NNRTIs | L100I, K101E/P, K103N/S, V106A/M, V108I, E138/A/G/K/Q/R, V179L, |
| | Y181C/I/V, Y188C/L/H, G190S/A, H221Y, P225H, F227C, M230I/L, |
| Pls | D30N,V32I , M46I/L, I47AV, G48V, I50V/L, I54V/M/L, Q58E, T74P, L76V, |
| | V82A/T/F/L/S, N83D, I84V, N88S,L90M |

Note: List generated from IAS\_USA Guideline, - 2019 2019 Resistance Mutations Update Volume 27 Issue 3, July/August 2019

\*Q151M Complex: Q151M usually occurs in combination with two or more of the following four accessory NRTI mutations A62V, V75I, F77L, and F116Y

## Susceptibility Scores

## Stanford Genotypic Susceptibility Score (GSS)

- To establish genotypic susceptibility to ART treatment, a genotypic sensitivity score will be calculated.
- Genotypic sensitivity to each drug will be assessed using the HIVdb, the Integrated Genotypic Resistance Interpretation System [Liu, 2006].
- In the HIVdb system, each HIV-1 drug resistance mutation is assigned a drug penalty score.
   The penalty scores for each drug resistance mutation are available at

NNRT1: https://nivdb.stanford.edu/dr-summary/mut-scores/NNRT1/

NRT1: https://hivdb.stanford.edu/dr-summary/mut-scores/NRT1/

PI: https://hivdb.stanford.edu/dr-summary/mut-scores/PI/

INST I: <a href="https://hivdb.stanford.edu/dr-summary/mut-scores/INST">https://hivdb.stanford.edu/dr-summary/mut-scores/INST</a>/. Scores for particular patterns of INST is are also available at <a href="https://hivdb.stanford.edu/dr-summary/pattern-scores/INST">https://hivdb.stanford.edu/dr-summary/pattern-scores/INST</a>//

The drug resistance estimate is obtained by adding together the penalty scores from all
mutations associated with resistance to that drug and then a numeric score (S-GSS) is applied
for each drug as shown below. The sum scores are titrated to fall within the following ranges:
susceptible, potential low-level resistance, low-level resistance, intermediate resistance, and
high-level resistance (see table below)

CCI - This section contained Clinical Outcome Assessment data collection questionnaire or indices, which are protected by third party copyright laws and therefore have been excluded.

 The HIVdb GSS will then be calculated for each subject defined as the sum of the resistance scores for each of their background drugs.

## Monogram Genotypic Susceptibility Score (GSS)

- Monogram GSS score will be reported in a listing, but will not be used for summary tables.
- Genotypic sensitivity to each drug will be assigned using the Monogram resistance score for each background drug provided in the database.

## Genotype

## **Amino Acid Changes**

For the DTG + 3TC arm a subject might have a M-GSS score of 0, 1 or 2, and in the TBR arm a subject might have a M-GSS score of 0, 1, 2, or 3 (since TBR is a 3-drug regimen).

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

## Phenotype

## Phenotypic Susceptibility

- Phenotypic susceptibility to all licensed antiretroviral drugs and DTG will be determined
  using PhenoSense HIV assays from Monogram Inc. and will be reported as fold change
  (FC) in IC50 relative to wild-type control virus NL4-3, i.e., FC of sample virus = IC50 of
  sample virus/IC50 of control virus.
- Since the maximum assay limit for FC for each ART varies from subject to subject, FC values that are greater than the maximum assay limit (e.g., '>100') will be interpreted as having a value equal to the smallest maximum assay limit for that ART in the study population for data analysis. Censored values will be presented 'as is' in the listings.
- Phenotypic susceptibilities will be categorised according to FC (based on Monogram PhenoSense assay). Clinical cut-offs (where available) or biological cut-offs by PhenoSense will be used to define the phenotypic susceptibility of background treatment.
- Replication capacity is generated as part of standard phenotypic assays.
- To establish susceptibility to background treatment, a phenotypic sensitivity score will be
  calculated. Phenotypic susceptibility to each drug in a subject's background regimen will
  be determined by applying drug-associated cutoffs as defined by the PhenoSense
  algorithm to the phenotypic fold resistance to that drug at a certain timepoint (e.g.,
  Screening or Baseline). A numeric score will be assigned to each background drug using
  two different methods: one with full sensitivity only (PSSf) and one with partial sensitivity
  included (PSSp).

#### PSS with Full Sensitivity Only (PSSf)

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

#### PSS with Partial Sensitivity Included (PSSp)

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

 Both PSSf and PSSp will be calculated separately for each subject defined as the sum of the resistance scores for each background drug.

| Drug | Abbreviation | Class | PhenoSense cutof |
|-----------------|--------------|-------|--------------------------|
| Abacavir | ABC | NRTI | (4.5 − 6.5) <sup>a</sup> |
| Lamivudine | 3TC | NRTI | 3.5 a |
| Didanosine | ddl | NRTI | (1.3 – 2.2) a |
| Stavudine | d4T | NRTI | 1.7 a |
| Zidovudine | AZT (ZDV) | NRTI | 1.9 |
| Emtricitabine | FTC | NRTI | 3.5 |
| Tenofovir | TDF | NRTI | (1.4 – 4) a |
| Delavirdine | DLV | NNRTI | 6.2 |
| Efavirenz | EFV | NNRTI | 3 |
| Nevirapine | NVP | NNRTI | 4.5 |
| Etravirine | ETR | NNRTI | (2.9-10)a |
| Rilpivirine | RPV | NNRTI | 2.0 |
| Fosamprenavir/r | FPV/r | PI | (4-11)a |
| Atazanavir/r | AT V/r | PI | 5.2ª |
| Indinavir/r | IDV/r | PI | 10 a |
| Lopinavir/r | LPV/r | PI | (9 – 55) a |
| Nelfinavir | NFV | PI | 3.6 |
| Saquinavir/r | SQV/r | PI | (2.3 – 12) a |
| Tipranavir/r | TPV/r | PI | (2 – 8) a |
| Darunavir/r | DRV/r | PI | (10 – 90) a |
| Ritonavir | RTV | PI | 2.5 |
| Enfuvirtide | T20 | FI | 6.48 |
| Raltegravir | RAL | INI | 1.5 |
| Elvitegravir | EVG | INI | 2.5 |
| Dolutegravir | DTG | INI | (4-13) a |
| Bictegravir | BIC | INI | (2.5-10) |

a. clinical cutoff (lower cutoff - higher cutoff)

## Phenotypic Susceptibility Score (PSS)

## Net Assessment and Overall susceptibility of ARTs

- Net assessment is an assessment of antiviral activity of ARTs using both genotypic
  and phenotypic test results interpreted through a proprietary algorithm (from Monogram
  Biosciences) and provides the overall susceptibility of the drug (Note: partially sensitive
  and resistant calls are considered resistant in this analysis).

## Decision tree approach for Monogram resistance data analyses

- We might have resistance data that come from mixed datasets: PSGT, PSIN, GSIN (primary assays) vs PSGT+IN (secondary assay)
- If one of the primary assay does not work for a specific timepoint, we might report the
  secondary assay if data is available. If all primary assays for a specific timepoint work
  then we report primary. For example, for baseline if the same assay section (PSGT,
  PSIN, GSIN) worked then we report primary. If at least one of PSGT or PSIN or GSIN
  didn't work then we report secondary PSGT+IN.
- Secondary assay testing results might not always be available.

## Background:

- DNA GenoSure Archive only provides geno data for PRO/RT and Integrase
- PSGT provides both geno and pheno data for PRO/RT (NRTI and NNRTI) only
- PSIN Provides pheno data on Integrase only
- GSIN Provides geno data on Integrase only
- PSGT+IN Secondary assay used if PSGT or GSIN assay fails; it provides both geno and pheno data on PRO, RT and Integrase

#### 13.6.8. Health Outcomes

## European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L)

The EQ-5D is a quality of life instrument that provides a EQ-5D-5L Utility Score and the EQ Visual Analogue scale (EQ VAS)

#### EQ-5D-5L

- The descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression with five levels for each dimension from level 1 = to level 5 =
- The number of possible health states is 5<sup>5</sup> = 3125.
- The health state is defined by combining the levels of answers from each of the 5 questions.
- Each health state is referred to in terms of a 5-digit code. For example, state 11111 indicates no
  problems on any of the 5 dimensions, while state 12345 indicates no problems with mobility,
  slight problems with washing or dressing, moderate problems with doing usual activities, severe
  pain or discomfort and extreme anxiety or depression.
- The health state 5-digit code is translated into the utility score, which is valued up to one (representing perfect health) with lower values meaning worse state, according to the methodology described in Devlin, 2016, Section 3.4. The UK values set described in Section 3.4 will be used for all subjects regardless of their country origin.
- The numerals 1-5 have no arithmetic properties and should not be used as a cardinal score.
- Ambiguous values (e.g. 2 boxes are ticked for a single dimension) should be treated as missing values.
- Any missing values should be imputed using LOCF.
- In Late switch Phase, as there is data collected at only one timepoint post-switch for TBR arm, the LOCF method will not be used. At W196 results will be presented on observed data

#### EQ visual Analogue scale (EQ VAS) 'Thermometer'

- Self-rated current health status
- Ranges from 0 (CCC)
  ) to 100 (CCC)

## Willingness to switch survey

- Assess the reason(s) for their participation and facilitate an understanding of subject's willingness to switch
- A single item question prior to randomisation.
- 7 reasons for willingness to participate in a clinical study where the current HIV medication may be switched check all that apply
- Any missing values will remain missing

## 13.6.9. Cut-off date for protocol deviations

#### Cut-off date

The following rules should be used to calculate cut-off date for protocol deviations up to and including Week 24:

- For subjects who have Week 24 viral load date (cut-off 1):
  - cut-off = Week 24 viral load date (used for snapshot algorithm) from LB (laboratory) dataset, or date of re-test date if patient had a re-test
- For subjects who do not have Week 24 viral load date (cut-off 2):
  - cut-off date = the earliest of (Day of Study Discontinuation from DS, date of Withdrawal Visit from SV, Study day of permanent treatment discontinuation from EX (for subjects randomised to DTG + 3TC) or CM (for patients randomised to TBR), study treatment start date + 210\*-1).

\*upper bound of week 24 window

Additional Statistical Programming Checks to identify 'Subjects with study withdrawal due to a reason of "Protocol Deviation" (as recorded in the eCRF) at or prior Week 24' will be performed.

- Consider subjects that have discontinued from the study prior or at Week 24 with 'Protocol deviation' as a reason in DS (study discontinuation).
- Cut-off date (cut-off 3):
- For subjects who have Week 24 viral load date -> cut-off = Week 24 viral load date (used for snapshot algorithm) from LB (laboratory) dataset.
- For subjects who withdrawn before Week 24 Snapshot HIVRNA sample taken or if missing data during week 24 window but on study-> cut-off = IP start date + 210\* - 1
- Compare the PD occurrence date (Day of Study Discontinuation from DS) to cut-off date (see paragraph above, please note: cut-off rules 1 and 2 defined above do not apply here)

 If cut-off date ≥ PD occurrence date, then deviations will result in exclusion from the per protocol set.

\*upper bound of week 24 window

Similar rules will be followed for Week 48, 96, and 144 will be detailed in a separate Protocol Deviation specification document. Please refer to latest version of the Protocol Deviation specification document prior to the analysis for full details of protocol deviation identification,

#### 13.6.10. PK Data

Not applicable to analyses post Week 48.

Below Limit of Quantification (BLQ) concentrations from any of the sparse PK samples will be set to missing, regardless of the week of collection.

## 13.6.11. eCRF Baseline Third Agent Class Determination

Baseline third agent will be determined as the third agent ingredient:

- still being taken at randomisation for TBR patients
- discontinued immediately prior to randomisation for DTG + 3TC patients.

## 13.7. Appendix 7: Reporting Standards for Missing Data

## 13.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject study completion (i.e. as specified in the protocol) was defined as: Randomly assigned to either treatment group, completed the Late Switch Phase at the Week 200 visit, and did not enter the Continuation Phase; |
| | Subjects randomised to either treatment group, completed the Randomised Late Switch Phase at the Week 200 visit, entered and completed the Continuation Phase, defined as remaining on study until: |
| | <ul> <li>DTG and 3TC FDC tablet is locally approved for use as a 2-drug<br/>regimen, and available through public health services or through the<br/>subject's usual health insurance payer, or</li> </ul> |
| | <ul> <li>the subject no longer derives clinical benefit, or</li> </ul> |
| | o the subject meets a protocol-defined reason for discontinuation, or |
| | o development of the DTG plus 3TC dual regimen is terminated. |
| | <ul> <li>Withdrawn subjects will not be replaced in the study.</li> <li>All available data from subjects who were withdrawn from the study will be listed.</li> </ul> |

## 13.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data are not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data are excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be</li> </ul> |
| Snapshot | <ul> <li>missing data and should not be displayed as such.</li> <li>In the Snapshot dataset, subjects without HIV-1 RNA data in the assessment window for the visit of interest (due to missing data or discontinuation of IP prior to the visit window) are classified as non-responders in the derivation of the proportion of subjects with HIV-1 RNA &lt; 50 c/mL (or &lt;400 c/mL). The nature of this missing data will be further classified in Snapshot summaries as either 'Virologic Failure' or 'No Virologic Data at Week X'; see Section 13.11 for full details. Further details of missing data as a result of COVID-19 and Snapshot sensivity analyses relevant to analyses at Week 96, Week 144 and W196 can be seen in Section 13.14.1.</li> </ul> |
| Element | Reporting Detail |
|---|---|
| LOCF | <ul> <li>In the LOCF dataset, missing values will be carried forward from the previous,<br/>non-missing available on-treatment assessment.</li> </ul> |
| Lipid LOCF | <ul> <li>If subjects initiate serum lipid-lowering agents Post-baseline, then the last available fasted On-treatment lipid values prior to the initiation will be used in place of future, observed On-treatment values.</li> <li>Imputation will continue even if the subject discontinues the lipid-lowering agent.</li> <li>Missing assessments will not be imputed.</li> <li>Subjects on lipid-lowering agents at baseline will be excluded from this dataset. This dataset will be used for all summaries of lipids data.</li> </ul> |
| Observed<br>Case (OC) | <ul> <li>This dataset uses only the data that is available at a particular timepoint, with no<br/>imputation for missing values.</li> </ul> |
| Lipid W196 | <ul> <li>If subjects initiate serum lipid-lowering agents Post-baseline/LS baseline, then the subsequent values will be set to missing.</li> <li>Subjects on lipid-lowering agents at baseline/LS baseline will be excluded from this dataset</li> <li>The observed case dataset will be used for all summaries of lipids data.</li> </ul> |

## 13.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Partial dates will be displayed as captured in subject listing displays.</li> </ul> |
| Exposure | <ul> <li>If study treatment stop date is missing, then for the purposes of calculating exposure, it will be imputed using the date of last visit or the recorded date of withdrawal/completion whichever is earlier.</li> <li>Partially Missing Stop Day: Last day of the month or last month of the year will be used, unless this is after the study completion date or withdrawal date; in this case the earliest of the two dates will be used. Note Study Treatment DTG+3TC is recorded on the Study Treatment CRFs and TBR treatment is recorded on the CONART CRFs.</li> </ul> |
| Adverse<br>Events and<br>Clinical Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE and Clinical Event start and end dates; that is, the day of the month may be missing: <ul> <li>If the full date cannot be ascertained, the following conventions will be applied for calculating the time to onset and the duration of the event: Completely missing dates: (i.e. no year specified) will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> <li>Partially Missing Start Day: First day of the month or first month of the year will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: T reatment States and Phases</li> <li>Partially Missing Stop Day: Last day of the month or last month of the year will be used, unless this is after the stop date of study treatment,</li> </ul> </li> </ul> |

| Element | Reporting Detail |
|---|---|
| | data cut off date or withdrawal date; in this case the earliest of the three dates will be used. The recorded partial date will be displayed in listings. |
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, the first day of the month will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, last day of the month will be used for the day and 'Dec' will be used for the month.</li> <li>For medications recorded in the eCRF as prior ART, the earlier of this imputed date or the day before IP start will be used.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 13.8. Appendix 8: Values of Potential Clinical Importance

| Element | Reporting Detail |
|---|---|
| Laboratory | The DAIDS grading for severity of laboratory toxicities and clinical adverse |
| Values and | events is included in the protocol. |
| Adverse<br>Events | The central laboratory will flag lab parameter toxicities directly in the provided datasets. |

## 13.9. Appendix 9: Population Pharmacokinetic (PopPK) Analyses

Not applicable to analyses post Week 48.

### 13.10. Appendix 10: Time to Event Details

### 13.10.1. TRDF Detailed Steps

### **TRDF Detailed steps**

For studies that have a Late Switch or Continuation Phase, ensure only data pertinent to the analysis is included, see study RAP for definition of Treatment Phase.

The steps below are for the derivation of TRDF at specific timepoints when the upper bound of the analysis window is used as a cut-off i.e. for the table only.

Randomised Period denotes period where subjects are still on their randomised treatment, prior to late switch of study treatment. This is also irrespective of blinding. Hence, Randomised Period also refers to Early Switch Phase.

Final step of the derivation is made in following order:

- [1] When one EVENT (1.2, 2.2, 3.2, 4.2) criterion is satisfied, select. In situations where more than one EVENT criteria satisfied, select the earliest event. If the earliest event date satisfies more than one criteria (e.g. subject had CVW and discontinuation), select CVW.
- [2] When one CENSOR (1.1, 2.1, 3.1, 4.1, 5.x) criterion is satisfied, select. Else in situations where more than one CENSOR criteria satisfied, select the latest censor day. If the latest event date satisfies more than one criteria, apply the ordering below.

| Condition | Censor<br>Status | Event Description/AVAL |
|---|---|---|
| 1. Subjects met CVW event criteria during the randomized period. | | |
| (Based on derived CVW confirmed prior to cut-off used for the analysis) | | |
| Then set <b>tempAVAL</b> = Study Day of first elevation immediately preceding CVW | | |
| 1.1 CVW event date is after the upper bound of the analysis visit window | CNSR=1 | EVNTDESC=Censored due to data cutoff. |
| i.e tempAVAL > upper bound of the analysis visit window for Week X | | AVAL=Upper bound of analysis visit window. |
| 1.2 CVW event date is on or before the upper bound of the analysis visit window | CNSR=0 | EVNTDESC=CVW. AVAL= tempAVAL. |
| i.e tempAVAL $\leq$ upper bound of the analysis visit window for Week X | | |

| TRDF Detail | ed steps | |
|---|---|---|
| 2. Subjects with study withdrawal due to treatment related adverse events during the randomized period | | |
| (defined as subjects that have reason for withdrawal =AE on disposition page and that the subject has at least one AE that is considered both: (i) drug related (AEREL=Y) and (ii) results in withdrawal from study (AEWD=Y)) | | |
| Then set <b>tempAVAL</b> = Earliest of (Day of Study Discontinuation [from Disposition page]), date of Withdrawal Visit [from Study Visit domain], Study day of permanent treatment discontinuation [from Exposure domain (for DTG + 3TC subject) or Concomitant Medication domain (for TBRsubjects)]). Assumption: Study day of permanent treatment discontinuation is included in the definition to account for cases where discontinuation information is recorded later. This is a conservative approach consistent with treatment discontinuation | | |
| preceding withdrawal. 2.1 Study withdrawal is after the upper | CNSR=1 | EVNTDESC=Censored due |
| bound of the analysis visit window | | to data cutoff. |
| i.e tempAVAL > upper bound of the analysis visit window | | AVAL=Upper bound of analysis visit window. |
| 2.2 Study withdrawal is on or before the upper bound of the analysis visit window i.e tempAVAL ≤ upper bound of the analysis visit window | CNSR=0 | EVNTDESC=Study Withdrawal Due to Treatment Related AE. AVAL= tempAVAL |
| 3: Subjects met protocol defined stopping criteria during the randomized period., | | |
| (Based on disposition page) | | |
| Then set <b>tempAVAL</b> =Earliest of (Day of Study Discontinuation [from Disposition page]), date of Withdrawal Visit [from Study Visit domain], Study day of permanent treatment discontinuation [from Exposure domain (for DTG + 3TC subject) | | |

| TRDF Detailed steps | | |
|---|---|---|
| or Concomitant Medication domain (for TBRsubjects)]). | | |
| 3.1 Protocol defined stopping criteria were met after the upper bound of the analysis visit window i.e tempAVAL > upper bound of the analysis visit window | CNSR=1 | EVNTDESC=Censored due to data cutoff. AVAL=Upper bound of analysis visit window. |
| 3.2 Protocol defined stopping criteria were met on or before the upper bound of the analysis visit window i.e tempAVAL ≤ upper bound of the analysis visit window | CNSR=0 | EVNTDESC=Study Withdrawal Due to Protocol Defined Criteria. AVAL=tempAVAL |
| 4: Subjects with study withdrawal due to lack of efficacy during the randomized period. | | |
| (Based on disposition page) | | |
| Then set <b>tempAVAL</b> = Earliest of (Day of Study Discontinuation [from Disposition page]), date of Withdrawal Visit [from Study Visit domain], Study day of permanent treatment discontinuation [from Exposure domain (for DTG + 3TC subject) or Concomitant Medication domain (for TBRsubjects)]). | | |
| 4.1 Study withdrawal is after the upper bound of the analysis visit window | CNSR=1 | EVNTDESC=Censored due to data cutoff. |
| i.e tempAVAL > upper bound of the analysis visit window | | AVAL=Upper bound of analysis visit window. |
| 4.2 Study withdrawal is on or before the upper bound of the analysis visit window i.e tempAVAL ≤ upper bound of the analysis visit window | CNSR=0 | EVNTDESC=Study Withdrawal Due to Lack of Efficacy AVAL= tempAVAL |
| If none of the above conditions met | | |
| 5: Subjects with study withdrawal for other reasons during the randomized period. (Based on disposition page) | | |

| TRDF Detailed steps | | |
|---|---|---|
| Then set <b>tempAVAL</b> = Earliest of (Day of Study Discontinuation [from Disposition page]), date of Withdrawal Visit [from Study Visit domain], Study day of permanent treatment discontinuation [from Exposure domain (for DTG + 3TC subject) or Concomitant Medication domain (for TBRsubjects)]). 5.1 Study withdrawal is after the upper | CNSR=1 | EVNTDESC=Censored due |
| i.e tempAVAL > upper bound of the analysis visit window | | to data cutoff. AVAL=Upper bound of analysis visit window. |
| 5.2 Study withdrawal is on or before the upper bound of the analysis visit window i.e tempAVAL ≤ upper bound of the analysis visit window | CNSR=1 | EVNTDESC=Censored due to Study Discontinuation for Other Reasons. AVAL=tempAVAL |
| 6: Subject completed the randomized period of the study. (Based on disposition page) | CNSR=1 | EVNTDESC= Censored as completed the Randomized Period. AVAL= Date of end of Treatment Phase |
| 7: Subject is ongoing in the study during the randomized period and have not yet completed the randomized period | CNSR=1 | EVNTDESC= Censored due to data cutoff. AVAL=Upper bound of analysis visit window. |
| Assumption: this will only be in cases where the reporting effort/analysis is performed midway through the randomized period | | |

### 13.10.2. TRDF Detailed Steps for the Kaplan-Meier plot

### TRDF Detailed steps

### The steps beloware for the derivation of TRDF overall i.e. for the Kaplan-Meier plot only.

Final step of the derivation is made in following order:

- [1] When one EVENT (conditions 1-4) criterion is satisfied, select. In situations where more than one EVENT criteria satisfied, select the earliest event. If the earliest event date satisfies more than one criteria (e.g. subject had CVW and discontinuation), select CVW.
- [2] When one CENSOR (conditions 5.x) criterion is satisfied, select. Else in situations where more than one CENSOR criteria satisfied, select the latest censor day. If the latest event date satisfies more than one criteria, apply the ordering below.

| Condition Censor Event Description/AVA | | |
|---|---|---|
| Condition | Status | Event Description/AVAL |
| Subjects met CVW event criteria during the randomized period. (Based on derived CVW confirmed prior to cut-off used for the analysis) | CNSR=0 | EVNTDESC=CVW. AVAL=Study Day of first elevation immediately preceding CVW. |
| 2. Subjects with study withdrawal due to treatment related adverse events during the randomized period (defined as subjects that have reason for withdrawal =AE on disposition page and that the subject has at least one AE that is considered both: (i) drug related (AEREL=Y) and (ii) results in withdrawal from study (AEWD=Y)) | CNSR=0 | EVNTDESC=Study Withdrawal Due to Treatment Related AE. AVAL=Earliest of (Day of Study Discontinuation [from Disposition page]), date of Withdrawal Visit [from Study Visit domain], Study day of permanent treatment discontinuation [from Exposure domain]). |
| 3: Subjects met protocol defined stopping criteria during the randomized period., (Based on disposition page) | CNSR=0 | EVNTDESC=Study Withdrawal Due to Protocol Defined Criteria. AVAL=Earliest of (Day of Study Discontinuation [from Disposition page]), date of Withdrawal Visit [from Study Visit domain], Study day of permanent treatment discontinuation [from Exposure domain]). |
| 4: Subjects with study withdrawal due to lack of efficacy during the randomized period. (Based on disposition page) | CNSR=0 | EVNTDESC=Study Withdrawal Due to Lack of Efficacy |

| TRDF Detailed steps | | |
|---|---|---|
| If none of the above conditions met | | AVAL= Earliest of (Day of Study Discontinuation [from Disposition page]), date of Withdrawal Visit [from Study Visit domain], Study day of permanent treatment discontinuation [from Exposure domain]) |
| 5: Subjects with study withdrawal for other reasons on or before the end of randomized period. (Based on disposition page) | CNSR=1 | EVNTDESC=Censored due to Study Discontinuation for Other Reasons. AVAL=Earliest of (Day of Study Discontinuation [from Disposition page]), date of Withdrawal Visit [from Study Visit domain], Study day of permanent treatment discontinuation [from Exposure domain]) |
| 6: Subject completed the randomized period of the study. (Based on disposition page) | CNSR=1 | EVNTDESC= Censored as completed the Randomized Period. AVAL= Date of completion of randomized study period |
| 7: Subject is ongoing in the study during the randomized period and have not yet completed the randomized period | CNSR=1 | EVNTDESC= Ongoing in the Study. AVAL=Last visit date |

- 1. Notes:
- 2. Randomised Period = Randomised Early Switch Phase
- 3. Efficacy visit windows should be used throughout for the upper bound of the analysis visit window
- 4. Subjects are considered to have completed the randomised period if they completed the Early Switch Phase.
- 5. By definition, a subject must be on-treatment for a CVW to be recorded therefore inclusion of study date of treatment discontinuation in the derivation is not required
- 6. EVNTDESC, AVAL & CNSR variables created for the following timepoints:
- 7. Week 24, 48, 96, 144 for the table analysis
- 8. Overall for the Kaplan-Meier plot

### 13.10.3. ERDF Detailed Steps

Similar algorithm will be applied for ERDF analyses and Kaplan-Meier figure, where condition 2 and 3 in Section 13.10.1 and Section 13.10.2 will not be considered.

### 13.11. Appendix 11: Snapshot

#### **Detailed Algorithm Steps**

### **Detailed steps**

Please note that the following scenarios will NOT be penalized Per Snapshot algorithm (i.e. please excluding these scenarios from **Condition** 1-4).

- Dose reduction, dropping a component, or change in formulation (e.g. 'Tivicay + Kivexa' to 'Triumeq' with the identical ingredients)
- Permitted Change (if a decision date is not collected in eCRF) / decision to permitted change is made prior to/on the first on-treatment viral load result
- Permitted change is made after the first on-treatment viral load result AND last on-treatment viral load prior to/on the date of change is <50 c/mL</li>
- Note: The only protocol-permitted substitutions are as follows:
  - A switch from a PI boosted with RTV to the same PI boosted with cobicistat is allowed.
  - A switch from a PI boosted with cobicistat to the same PI boosted with RTV is allowed.

Note the same process will be mapped out for Week 24, Week 96, Week 144 and Week 196

Please refer to Section 13.14.1 for further details of Snapshot modifications in presence of COVID-19 missing data (relevant to analyses at Week 96, Week 144 and Week 196).

| Condition | Response | Reasons |
|---|---|---|
| ('Week 48' indicates Week 48 window) | | |
| 1. If <i>non-permitted</i> change in background therapy <i>prior to</i> Week 48 | HIV1-RNA<br>≥ 50 | Change in background therapy |
| 2. If <i>permitted</i> change in background therapy <i>prior to</i> Week 48 AND the latest on-treatment VL prior to/on the date of change is $\geq 50$ c/m [a] | HIV1-RNA<br>≥ 50 | Change in background therapy |
| 3: If <i>non-permitted</i> change in background therapy <i>during</i> Week 48 | | |
| <ul> <li>Last on-treatment VL during Week 48 prior<br/>to/on the date of change ≥ 50 c/mL</li> </ul> | HIV1-RNA<br>≥ 50 | Data in window not below 50 |
| • Last on-treatment VL during Week 48 prior to/on the date of change <50 c/mL | HIV1-RNA<br>< 50 | |

| <ul> <li>No VL during Week 48 prior to/on the date<br/>of change</li> </ul> | HIV1-RNA<br>≥ 50 | Change in background therapy |
|---|---|---|
| 4: If <i>permitted</i> change in background therapy <i>during</i> Week 48 AND the last on-treatment VL prior to/on the date of change is $\geq 50$ c/mL [a] | | |
| 4.1 this last on-treatment VL occurs prior to Week 48 | HIV1-RNA<br>≥ 50 | Change in background therapy |
| 4. 2 this last on-treatment VL occurs during Week 48 but prior to/on the date of change | HIV1-RNA<br>≥ 50 | Data in window not below 50 |
| 5: If none of the above conditions met | | |
| 5.1 VL available during Week 48 | | |
| • Last on-treatment VL during Week 48 ≥ 50 c/mL | HIV1-RNA<br>≥ 50 | Data in window not below 50 |
| Last on-treatment VL during Week 48 <50 c/mL | HIV1-RNA<br>< 50 | |
| b. No VL during Week 48 | | |
| i. if subjects still on study (i.e. IP has not been permanently stopped up to Week 48) | No virologic<br>data at<br>Week 48<br>Window | On study but<br>missing data in<br>window |
| ii. If subjects withdraw before/during Week 48 due to | | |
| 1. Safety reasons (e.g. AE/death, liver chemistry stopping criteria, renal toxicity withdrawal criteria, QTc withdrawal criteria et al, as recorded in eCRF Study Conclusion form) | | Disc due to<br>AE/death |
| 2. Non-safety related reasons (e.g. Lack of efficacy, protocol deviation, withdrew consent, loss to follow-up, study closed/terminated, investigator discretion et al, as recorded in eCRF Study Conclusion Form) | | |

| Last on-treatment VL <50 c/mL OR no<br>on-treatment VL available during study | No virologic<br>Data at<br>Week 48<br>Window | Disc for other reasons |
|---|---|---|
| • Last on-treatment $VL \ge 50$ c/mL AND withdrawal due to Lack of efficacy | HIV1-RNA<br>≥ 50 | Disc. for lack of efficacy |
| <ul> <li>Last on-treatment VL ≥ 50 c/mL AND<br/>withdrawal due to all other non-safety<br/>related reasons</li> </ul> | HIV1-RNA<br>≥ 50 | Dis. for other reason while not below 50 |

[a]: Excluding permitted change in background therapy where change or decision to change is made prior to/on the first on-treatment viral result

### Examples from FDA guidance

#### Data in Window

Virologic outcome should be determined by the last available measurement while the patient is on treatment and continued on trial within the time window:

• HIV-RNA = 580 copies/mL at Day 336, HIV-RNA below 50 copies/mL on Day 350. This should be categorized as HIV-RNA below 50 copies/mL.

#### No Data in Window

Discontinued study due to Adverse Event or Death:

- Any patient who discontinues because of an AE or death before the window should be classified as *Discontinued due to AE or Death* (as appropriate), regardless of the HIV-RNA result, even if the HIV-RNA is below 50 copies/mL at the time of discontinuation.
- However, if a patient has an HIV-RNA value in the time window and also discontinues in the time window, the viral load data should be used to classify the patient's response.
   This is the Virology First hierarchy:
  - a. HIV-RNA below 50 copies/mL at Day 336 and discontinues because of AE or even dies on Day 360 — this person is categorized as having HIV-RNA below 50 copies/mL.
  - b. HIV-RNA is 552 copies/mL on Day 336 and the patient discontinues on Day 360, the patient is categorized as having HIV-RNA greater than or equal to 50 copies/mL.

#### Discontinued for Other Reasons:

- Only patients who have achieved virologic suppression can be counted as *Discontinued* for Other Reasons.
- If a patient discontinues the study before the window because of *lack of efficacy* then
  the patient should be included in the HIV-RNA greater than or equal to 50 row and not in
  the Discontinued for Other Reasons row.

- If a patient discontinues because of subject withdrew consent and his or her HIV-1 RNA
  result at the time of discontinuation was equal to or above 50 copies/mL, then he or she
  should be categorized as HIV-RNA greater than or equal to 50 and NOT as
  Discontinued for Other Reasons.
- If a patient discontinued because of *Lost to Follow-Up* and the last HIV-RNA result was 49 copies/mL, then the patient can be categorized as Discontinued for Other Reasons.
- If patients changed background treatment not permitted by protocol— they should be considered an efficacy failure and captured in the HIV-RNA greater than or equal to 50 copies/mL row.

### On study but missing data in window:

- If there are no data during Days 294 to 377, but there is an HIV-RNA below 50 copies/mL on Day 380, this patient should be considered On Study but Missing Data in Window.
- If there are no data during Days 294 to 377, but there is an HIV-RNA equal to or above 50 copies/mL on Day 280, this patient also should be classified as On Study but Missing Data in Window.

#### Optimized Background Therapy Substitutions After Randomisation

- OBT substitutions (in-class or cross-class) permitted per protocol for documented toxicity reasons can be permitted on or before the first trial visit without penalty.
- If OBT substitutions for toxicity reasons occur after the first trial visit, then patients should be categorized as having HIV-RNA greater than or equal to 50 copies/mL if they have HIV-RNA above 50 copies/mL at the time of switch.

## 13.12. Appendix 12: Abbreviations & Trade Marks

### 13.12.1. Abbreviations

| Abbreviation | Description |
|---|---|
| A&R | Analysis and Reporting |
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| $CV_b/CV_w$ | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DOB | Date of Birth |
| DOV | Date of Visit |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| ERDF | Efficacy Related Discontinuation Failure |
| GSK | GlaxoSmithK line |
| GUI | Guidance |
| IA | Interim Analysis |
| ICH | International Conference on Harmonisation |
| IDMC | Independent Data Monitoring Committee |
| IDSL | - |
| IMMS | Integrated Data Standards Library International Modules Management System |
| IP IVINS | · · |
| | Investigational Product Intent-To-Treat |
| ITT<br>LOC | Last Observation Carries Forward |
| MMRM | Mixed Model Repeated Measures |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | |
| PK | Protocol Deviation Management Plan Pharmacokinetic |
| PP | Per Protocol |
| QC<br>QTcF | Quality Control Frederica's QT Interval Corrected for Heart Rate |
| RAMOS | Randomisation & Medication Ordering System |
| RAP | Reporting & Analysis Plan |
| SAC | Statistical Analysis Complete |
| | · |
| SDTM<br>SOP | Study Data Tabulation Model Standard Operation Procedure |
| | 1 |
| TAE | Therapeutic Area Tanafavin alafanamida fumarata |
| TAF | Tenofovir alafenamide fumarate |

| Abbreviation | Description |
|--------------|-------------------------------------------|
| TBR | TAF based regimen |
| TFL | Tables, Figures & Listings |
| TRDF | Treatment Related Discontinuation Failure |

### 13.12.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| Epivir |
| Tivicay |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| Monogram Inc |
| NONMEM |
| SAS |
| WinNonlin |

# 13.13. Appendix 13: Model Checking and Diagnostics for Statistical Analyses

### 13.13.1. Statistical Analysis Assumptions

| Endpoint(s) | Change from Baseline in bone/renal/inflammatory biomarkers, EQ5D, weight, BMI, lipids and HOMA-IR |
|---|---|
| Analysis | MMRM |

- Model assumptions will be applied, but appropriate adjustments maybe made based on the data.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- An unstructured covariance structure for the R matrix will be estimated by treatment group by specifying 'type=UN' and 'group=treat' on the REPEATED line.
  - o In the event that this model fails to converge, alternative correlation structures may be considered such as CSH or CS.
  - Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure.
- Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.

# 13.14. Appendix 14: COVID-19 Modified Analyses and Supportive Sensitivity Analyses

This section outlines the additional analyses that will be performed at Week 96 onwards to account for the effect of COVID-19.

### 13.14.1. Efficacy Analyses (Snapshot)

The main efficacy analysis remains that performed on the ITT-E analysis. Study Outcomes based on the main Table 2.4-Table 2.6 will be reported in line with the Modified Snaphot Algorithm (Section 13.14.1.2) that presents additional subcategories related to COVID-19 missing and intercurrent event data (otherwise top-level outcomes of >=50 c/mL, <50 c/mL and No Virologic Data remain unaffected). Summary tables to test for non-inferiority (Table 2.1-Table 2.3, Table 2.7, Table 2.8 and Table 2.34) will remain unchanged.

A supplemental analysis for study outcomes (Table 2.38) and treatment comparison of HIV-1 RNA >=50 c/mL endpoint (Table 2.36) and HIV-1 RNA <50 c/mL endpoint (Table 2.37) will be performed on the Efficacy Evaluable Population, which excludes subjects with no Week 96 data due to COVID-19. Subjects with no HIV-1 RNA recorded within the Week 96 analysis visit window will be excluded either as a result of discontinuation from the study due to COVID-19 as recorded on study conclusion page or still on-study but no Week 96 data as a result of COVID-19, as recorded in the protocol deviations log. (If COVID-19 is not recorded as a reason for discontinuation from study on the study conclusion page, then this may be captured from protocol deviations and/or AE page.) In the event that there is a higher rate of primary endpoint missing data observed than expected, an assessment will be made as to whether this analysis will be supplemented or replaced with an imputation-based analysis where subjects' last-on treatment HIV-1 RNA prior to Week 96 will be used in lieu of missing Week 96 HIV-1 RNA data as a result of COVID-19. Imputation will only be considered for subjects with missing data as a result of COVID-19 (i.e. discontinued due to COVID-19 or on study but missing data due to COVID-19). Following imputation, the Snapshot algorithm will be performed in the same way as described in Section 13.11, and Study Outcomes and non-inferority test outputs will be performed. The above supplemental analysis on Efficacy Evaluable Population performed at Week 144. The main Study Outcomes analyses for subjects with HIV-1 RNA <40 c/mL and HIV-1 RNA <40 c/mL and Target Not Detected based on ITT-E population in Table 2.31 and Table 2.35) will be reported in line with the Modified Snapshot Algorithm (Section 13.14.1.2, which presents additional subcategories related to COVID-19 missing and intercurrent event data. The corresponding analyses for the comparison in proportions of subjects with HIV-1 RNA <40 c/mL and HIV-1 RNA <40 c/mL and Target Not Detected (Table 2.27 and Table 2.28, respectively) will remain unchanged. A supplemental analysis for HIV-1 RNA <40 c/mL and Target Not Detected based on the Evaluable Efficacy Population, which excludes subjects with no Week 96 data due to COVID-19 as above. Study Outcomes (Table 2.39) and test for comparison (Table 2.40) will be reported.

Refer to shells document for further details.

### 13.14.1.1. Change in Study Treatment

Given that subjects with any changes in study treatment should be withdrawn from study per protocol instructions, it is anticipated that there will be minimal (if any) changes in study treatment Snapshot outcomes. However, in the event of any unforeseen change in study treatment events then change in study treatment outcomes will be reported by COVID-19 and non-COVID-19 subcategories in line with steps 1-4 of the Modified Snapshot Algorithm rules as presented in Section 13.14.1.2.

### 13.14.1.2.Modified Snapshot Algorithm

The below Modified Snapshot Algorithm will be used to determine Snapshot outcomes taking into account COVID-19 related events. The Modified Snapshot Estimand still reports high-level categories (>=50 c/mL, <50 c/mL and No Virologic Data) in exactly the same way as the standard FDA Snapshot Algorithm in Section 13.11, however it reports additional subcategories to account for outcomes related to COVID-19.

| Condition | Response | Reasons |
|---|---|---|
| ( 'Week 48' indicates Week 48 window) | | |
| If <i>non-permitted</i> change in background therapy <i>prior to</i> Week 48 (Non-COVID-19 switch) | HIV1-RNA ≥<br>50 | Change in<br>background therapy<br>(Non- COVID-19<br>related) |
| 1.2 If <b>non-permitted</b> change in background therapy <b>prior to</b> Week 48 (COVID-19 switch) | HIV1-RNA ≥<br>50 | Change in background therapy (COVID-19 related) |
| 2.1 If <b>permitted</b> change (not related to COVID-19) in background therapy <b>prior to</b> Week 48 AND the latest on-treatment VL prior to/on the date of change is ≥ 50 c/mL | HIV1-RNA ≥<br>50 | Change in background therapy (Non- COVID-19 related) |
| 2.2 If <b>permitted</b> change (related to COVID-19) in background therapy <b>prior to</b> Week 48 AND the latest on-treatment VL prior to/on the date of change is ≥ 50 c/mL | HIV1-RNA ≥<br>50 | Change in background therapy COVID-19 related) |
| If <i>non-permitted</i> change in background therapy<br>during Week 48 | | |
| <ol> <li>3.1 Last on-treatment VL during Week 48 prior<br/>to/on the date of change ≥ 50 c/mL</li> </ol> | HIV1-RNA ≥<br>50 | Data in window not below 50 |
| 3. 3.2 Last on-treatment VL during Week 48 prior to/on the date of change <50 c/mL | HIV1-RNA < 50 | |
| 4. 3.3.1 No VL during Week 48 prior to/on the date of change (non-COVID-19 related) | HIV1-RNA ≥<br>50 | Change in<br>background therapy<br>(Non- COVID-19<br>related) |
| 5. 3.3.2 No VL during Week 48 prior to/on the date of change (COVID-19 related) | HIV1-RNA ≥<br>50 | Change in background therapy (COVID-19 related) |

| Condition | | Response | Reasons |
|---|---|---|---|
| ( 'Week 48' indicates Week 48 window) | | | |
| We | nitted change in background therapy during sek 48 AND the last on-treatment VL prior on the date of change is ≥ 50 c/mL [a] | | |
| | this last on-treatment VL occurs prior to<br>Veek 48 (non-COVID-19 related switch) | HIV1-RNA ≥<br>50 | Change in background therapy (Non- COVID-19 related) |
| | this last on-treatment VL occurs prior to Veek 48 (COVID-19 related switch) | HIV1-RNA ≥ 50 | Change in background therapy COVID-19 related) |
| | s last on-treatment VL occurs during Week<br>8 but prior to/on the date of change | HIV1-RNA ≥<br>50 | Data in window not below 50 |
| | of the above conditions met | | |
| 5.1 VL | available during Week 48 | | |
| c/mL | ast on-treatment VL during Week 48 ≥ 50 | HIV1-RNA ≥<br>50 | Data in window not below 50 |
| c/mL | ast on-treatment VL during Week 48 <50 | HIV1-RNA <<br>50 | |
| 5.2 No | VL during Week 48 | | |
| | Participants unable to attend Week 48 visit due to COVID-19, but otherwise considered still on-study (i.e. The on-treatment period continues beyond the upper bound of Week 48 window. For example, for oral treatment, a participant with IP stop date+1> Day 378 of the upper bound of Week 48 window, would be considered 'on study' for Week 48 snapshot assessment) | No virologic<br>data at Week<br>48 Window | On study but missing data in window (COVID-19 related) |
| | If participants still on study but participant has missed visit not due to COVID-19 (i.e. The on-treatment period continues beyond the upper bound of Week 48 window. For example, for oral treatment, a participant with IP stop date+1> Day 378 of the upper bound of Week 48 window, would be considered 'on study' for Week 48 snapshot assessment) | No virologic<br>data at Week<br>48 Window | On study but missing<br>data in window<br>(Non- COVID-19<br>related) |
| 5.3.2 | If participants withdraw before/during Week 48 due to: | | |
| 5.3.2.1 | Non-COVID-19 Safety reasons (e.g. non-COVID-19 AE/death, liver chemistry stopping criteria, renal toxicity withdrawal criteria, QTc withdrawal criteria, as | No virologic<br>data at Week<br>48 Window | Disc. due to<br>AE/death<br>(Non- COVID-19<br>related) |

| Condition | Response | Reasons |
|---|---|---|
| ( 'Week 48' indicates Week 48 window) | | |
| recorded in eCRF Conclusion form where | | |
| related to pandemic not equal to 'Yes') | | D: 1 ( |
| 5.3.2.2 COVID-19 safety reasons eCRF (e.g. | No virologic | Disc. due to |
| AE/death resulting from COVID-19 as | data at Week | AE/death |
| recorded in the eCRF Conclusion form | 48 Window | (COVID-19 related) |
| where related to pandemic='Yes') | | |
| 5.3.2.3 Non-safety and non-COVID-19 related | | |
| reasons (e.g. Lack of efficacy, protocol | | |
| deviation, withdrew consent, loss to follow- | | |
| up, study closed/terminated, investigator | | |
| discretion et al, as recorded in eCRF Study | | |
| Conclusion Form and pandemic-related not | | |
| equal to 'Yes') | | |
| 5.3.2.3.1 Last on-treatment VL <50 c/mL OR no | No virologic | Disc. for other |
| on-treatment VL available during study | Data at Week | reasons |
| | 48 Window | (Non- COVID-19 |
| | | related) |
| 5.3.2.3.2 Last on-treatment VL ≥ 50 c/mL AND | HIV1-RNA ≥ | Disc. for lack of |
| withdrawal due to Lack of efficacy | 50 | efficacy |
| | | (Non- COVID-19 |
| | | related) |
| 5.3.2.3.3 Last on-treatment VL ≥ 50 c/mL AND | HIV1-RNA ≥ | Disc. for other reason |
| withdrawal due to all other non-safety related | 50 | while not below 50 |
| reasons | | (Non- COVID-19 |
| | | related) |
| 5.3.2.4 Non-safety and COVID-19 related reasons | | |
| (e.g. Withdrawal of consent, lack of efficacy, | | |
| protocol deviation, investigator discretion et | | |
| al. as recorded in eCRF Study Conclusion | | |
| Form and pandemic-related='Yes') | | |
| 5.3.2.4.1 Last on-treatment VL <50 c/mL OR no | No virologic | Disc. for other |
| on-treatment VL available during study | Data at Week | reasons |
| | 48 Window | (COVID-19 related) |
| 5.3.2.4.2 Last on-treatment VL ≥ 50 c/mL AND | HIV1-RNA ≥ | Disc. for lack of |
| withdrawal due to Lack of efficacy | 50 | efficacy |
| , | | (COVIĎ-19 related) |
| 5.3.2.4.3 Last on-treatment VL ≥ 50 c/mL AND | LII/A DNIA ~ | Dieg for other reces |
| | HIV1-RNA ≥<br>50 | Disc. for other reason while not below 50 |
| withdrawal due to all other non-safety related | 30 | (COVID-19 related) |
| reasons | | (סט אום- ופו פוריםוא סטן) |

### 13.15. Appendix 15: List of Data Displays

### 13.15.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|-------------|
| Study Population | 1.01 to 1.n | 1.01 to 1.n |
| Efficacy | 2.01 to 2.n | 2.01 to 2.n |
| Safety | 3.01 to 3.n | 3.01 to 3.n |
| Virology | 4.01 to 4.n | 4.01 to 4.n |
| Pharmacokinetic | 5.01 to 5.n | 5.01 to 5.n |
| Health Outcomes | 6.01 to 6.n | 6.01 to 6.n |
| Section | List | ings |
| ICH Listings | 1 t | 0 X |
| Other Listings | y t | 0 Z |

### 13.15.2. Mock Example Shell Referencing

Non-IDSL specifications will be referenced as indicated and if required example mockup displays provided in Appendix 16: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 13.15.3. Deliverables

| Delivery [Priority] [1] | Description |
|-------------------------|------------------------------------------------|
| DS [X] | During Study |
| IA SAC [X] | Interim Analysis Statistical Analysis Complete |
| SAC [X] | Final Statistical Analysis Complete |

#### NOTES

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort

### 13.15.4. Study Population Tables

Note that where the Deliverable column states 'All', this refers to all reporting efforts i.e. Weeks 24, 48, 96, 144, and 196.

Note: For W196 combined outputs (combining Early and Late Switch Phase outputs for DTG+3TC arm and Late Switch Phase for TBR arm), population presented in output header will be oveall Safety/ITTE/CVW/Viral Genotypic/Viral Phenotypic but Treatment Lable for Early Switch DTG+3TC as ES DTC+3TC and for Late Switch TBR arm as 'LS DTG+3TC'. For outputs on change from baseline summary or post-baseline events, Baseline for LS DTG+3TC should be labelled as 'LS Baseline'.

Note: For outputs which uses LS Baseline in the title or template add the footnote "LS Baseline - Baseline for LS DTG/3TC, the latest available pre-switch data". Also in any existing footnote for baseline replace "Baseline" with "Baseline"LS Baseline".

Note: For all outputs, Early Switch DTG+3TC and should be labelled as ES DTC+3TC and Late Switch TBR arm as 'LS DTG+3TC'.

Note: The following footnote should be added for all Listings' Note: TBR subjects are switched to DTG+3TC in Late Switch Phase from Week 148'

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | Disposition | | | | |
| 1.1. | ITT-E | ES1 | Summary of Subject Disposition for the Subject<br>Conclusion Record - Early Switch Phase | Not repeated Present the disposition by Overall Related to COVID-19 Not Related to COVID-19 | Weeks 24,<br>48, 96 and<br>144 |
| 1.101 | ITT-E | ES1 | Summary of Subject Disposition for the Subject Conclusion Record - DTG <u>+ 3TC</u> arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | Present the disposition by Overall Related to COVID-19 Not Related to COVID-19 | Week 196 |

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.2. | | | | No longer required | |
| 1.3. | ITT-E | ES4 | Summary of Subject Disposition at Each Study Epoch | | |
| 1.4. | All<br>Subjects<br>Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Not repeated | Weeks 24, 48,<br>96, 144 |
| 1.5. | All<br>Subjects<br>Screened | NS1 | Summary of Number of Subjects Enrolled by Country and Site ID | Not repeated | Weeks 24, 48,<br>96, 144 |
| 1.6. | ITT-E | POP_T1 | Summary of Reasons for Withdrawal by Visit- Early Switch Phase | No longer required | Weeks 24, 48,<br>96 |
| 1.601 | ITT-E | POP_T1 | Summary of Reasons for Withdrawal by Visit - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | Week 196<br>(including<br>W200) |
| Protoco | ol Deviation | | | | |
| 1.7. | ITT-E | DV1 | Summary of Important Protocol Deviations- Early Switch Phase | Not repeated | Weeks 24, 48,<br>96, 144 |
| 1.701 | ITT-E | DV1 | Summary of Important Protocol Deviations - DTG <u>+ 3TC</u> arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | Week 196<br>(including<br>W200) |
| 1.8. | ITT-E | DV1 | Summary of Protocol Deviations Leading to Exclusion from the Per-Protocol Population- Early Switch Phase | Not repeated | Weeks 24, 48,<br>96, 144 |

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Populat | ion Analyse | d | | | • |
| 1.9. | All<br>Subjects<br>Screened | SP1 | Summary of Study Populations | | All |
| 1.10. | | | | No longer required | |
| Demogr | aphic and B | aseline Chara | acteristics | <u>l</u> | |
| 1.11. | ITT-E | DM1 | Summary of Demographic Characteristics | Not repeated | Weeks 24, 48,<br>96, 144 |
| 1.1102 | LS-ITT-E | DM1 | Summary of Demographic Characteristics - TBR arm – Late Switch Phase | | Week 196 |
| 1.12. | All<br>Subjects<br>Screened | DM11 | Summary of Age Ranges | Not repeated | Weeks 24, 48,<br>96 |
| 1.13. | ITT-E | DM5 | Summary of Race and Racial Combinations | Not repeated | Weeks 24, 48,<br>96 |
| 1.14. | ITT-E | DM6 | Summary of Race and Racial Combinations Details | Not repeated | Weeks 24, 48,<br>96, 144 |
| 1.1402 | LS-ITT-E | DM6 | Summary of Race and Racial Combinations Details -<br>TBR arm – Late Switch Phase | | Week 196 |
| 1.15. | ITT-E | POP_T2 | Summary of Hepatitis Status at Entry | Not repeated | Weeks 24, 48,<br>96, 144 |

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.1502 | LS-ITT-E | POP_T2 | Summary of Hepatitis Status at Entry - TBR arm – Late Switch Phase | For Late switch Phase at study entry and any new event through W144 | Week 196 |
| 1.16. | ITT-E | CDC1 | Summary of CDC Classification of HIV Infection at Baseline | Not repeated | Weeks 24, 48,<br>96, 144 |
| 1.1602 | LS-ITT-E | CDC1 | Summary of CDC Classification of HIV Infection at Baseline - TBR arm - Late Switch Phase | | Week 196 |
| 1.17. | ITT-E | RF1 | Summary of HIV Risk Factors | Not repeated | Weeks 24, 48,<br>96, 144 |
| 1.1702 | LS-ITT-E | RF1 | Summary of HIV Risk Factors - TBR arm – Late Switch Phase | | Week 196 |
| 1.18. | ITT-E | POP_T3 | Summary of Screening Cardiovascular Risk<br>Assessments | Not repeated | Weeks 24, 48,<br>96, 144 |
| 1.1802 | LS-ITT-E | POP_T3 | Summary of Screening Cardiovascular Risk<br>Assessments - TBR arm – Late Switch Phase | Framingham risk score from W144. Add footnote to indicate this | Week 196 |
| 1.19. | ITT-E | POP_T4 | Summary of Distribution of CD4+ Cell Count (cells/mm^3) Results at Screening and Baseline | Not repeated | Weeks 24, 48,<br>96, 144 |
| 1.1902 | LS-ITT-E | POP_T4 | Summary of Distribution of CD4+ Cell Count (cells/mm^3) Results at LS Baseline - TBR arm – Late Switch Phase | | Week 196 |
| Prior an | Prior and Concomitant Medications, Medical Conditions | | | | |
| 1.20. | ITT-E | MH1 | Summary of Current Medical Conditions - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.2001 | ITT-E | MH1 | Summary of Current Medical Conditions - DTG <u>+ 3TC</u> arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | Week 196 |
| 1.21. | ITT-E | MH1 | Summary of Past Medical Conditions | Not repeated | Weeks 24, 48,<br>96, 144 |
| 1.2101 | LS-ITT-E | MH1 | Summary of Past Medical Conditions - TBR arm – Late<br>Switch Phase | | Week 196 |
| 1.22. | ITT-E | CM1 | Summary of Concomitant Medications by Ingredient AT C<br>Level 1- Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 1.2201 | ITT-E | CM1 | Summary of Concomitant Medications by Ingredient ATC Level 1 - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | Week 196<br>(including<br>W200) |
| 1.23. | ITT-E | CM8 | Summary of Concomitant Medication Ingredient Combinations - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 1.2301 | ITT-E | CM8 | Summary of Concomitant Medication Ingredient Combinations - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | Week 196<br>(including<br>W200) |
| 1.24. | ITT-E | CM1b | Summary of Concomitant Medications by Combination Term ATC Level 1- Early Switch Phase | Not repeated | Weeks 24, 48,<br>96, 144 |
| 1.2401 | ITT-E | CM1b | Summary of Concomitant Medications by Combination Term ATC Level 1 - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | Week 196<br>(including<br>W200) |

| Study P | opulation Ta | ables | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.25. | ITT-E | POP_T5 | Summary of Antiretroviral Therapy Stopped Prior to Screening | Not repeated | Weeks 24, 48,<br>96, 144 |
| 1.26. | ITT-E | POP_T5 | Summary of Antiretroviral Therapy Received at Screening | Not repeated | Weeks 24, 48,<br>96, 144 |
| 1.2602 | LS-ITT-E | POP_T5 | Summary of Antiretroviral Therapy Received at Screening - TBR arm – Late Switch Phase | | Week 196 |
| 1.27. | ITT-E | MH4 | Summary of Current Cardiac, Gastrointestinal,<br>Metabolism and Nutrition, Psychiatric, Renal and Urinary,<br>and Nervous System Conditions | Not repeated | Weeks 24, 48,<br>96, 144 |
| 1.2701 | ITT-E | MH4 | Summary of Current Cardiac, Gastrointestinal, Metabolism and Nutrition, Psychiatric, Renal and Urinary, and Nervous System Conditions - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | Week 196<br>(including<br>W200) |
| 1.28. | ITT-E | MH4 | Summary of Past Cardiac, Gastrointestinal, Metabolism and Nutrition, Psychiatric, Renal and Urinary, and Nervous System Conditions | Not repeated | Weeks 24, 48,<br>96, 144 |
| 1.2801 | LS-ITT-E | MH4 | Summary of Past Cardiac, Gastrointestinal, Metabolism and Nutrition, Psychiatric, Renal and Urinary, and Nervous System Conditions - DTG + 3TC arm (Early and Late Switch Phase) | | Week 196 |
| 1.29. | ITT-E | POP_T6 | Summary of Lipid Modifying Agent Use at Baseline | Not repeated | Weeks 24, 48,<br>96, 144 |

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.2902 | LS-ITT-E | POP_T6 | Summary of Lipid Modifying Agent Use at LS Baseline - TBR arm – Late Switch Phase | | Week 196 |
| 1.30. | ITT-E | POP_T6 | Summary of Lipid Modifying Agent Use Starting Post-<br>Baseline- Early Switch Phase | Not repeated | Weeks 24, 48,<br>96, 144 |
| 1.3001 | ITT-E | POP_T6 | Summary of Lipid Modifying Agent Use Starting Post-<br>Baseline - DTG + 3TC arm (Early and Late Switch<br>Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | Week 196<br>(including<br>W200) |
| 1.31. | ITT-E | POP_T7 | Summary of History of Depression and Anxiety at Baseline | Not repeated | Weeks 24, 48,<br>96, 144 |
| 1.3102 | LS-ITT-E | POP_T7 | Summary of History of Depression and Anxiety at LS Baseline - TBR arm – Late Switch Phase | LS Baseline – at study entry or through W144 | Week 196 |
| 1.32. | ITT-E | POP_T8 | Summary of Baseline Third Agent Class | Not repeated | Weeks 24, 48,<br>96, 144 |
| 1.3202 | LS-ITT-E | POP_T8 | Summary of Baseline Third Agent Class - TBR arm - Late Switch Phase | | Week 196 |
| 1.33. | ITT-E | NS1 | Summary of Number of Subjects Enrolled by Country and Site ID –ITT-E | Not repeated | Weeks 24, 48,<br>96 |
| 1.3302 | LS-ITT-E | NS1 | Summary of Number of Subjects Enrolled by Country and Site ID – TBR arm - Late Switch Phase | | W196 |
| 1.34. | ITT-E | POP_T9 | Summary of Number of Subjects Attending Nominal and Actual Analysis Visits - Early Switch Phase | Not repeated | Weeks 24, 48, 96 |
| 1.35. | | | | No longer required | |

| Study Po | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.36. | ITT-E | POP_T10 | Summary of Antiretroviral Therapy at Screening by Regimen | Not repeated | Weeks 24, 48,<br>96, 144 |
| 1.3602 | LS-ITT-E | POP_T10 | Summary of Antiretroviral Therapy at Screening by Regimen - TBR arm - Late Switch Phase | | W196 |
| 1.37. | ITT-E | POP_T11 | Summary of Distribution of Quantitative Plasma HIV-1 RNA Results at Baseline | Not repeated | 48, 96, 144 |
| 1.3702 | LS-ITT-E | POP_T11 | Summary of Distribution of Quantitative Plasma HIV-1<br>RNA Results at LS Baseline - TBR arm - Late Switch<br>Phase | | Week 196 |
| 1.38. | ITT-E | POP_T12 | Summary of Time since First Antiretroviral Therapy until Day 1 - Early Switch Phase | Not repeated | Week 24, 48,<br>96, 144 |
| 1.3802 | LS-ITT-E | POP_T12 | Summary of Time since First Antiretroviral Therapy until Day 1 - TBR arm - Late Switch Phase | | W196 |
| 1.39. | ITT-E | POP_T13 | Summary of Misrandomized Strata or Treatment | Not required | 48, 96, 144 |
| 1.40. | ITT-E | POP_T5 | Summary of On-Treatment Antiretroviral Therapy Starting after Day 1- Early Switch Phase | Not repeated | 48, 96, 144 |
| 1.4001 | ITT-E | POP_T5 | Summary of On-Treatment Antiretroviral Therapy Starting after Day 1 for DTG + 3TC arm (Early and Late Switch Phase) and Starting after switch for TBR arm (Late Switch Phase) | | Week 196<br>(including<br>W200) |
| 1.41. | ITT-E | POP_T5 | Summary of Antiretroviral Therapy Starting after Treatment Discontinuation- Early Switch Phase | Not repeated | 48, 96, 144 |

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.4101 | ITT-E | POP_T5 | Summary of Antiretroviral Therapy Starting after Treatment Discontinuation - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | Week 196<br>(including<br>W200) |
| 1.42. | ITT-E | POP_T10 | Summary of On-Treatment Antiretroviral Therapy Starting after Screening by Regimen-Early Switch Phase | Not repeated | 48, 96, 144 |
| 1.4201 | ITT-E | POP_T10 | Summary of On-Treatment Antiretroviral after Day 1 for DTG + 3TC arm (Early and Late Switch Phase) and after switch for TBR arm (Late Switch Phase) by Regimen | | Week 196<br>(including<br>W200) |
| 1.43. | ITT-E | POP_T10 | Summary of Antiretroviral Therapy Starting after Treatment Discontinuation by Regimen-Early Switch Phase | Not repeated | 48, 96, 144 |
| 1.4301 | ITT-E | POP_T10 | Summary of Antiretroviral Therapy Starting after Treatment Discontinuation by Regimen - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | Week 196<br>(including<br>W200) |
| 1.44. | ITT-E | DV1 | Summary of Important COVID-19 Protocol Deviations - Early Switch Phase | Not repeated | 96, 144 |
| 1.4401 | ITT-E | DV1 | Summary of Important COVID-19 Protocol Deviations - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | Week 196<br>(including<br>W200) |
| 1.45. | ITT-E | DV1 | Summary of Important non-COVID-19 Protocol Deviations - Early Switch Phase | Not repeated | 96, 144 |

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Populati<br>on | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.46. | ITT-E | PAN4 | Summary of COVID-19 Pandemic Visit Impacts - Early Switch Phase | Not repeated | 144 |
| 1.4601 | ITT-E | PAN4 | Summary of COVID-19 Pandemic Visit Impacts - DTG <u>+</u> 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | Week 196<br>(including<br>W200) |

# 13.15.5. Efficacy Tables

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Primary | Efficacy Anal | ysis | | | |
| 2.1. | ITT-E | EFF_T1 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA ≥ 50 c/mL at Week X – Snapshot Analysis - Early Switch Phase | No longer required | Weeks 24, 48,<br>96 and 144 |
| 2.2. | Per-<br>Protocol | EFF_T1 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA ≥ 50 c/mL at Week X – Snapshot Analysis - PP - Early Switch Phase | No longer required | Weeks 24, 48,<br>96 and 144 |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.3. | ITT | EFF_T1 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA ≥ 50 c/mL at Week X – Snapshot Analysis – ITT - Early Switch Phase | No longer required | Weeks 24, 48,<br>96 and 144 |
| 2.4. | ITT-E | TBC | Summary of Study Outcomes (Plasma HIV-1 RNA ≥ / < 50 c/mL) at Week X – Snapshot Analysis - Early Switch Phase | See Modified Snapshot in<br>Section 13.14.1<br>Not repeated | Weeks 24, 48,<br>96 and 144 |
| 2.401 | ITT-E | TBC | Summary of Study Outcomes (Plasma HIV-1 RNA $\geq$ / < 50 c/mL) at Week X – Snapshot Analysis - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | W196 |
| 2.5. | Per-<br>Protocol | TBC | Summary of Study Outcomes (Plasma HIV-1 RNA $\geq$ / < 50 c/mL) at Week X – Snapshot Analysis - PP - Early Switch Phase | See Modified Snapshot in<br>Section 13.14.1<br>No longer required | Weeks 24, 48,<br>96 and 144 |
| 2.6. | ITT | ТВС | Summary of Study Outcomes (Plasma HIV-1 RNA ≥ / < 50 c/mL) at Week X – Snapshot Analysis- ITT - Early Switch Phase | See Modified Snapshot in<br>Section 13.14.1<br>No longer required | Weeks 24, 48,<br>96 and 144 |
| 2.7. | ITT-E | EFF_T1 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA ≥ 50 c/mL at Week X – Snapshot Analysis (Sparse Data Sensitivity Analysis) - Early Switch Phase | No longer required | Weeks 24, 48,<br>96 and 144 |

| Efficacy: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Second | lary Efficacy Ar | nalyses | | | |
| 2.8. | ITT-E | EFF_T2 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week X – Snapshot Analysis - Early Switch Phase | No longer required | Weeks 24, 48,<br>96 and 144 |
| 2.9. | | | | No longer required | |
| 2.10. | | | | No longer required | |
| 2.11. | ITT-E | EFF_T5 | Summary of Proportion of Subjects with Plasma HIV-1<br>RNA ≥50 c/mL by Visit – Snapshot Analysis - Early Switch<br>Phase | No longer required | Weeks 24, 48,<br>96 and 144 |
| 2.12. | ITT-E | EFF_T5 | Summary of Proportion of Subjects with Plasma HIV-1<br>RNA <50 c/mL by Visit – Snapshot Analysis - Early Switch<br>Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 2.1201 | ITT-E | EFF_T5 | Summary of Proportion of Subjects with Plasma HIV-1<br>RNA <50 c/mL by Visit – Snapshot Analysis - DTG + 3TC<br>arm (Early and Late Switch Phase) and TBR arm (Late<br>Switch Phase) | | W196 |
| 2.13. | ITT-E | EFF_T6 | Summary of Proportion of Subjects with Plasma HIV-1<br>RNA <50 c/mL at Week X by Subgroup – Snapshot<br>Analysis - Early Switch Phase | No longer required | Weeks 24, 48,<br>96 and 144 |
| 2.14. | | | | No longer required | |
| 2.15. | ITT-E | EFF_T3 | Summary of Study Outcomes (Plasma HIV-1 RNA ≥ / < 50 c/mL) at Week X by Subgroup - Snapshot Analysis - Early Switch Phase | No longer required | Weeks 24, 48,<br>96 and 144 |

| Efficacy: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.16. | ITT-E | EFF_T8 | Summary of Change from Baseline in Plasma HIV-1 RNA (log10 c/mL) by Visit - Early Switch Phase | No longer required | Weeks 24, 48,<br>96 |
| 2.17. | ITT-E | EFF_T9 | Summary of Change from Baseline in CD4+ count (cells/mm3) by Visit - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 2.1701 | ITT-E | EFF_T9 | Summary of Change from Baseline in CD4+ count (cells/mm3) by Visit - DTG + 3TC arm - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS baseline for TBR arm | Week 196<br>(including<br>W200) |
| 2.18. | ITT-E | EFF_T9 | Summary of Change from Baseline in in CD4+/CD8+ count ratio (cells/mm3) by Visit - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 2.1801 | ITT-E | EFF_T9 | Summary of Change from Baseline in in CD4+/CD8+ count ratio (cells/mm3) by Visit - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS baseline for TBR arm | W196 |
| 2.19. | ITT-E | EFF_T10 | Summary of Post-Baseline HIV-1 Associated Conditions Including and Excluding Recurrences – Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 2.1901 | ITT-E | EFF_T10 | Summary of Post-Baseline HIV-1 Associated Conditions Including and Excluding Recurrences - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS baseline for TBR arm | Week 196<br>(including<br>W200) |
| 2.20. | | | | No longer required | |
| 2.21. | ITT-E | EFF_T11 | Summary of Post-Baseline HIV-1 Disease Progressions - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.2101 | ITT-E | EFF_T11 | Summary of Post-Baseline HIV-1 Disease Progressions - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS baseline for TBR arm | Week 196<br>(including<br>W200) |
| 2.22. | ITT-E | EFF_T12 | Cumulative Proportion of Subjects Meeting Confirmed Virologic Withdrawal Criteria by Visit - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 2.2201 | ITT-E | EFF_T12 | Cumulative Proportion of Subjects Meeting Confirmed Virologic Withdrawal Criteria by Visit - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | W196 |
| 2.23. | ITT-E | EFF_T13 | Distribution of Quantitative Plasma HIV-1 RNA Results at Suspected and Confirmed Virologic Withdrawal - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 2.24. | ITT-E | EFF_T14 | Summary of Change from Baseline in in CD4+ count (cells/mm3) at Week X by Subgroup - Early Switch Phase | No longer required | Weeks 24, 48,<br>96 and 144 |
| 2.25. | ITT-E | EFF_T15 | Summary of Kaplan-Meier Estimates of Proportion of Subjects Without Confirmed Virologic Withdrawal at Week X - Treatment Related Discontinuation = Failure - Early Switch Phase | No longer required | Weeks 24, 48,<br>96 and 144 |
| 2.26. | ITT-E | EFF_T15 | Summary of Kaplan-Meier Estimates of Proportion of Subjects Without Confirmed Virologic Withdrawal at Week X - Efficacy Related Discontinuation = Failure - Early Switch Phase | No longer required | Weeks 24, 48,<br>96 and 144 |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.27. | ITT-E | EFF_T2 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA <40 c/mL at Week X – Snapshot Analysis - Early Switch Phase | No longer required | Weeks 24, 48,<br>96 and 144 |
| 2.28. | ITT-E | EFF_T2 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA <40 c/mL and Target Not Detected Status at Week X - Snapshot Analysis - Early Switch Phase | No longer required | Weeks 24, 48,<br>96 and 144 |
| 2.29. | | | | No longer required | |
| 2.30. | | | | No longer required | |
| 2.31. | ITT-E | EFF_T3 | Summary of Study Outcomes (<40 c/mL and Target Not Detected Status) at Week X – Snapshot - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 2.3101 | ITT-E | EFF_T3 | Summary of Study Outcomes (<40 c/mL and Target Not Detected Status) at Week X – Snapshot - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | W196 |
| 2.32. | | | | No longer required | |
| 2.33. | ITT-E | EFF_T6 | Summary of Change from Baseline in CD4+/CD8+ Count Ratio (cells/mm3) at Week X by Subgroup - Early Switch Phase | No longer required | Weeks 24, 48,<br>96 and 144 |
| 2.34. | ITT-E | EFF_T14 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week X – Snapshot Analysis - Withdrawal Bias Sensitvity Analysis - Early Switch Phase | No longer required | Weeks 24, 48,<br>96 and 144 |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.35. | ITT-E | EFF_T2 | Summary of Study Outcomes (<40 c/mL) at Week X - Snapshot Analysis - Early Switch Phase | Not repeated | 48, 96 and<br>144 |
| 2.3501 | ITT-E | EFF_T2 | Summary of Study Outcomes (<40 c/mL) at Week X - Snapshot Analysis - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | W196 |
| 2.36. | EEP | EFF_T1 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA ≥ 50 c/mL at Week X – Snapshot Analysis (Evaluable Efficacy Population) - Early Switch Phase | No longer required | 96, 144 |
| 2.37. | EEP | EFF_T1 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA < 50 c/mL at Week X – Snapshot Analysis (Evaluable Efficacy Population) - Early Switch Phase | No longer required | 96, 144 |
| 2.38. | EEP | EFF_T2 | Summary of Study Outcomes (Plasma HIV-1 RNA ≥ / < 50 c/mL) at Week X – Snapshot Analysis (Evaluable Efficacy Population) - Early Switch Phase | No longer required | 96, 144 |
| 2.39. | EEP | EFF_T2 | Summary of Study Outcomes (<40 c/mL and Target Not Detected Status) at Week X – Snapshot (Evaluable Efficacy Population) - Early Switch Phase | No longer required | 96, 144 |
| 2.40. | EEP | EFF_T1 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA <40 c/mL and Target Not Detected Status at Week X - Snapshot Analysis (Evaluable Efficacy Population) - Early Switch Phase | No longer required | 96, |

# 13.15.6. Efficacy Figures

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Primar | y Efficacy Ana | alyses | | | |
| 2.1 | | | | No longer required | |
| Secon | dary Efficacy A | Analyses | | | <b>,</b> |
| 2.2. | | | | No longer required | |
| 2.3. | ITT-E | EFF_F2 | Unadjusted Treatment Difference in Proportion (95% CI) of Subjects with HIV-1 RNA <50 c/mL at Week X by Subgroup – Snapshot Analysis - Early Switch Phase | No longer required | Weeks 24, 48,<br>96 |
| 2.4. | ITT-E | EFF_F3 | Individual Plasma HIV-1 RNA and CD4+ Profiles by Visit for subjects with at least one viral load ≥50 c/MI - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96, 144 |
| 2.401 | ITT-E | EFF_F3 | Individual Plasma HIV-1 RNA and CD4+ Profiles by Visit for subjects with at least one viral load ≥50 c/MI - DTG + 3TC arm - Early and Late Switch Phase | | W196 |
| 2.402 | LS-ITT-E | EFF_F3 | Individual Plasma HIV-1 RNA and CD4+ Profiles by Visit for subjects with at least one viral load ≥50 c/MI - TBR arm - Late Switch Phase | | W196 |
| 2.5. | | | | No longer required | |
| 2.6. | ITT-E | EFF_F4 | Kaplan-Meier Plot of Time to Failure - Treatment Related Discontinuation = Failure (TRDF) - Early Switch Phase | No longer required | Weeks 24, 48,<br>96 |
| 2.7. | ITT-E | EFF_F4 | Kaplan-Meier Plot of Time to Failure - Efficacy Related Discontinuation = Failure (ERDF) - Early Switch Phase | No longer required | Weeks 24, 48,<br>96 |

# 13.15.7. Safety Tables

| Safety: T | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Exposur | е | | | | • |
| 3.1. | Safety | SAFE_T1 | Summary of Extent of Exposure to Investigational Product / Study Treatment – Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 3.2. | Safety | SAFE_T1 | Summary of Extent of Exposure to Investigational Product / Study Treatment - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | Week 144,<br>W196(includin<br>g W200 |
| 3.3. | LS-Safety | SAFE_T1 | Summary of Extent of Exposure to Investigational Product / Study Treatment - TBR - Late Switch Phase | No longer required | Week 144 |
| Adverse | Events (AEs) | | | | |
| 3.4. | Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 3.401 | Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term - DTG <u>+ 3TC</u> - Early and Late Switch Phase | DTG+3TC arm only No longer required | Week 144 |
| 3.402 | LS-Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term - TBR - Late Switch Phase | TBR arm which has switched over to DTG+3TC only No longer required | Week 144 |
| 3.5. | | | | No longer required | |
| 3.6. | Safety | AE5A | Summary of All Adverse Events by Maximum Grade - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |

| Safety: 1 | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.601 | Safety | AE5A | Summary of All Adverse Events by System Organ Class and Preferred Term and by Maximum Grade - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | W196(includin<br>g W200) |
| 3.7. | Safety | AE3 | Summary of Common (>=2%) Adverse Events by Overall Frequency- Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 3.701 | Safety | AE3 | Summary of Common (>=2%) Adverse Events by Overall Frequency - DTG <u>+ 3TC</u> arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | W196<br>(including<br>W200) |
| 3.8. | Safety | AE3 | Summary of Common (>=2%) Grade 2-5 Adverse Events by Overall Frequency-Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 3.801 | Safety | AE3 | Summary of Common (>=2%) Grade 2-5 Adverse Events by Overall Frequency- DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | W196<br>(including<br>W200 |
| 3.9. | Safety | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term – Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 3.10. | Safety | AE5A | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Grade - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 3.1001 | Safety | AE5A | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Grade - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | Week 144,<br>W196(includin<br>g W200 |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 3.1002 | LS-Safety | AE5A | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Grade – TBR - Late Switch Phase | TBR arm which has switched over to DTG+3TC only No longer required | Week 144 |
| 3.11. | Safety | AE15 | Summary of Common (>=2%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subject and Occurrences) - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 3.1101 | Safety | AE15 | Summary of Common (>=2%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subject and Occurrences) - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | W196(includin<br>g W200 |
| 3.12. | Safety | AE3 | Summary of Common (>=0.5%) Drug-Related Grade 2-5 Adverse Events by Overall Frequency- Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 3.1201 | Safety | AE3 | Summary of Common (>=0.5%) Drug-Related Grade 2-5 Adverse Events by Overall Frequency - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | W196(includin<br>g W200 |
| 3.13. | | | | No longer required | |

| Safety: T | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Serious | and Other Sign | ificant Adver | se Events | | |
| 3.14. | Safety | AE16 | Summary of Serious Adverse Events by System Organ<br>Class and Preferred Term (Number of Subjects and<br>Occurrences) - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 3.1401 | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | Week 144,<br>W196(includin<br>g W200) |
| 3.1402 | LS-Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – TBR - Late Switch Phase | TBR arm which has switched over to DTG+3TC only No longer required | Week 144 |
| 3.15. | Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term /by Overall Frequency - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96, 144 |
| 3.1501 | Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term /by Overall Frequency - DTG + 3TC - Early and Late Switch Phase | DTG+3TC arm only No longer required | Week 144, |
| 3.1502 | LS-Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term /by Overall Frequency – TBR - Late Switch Phase | TBR arm which has switched over to DTG+3TC only No longer required | Week 144, |

| Safety: T | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.16. | Safety | AE5A | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by Maximum Grade - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96, 144 |
| 3.1601 | Safety | AE5A | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by Maximum Grade - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | W196(includin<br>g W200) |
| 3.17. | | | | No longer required | |
| 3.18. | Safety | AE3 | Summary of Serious Adverse Events by System Organ Class - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 3.1801 | Safety | AE3 | Summary of Serious Adverse Events by System Organ Class - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | W196(includin<br>g W200 |
| 3.19. | | | | No longer required | |
| 3.20. | Safety | AE1 | Summary of Drug-Related Serious Adverse Events by System Organ Class - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 3.2001 | Safety | AE1 | Summary of Drug-Related Serious Adverse Events by System Organ Class - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | W196(includin<br>g W200 |
| 3.21. | | | | No longer required | |

| Safety: 7 | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Laborat | ory: Chemistry | | | | <u> </u> |
| 3.22. | Safety | LB1 | Summary of Chemistry Changes from Baseline by Visit - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 3.2201 | Safety | LB1 | Summary of Chemistry Changes from Baseline by Visit - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | W196<br>(including<br>W200) |
| 3.23. | Safety | SAFE_T3 | Summary of Maximum Post-Baseline Emergent Chemistry Toxicities - Lipid LOCF - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96, 144 |
| 3.2301 | Safety | SAFE_T3 | Summary of Maximum Post-Baseline Emergent Chemistry Toxicities - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | Week 144,<br>W196<br>(including<br>W200) |
| 3.24. | Safety | LB1 | Summary of Fasting Lipids by Visit - Lipid LOCF - Early Switch Phase | Not required | Weeks 24, 48,<br>96 |
| 3.25. | | | | No longer required | |
| 3.26. | Safety | LB1 | Summary of Fasting Lipids Percentage Changes from Baseline by Visit - Lipid LOCF - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96, 144 |
| 3.27. | | | | Not required | |
| 3.2601 | Safety | LB1 | Summary of Fasting Lipids Percentage Changes from Baseline by Visit - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | W196 |

| Safety: T | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.28. | | | | No longer required | |
| 3.29. | | | | No longer required | |
| 3.30. | Safety | SAFE_T5 | Summary of Changes in NCEP Lipid Baseline Category to Week X Category - Lipid LOCF – Early Switch Phase | Triglycerides, HDL, LDL<br>Cholesterol, Total Cholesterol<br>(mmol/L) NCEP Categories<br>Not repeated | Weeks 24, 48,<br>96, 144 |
| 3.3001 | Safety | SAFE_T5 | Summary of Changes in NCEP Lipid Baseline Category to Week X Category - DTG <u>+ 3TC</u> arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | Triglycerides, HDL, LDL<br>Cholesterol, Total Cholesterol<br>(mmol/L) NCEP Categories<br>LS Baseline for TBR arm | W196 |
| 3.31. | | | | No longer required | |
| 3.32. | Safety | SAFE_T6 | Summary of Changes in Total Cholesterol /HDL Ratio<br>Baseline Category to Week X - Lipid LOCF - Early Switch<br>Phase | Not repeated | Weeks 24, 48,<br>96, 144 |
| 3.3201 | Safety | SAFE_T6 | Summary of Changes in Total Cholesterol /HDL Ratio Baseline Category to Week 196 - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | W196 |
| 3.33. | | | | No longer required | |

| Safety: T | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Laborato | ry: Hematolog | y | | | |
| 3.34. | Safety | LB1 | Summary of Hematology Changes from Baseline - Early Switch Phase | Not repeated | Weeks 24, 48, 96,,4 |
| 3.3401 | Safety | LB1 | Summary of Hematology Changes from Baseline - DTG <u>+</u> <u>3TC</u> arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | W196<br>(including<br>W200) |
| 3.35. | Safety | SAFE_T3 | Summary of Maximum Post-Baseline Emergent<br>Hematology Toxicities - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96, 144 |
| 3.3501 | Safety | SAFE_T3 | Summary of Maximum Post-Baseline Emergent Hematology Toxicities - DTG <u>+ 3TC</u> arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | W196<br>(including<br>W200) |
| Laborato | ry: Urinalysis | | | | |
| 3.36. | | | | No longer required | |
| Biomark | ers | | | | |
| 3.37. | Safety | LB1 | Summary of Change from Baseline in Bone Biomarkers by Visit - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96, 144 |
| 3.3701 | Safety | LB1 | Summary of Change from Baseline in Bone Biomarkers by Visit - DTG <u>+ 3TC</u> arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | W196 |
| 3.38. | Safety | LB1 | Summary of Change from Baseline in Renal Biomarkers by Visit - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96, 144 |

| Safety: T | 1 | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.3801 | Safety | LB1 | Summary of Change from Baseline in Renal Biomarkers by Visit - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | W196 |
| 3.39. | Safety | LB1 | Summary of Change from Baseline in Renal Biomarkers by Visit - Loge Transformed Data - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96, 144 |
| 3.3901 | Safety | LB1 | Summary of Change from Baseline in Renal Biomarkers by Visit - Loge Transformed Data - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | W196 |
| 3.40. | | | | No longer required | |
| 3.41. | Safety | SAFE_T7 | Statistical Analysis of Change from Baseline Bone<br>Biomarkers – MMRM - Early Switch Phase | No longer required | Weeks 24, 48,<br>96, 144 |
| 3.42. | Safety | SAFE_T7 | Statistical Analysis of Change from Baseline in Renal Biomarkers – MMRM - Early Switch Phase | No longer required | Weeks 24, 48,<br>96, 144 |
| 3.43. | Safety | SAFE_T7 | Statistical Analysis of Change from Baseline in Renal<br>Biomarkers - Loge Transformed Data - MMRM - Early<br>Switch Phase | No longer required | Weeks 24, 48,<br>96, 144 |
| 3.44. | | | | No longer required | |

| Safety: T | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Laborate | ory: Hepatobilia | ry (Liver) | | | |
| 3.45. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96, 144 |
| 3.4501 | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | W196<br>(including<br>W200) |
| 3.46. | Safety | LIVER10 | Summary of Subjects Meeting Hepatobiliary Abnormality<br>Criteria – All Post-Baseline Abnormalities - Early Switch<br>Phase | Not repeated | Weeks 24, 48,<br>96, 144 |
| 3.4601 | Safety | LIVER10 | Summary of Subjects Meeting Hepatobiliary Abnormality Criteria – All Post-Baseline Abnormalities - DTG + 3TC am (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | Week 144,<br>W196<br>(including<br>W200) |
| Other | | | | | |
| 3.47. | Safety | SAFE_T8 | Summary of True Positive Suicidal Indication Alerts Based on eCSSRS by Visit - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96, 144 |
| 3.4701 | Safety | SAFE_T8 | Summary of True Positive Suicidal Indication Alerts Based on eCSSRS by Visit - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | W196 |
| 3.48. | Safety | SAFE_T9 | Summary of Subjects with C-SSRS Suicidal Ideation or Behaviour at Baseline - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96, 144 |
| 3.49. | Safety | SAFE_T9 | Summary of Subjects with Post Baseline C-SSRS Suicidal Ideation or Behaviour - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96, 144 |

| Safety: T | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.4901 | Safety | SAFE_T9 | Summary of Subjects with Post Baseline C-SSRS Suicidal Ideation or Behaviour - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | W196 |
| 3.50. | Safety | SAFE_T10 | Summary of Characteristics of Post Baseline Anxiety Adverse Events of Special Interest - Early Switch Phase | Not repeated | All |
| 3.5001 | Safety | SAFE_T10 | Summary of Characteristics of Post Baseline Anxiety Adverse Events of Special Interest - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | Week 196<br>(including<br>W200) |
| 3.51. | Safety | SAFE_T10 | Summary of Characteristics of Post Baseline Depression<br>Adverse Events of Special Interest - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96, 144 |
| 3.5101 | Safety | SAFE_T10 | Summary of Characteristics of Post Baseline Depression Adverse Events of Special Interest - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | Week 196<br>(including<br>W200) |
| 3.52. | Safety | SAFE_T10 | Summary of Characteristics of Post Baseline Suicidality and Self Injury Adverse Events of Special Interest - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96, 144 |
| 3.5201 | Safety | SAFE_T10 | Summary of Characteristics of Post Baseline Suicidality and Self Injury Adverse Events of Special Interest - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | Week 196<br>(including<br>W200) |
| 3.53. | Safety | SAFE_T10 | Summary of Characteristics of Post Baseline Insomnia<br>Adverse Events of Special Interest - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96, 144 |

| Safety: T | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.5301 | Safety | SAFE_T10 | Summary of Characteristics of Post Baseline Insomnia Adverse Events of Special Interest - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | Week 196<br>(including<br>W200) |
| 3.54. | Safety | SAFE_T10 | Summary of Characteristics of Post Baseline Rash<br>Adverse Events of Special Interest - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96, 144 |
| 3.5401 | Safety | SAFE_T10 | Summary of Characteristics of Post Baseline Rash<br>Adverse Events of Special Interest - DTG + 3TC arm (Early<br>and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | Week 196<br>(including<br>W200) |
| 3.55. | Safety | SAFE_T10 | Summary of Characteristics of Post Baseline Nightmare/Abnormal Dreams Adverse Events of Special Interest - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 3.5501 | Safety | SAFE_T10 | Summary of Characteristics of Post Baseline Nightmare/Abnormal Dreams Adverse Events of Special Interest - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | Week 196<br>(including<br>W200) |
| 3.56. | Safety | SAFE_T10 | Summary of Characteristics of Post Baseline Drug Hypersensitivity Adverse Events of Special Interest - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 3.5601 | Safety | SAFE_T10 | Summary of Characteristics of Post Baseline Drug Hypersensitivity Adverse Events of Special Interest - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | Week 196<br>(including<br>W200) |

| Safety: T | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.57. | Safety | SAFE_T11 | Summary of Onset and Duration of the First Occurrence of Post Baseline Anxiety Adverse Events of Special Interest - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 3.5701 | Safety | SAFE_T11 | Summary of Onset and Duration of the First Occurrence of Post Baseline Anxiety Adverse Events of Special Interest - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | Week 196<br>(including<br>W200) |
| 3.58. | Safety | SAFE_T11 | Summary of Onset and Duration of the First Occurrence of Post Baseline Depression Adverse Events of Special Interest - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 3.5801 | Safety | SAFE_T11 | Summary of Onset and Duration of the First Occurrence of Post Baseline Depression Adverse Events of Special Interest - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | Week 196<br>(including<br>W200) |
| 3.59. | Safety | SAFE_T11 | Summary of Onset and Duration of the First Occurrence of Post Baseline Suicidality and Self Injury Adverse Events of Special Interest - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 3.5901 | Safety | SAFE_T11 | Summary of Onset and Duration of the First Occurrence of Post Baseline Suicidality and Self Injury Adverse Events of Special Interest - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | Week 196<br>(including<br>W200) |
| 3.60. | Safety | SAFE_T11 | Summary of Onset and Duration of the First Occurrence of Post Baseline Insomnia Adverse Events of Special Interest - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |

| Safety: T | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.6001 | Safety | SAFE_T11 | Summary of Onset and Duration of the First Occurrence of Post Baseline Insomnia Adverse Events of Special Interest - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | Week 196<br>(including<br>W200) |
| 3.61. | Safety | SAFE_T11 | Summary of Onset and Duration of the First Occurrence of Post Baseline Rash Adverse Events of Special Interest - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 3.6101 | Safety | SAFE_T11 | Summary of Onset and Duration of the First Occurrence of Post Baseline Rash Adverse Events of Special Interest - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | Week 196<br>(including<br>W200) |
| 3.62. | Safety | SAFE_T11 | Summary of Onset and Duration of the First Occurrence of Post Baseline Nightmare/Abnormal Dreams Adverse Events of Special Interest - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 3.6201 | Safety | SAFE_T11 | Summary of Onset and Duration of the First Occurrence of Post Baseline Nightmare/Abnormal Dreams Adverse Events of Special Interest - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | Week 196<br>(including<br>W200) |
| 3.63. | Safety | SAFE_T11 | Summary of Onset and Duration of the First Occurrence of Post Baseline Drug Hypersensitivity Adverse Events of Special Interest - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 3.6301 | Safety | SAFE_T11 | Summary of Onset and Duration of the First Occurrence of Post Baseline Drug Hypersensitivity Adverse Events of Special Interest - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | Week 196<br>(including<br>W200) |
| 3.64. | | | | No longer required | |

| Safety: 7 | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL/<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.65. | | | | No longer required | |
| 3.66. | | | | No longer required | |
| 3.67. | | | | No longer required | |
| 3.68. | | | | No longer required | |
| 3.69. | | | | No longer required | |
| 3.70. | | | | No longer required | |
| 3.71. | Safety | SAFE_T15 | Summary of Post Baseline Depression and Suicidal and Self-Injury Adverse Events by AE of Special Interest, Maximum DAIDS Toxicity Grade, and Prior History of Depression and Anxiety - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96, 144 |
| 3.7101 | Safety | SAFE_T15 | Summary of Post Baseline Depression and Suicidal and Self-Injury Adverse Events by AE of Special Interest, Maximum DAIDS Toxicity Grade, and Prior History of Depression and Anxiety - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | W196(includin<br>g W200 |
| 3.72. | | | | No longer required | |
| 3.73. | Safety | LB1 | Summary of Change from Baseline in HOMA-Insulin<br>Resistance at Week X - Loge Transformed Data - Early<br>Switch Phase | No longer required | Weeks 24, 48,<br>96 and 144 |
| 3.74. | Safety | SAFE_T7 | Statistical Analysis of Change from Baseline in HOMA-<br>Insulin Resistance at Week X - Loge Transformed Data –<br>MMRM - Early Switch Phase | No longer required | 48, 96, 144 |

| Safety: T | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.75. | Safety | LB1 | Summary of Change from Baseline in Weight (kg) by Visit - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96, 144 |
| 3.7501 | Safety | LB1 | Summary of Change from Baseline in Weight (kg) by Visit - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | W196<br>(including<br>W200) |
| 3.76. | Safety | LB1 | Summary of Change from Baseline in BMI (kg/m2) by Visit - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96, 144 |
| 3.7601 | Safety | LB1 | Summary of Change from Baseline in BMI (kg/m2) by Visit - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | W196<br>(including<br>W200) |
| 3.77. | Safety | SAFE_T7 | Statistical Analysis of Change from Baseline in Weight (kg) – MMRM - Early Switch Phase | No longer required | Weeks 24, 48,<br>96,,144 |
| 3.78. | Safety | SAFE_T7 | Statistical Analysis of Change from Baseline in BMI (kg/m2) – MMRM - Early Switch Phase | No longer required | Weeks 24, 48,<br>96, 144 |
| 3.79. | | | | No longer required | |
| 3.80. | | | | | W196 |
| 3.81. | Safety | SAFE_T16 | Summary of HOMA-IR Shifts from Baseline to Week X - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96, 144 |
| 3.8101 | Safety | SAFE_T16 | Summary of HOMA-IR Shifts from Baseline to Week X - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | W196 |
| 3.82. | | | | No longer required | |

| Safety: 7 | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.83. | Safety | New shell | Sumamry of Chemistry by Visit - Early Switch Phase | Not required | All |
| 3.84. | Safety | New shell | Summary of Hematology by Visit - Early Switch Phase | Not required | All |
| 3.85. | Safety | New shell | Summary of Weight (kg) by Visit - Early Switch Phase | Not required | All |
| 3.86. | Safety | New shell | Summary of BMI (kg/m2) by Visit - Early Switch Phase | Not required | All |
| 3.87. | | | | No longer required | |
| 3.88. | | | | No longer required | |
| 3.89. | | | | No longer required | |
| 3.90. | | | | No longer required | |
| 3.91. | | | | No longer required | |
| 3.92. | | | | No longer required | |
| 3.93. | | | | No longer required | |
| 3.94. | | | | No longer required | |
| 3.95. | | | | No longer required | |
| 3.96. | Safety | LB1 | Summary of Change from Baseline in Inflammatory Biomarkers - Loge Transformed Data - Early Switch Phase | Not repeated | 48,96,144 |
| 3.9601 | Safety | LB1 | Summary of Change from Baseline in Inflammatory Biomarkers - Loge Transformed Data - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | W196 |

| Safety: 1 | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.97. | Safety | SAFE_T7 | Statistical Analysis of Change from Baseline in Inflammatory Biomarkers at Week X – Loge Transformed Data – MMRM – Early Switch Phase | No longer required | 48,96,144 |
| 3.98. | Safety | SAFE_T18 | Summary of Proportion of Subjects with Change from Baseline in Weight (>=3%, >=5% and >=10%) at Week X – Early Switch Phase | Not repeated | 48,96,144 |
| 3.9801 | Safety | SAFE_T18 | Summary of Proportion of Subjects with Change from Baseline in Weight (>=3%, >=5% and >=10%) at Week X - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | W196<br>(including<br>W200) |
| 3.99. | Safety | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term up to the End of the Week 144 Reporting Window (USPI) - Early Switch Phase | Not repeated | 48,96,144 |
| 3.9901 | Safety | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term up to the End of the Week 196 Reporting Window (USPI) - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | W196<br>(including<br>W200) |
| 3.100 | Safety | AE3 | Summary of Common (>=0.5%) Drug-Related Grade 2-5<br>Adverse Events by Overall Frequency up to the End of the<br>Week X Reporting Window (USPI) - Early Switch Phase | Not repeated | 48,96,144 |

| Safety: Ta | ables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.10001 | Safety | AE3 | Summary of Common (>=0.5%) Drug-Related Grade 2-5 Adverse Events by Overall Frequency up to the End of the Week X Reporting Window (USPI) - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | W196<br>(including<br>W200) |
| 3.101 | Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term /by Overall Frequency up to the End of the Week X Reporting Window (USPI) - Early Switch Phase | Not repeated | 48,96,144 |
| 3.10101 | Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term /by Overall Frequency up to the End of the Week X Reporting Window (USPI) - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | W196<br>(including<br>W200) |
| 3.102 | Safety | SAFE_T2 | Summary of Cumulative Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by Visit - Early Switch Phase | No longer required | 48,96,144 |
| 3.103 | Safety | SAFE_T14 | Summary of BMI Shifts from Baseline to Week X - Early Switch Phase | No longer required | 48,96 |
| 3.104 | Safety | SAFE_T10 | Summary of Characteristics of Post Baseline Increase in<br>Weight Adverse Events of Special Interest - Early Switch<br>Phase | Not repeated | 48,96,144 |

| Safety: T | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.10401 | Safety | SAFE_T10 | Summary of Characteristics of Post Baseline Increase in Weight Adverse Events of Special Interest - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | W196<br>(including<br>W200) |
| 3.105 | Safety | SAFE_T10 | Summary of Characteristics of Post Baseline Decrease in<br>Weight Adverse Events of Special Interest - Early Switch<br>Phase | Not repeated | 48,96,144 |
| 3.10501 | Safety | SAFE_T10 | Summary of Characteristics of Post Baseline Decrease in Weight Adverse Events of Special Interest - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | W196<br>(including<br>W200) |
| 3.106 | Safety | SAFE_T7 | Statistical Analysis of Change from Baseline in Fasting<br>Lipids - Loge Transformed Data - MMRM - Lipid LOCF -<br>Early Switch Phase | No longer required | 96, 144 |
| 3.107 | Safety | SAFE_T7 | Statistical Analysis of Variables Associated with >=2<br>HOMA-IR at Week 48 - Logistic Regression - Early Switch<br>Phase | May not be performed depending on scope of missing data No longer required | 96, 144 |
| 3.108 | Safety | SAFE_T3 | Summary of Maximum Post-Baseline Emergent Clinical Chemistry Toxicities to the End of the Week X Reporting Window (USPI) – LOCF - Early Switch Phase | Not repeated | 96, 144 |
| 3.10801 | Safety | SAFE_T3 | Summary of Maximum Post-Baseline Emergent Clinical Chemistry Toxicities to the End of the Week X Reporting Window (USPI) – LOCF - DTG <u>+ 3TC</u> arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | W196<br>(including<br>W200) |

| Safety: T | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.109 | | | | No longer required | 96, 144 |
| 3.110 | Safety | SAFE_T3 | Summary of Maximum Post-Baseline Emergent<br>Hematology Toxicities to the End of the Week X Reporting<br>Window (USPI) - Early Switch Phase | For Week 144: Up to end of<br>Week 144 visit window (i.e.<br>Week 144 + 4)<br>Not repeated | 96, 144 |
| 3.11001 | Safety | SAFE_T3 | Summary of Maximum Post-Baseline Emergent Hematology Toxicities to the End of the Week X Reporting Window (USPI) - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | W196<br>(including<br>W200) |
| 3.111 | Safety | PAN1 | Summary of COVID-19 Assessments - Early Switch Phase | Not repeated | From week 96 onwards |
| 3.11101 | Safety | PAN1 | Summary of COVID-19 Assessments - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | W196 |
| 3.112 | Safety | PAN10 | Summary of Exposure Adjusted Adverse Event Incidence<br>Rates Over Time Overall and by Country, Gender and Age<br>- Early Switch Phase | No longer required | 96, 144 |
| 3.113 | Safety | AE5A | Summary of All Adverse Events by Maximum Grade<br>Adverse Events Reported After the End of the Week 48<br>Analysis Window - Early Switch Phase | No longer required | 96, 144 |

| Safety: T | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.114 | Safety | AE5A | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Grade Adverse Events Reported After the End of the Week 48 Analysis Window - Early Switch Phase | No longer required | 96, 144 |
| 3.115 | Safety | AE16 | Summary of Serious Adverse Events by System Organ<br>Class and Preferred Term (Number of Subjects and<br>Occurrences) Adverse Events Reported After the End of<br>the Week 48 Analysis Window - Early Switch Phase | No longer required | 96, 144 |
| 3.116 | Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term Adverse Events Reported After the End of the Week 48 Analysis Window - Early Switch Phase | No longer required | 96, 144 |
| 3.117 | Safety | SAFE_T7 | Statistical Analysis of Change from Baseline in Weight (kg) by Visit - MMRM by Baseline BMI - Early Switch Phase | By BMI categories No longer required | 96, 144 |
| 3.118 | Safety | New shell | Summary of Waist to Height Ratio and Waist to Hip Ratio at Week 144 | Not repeated | 144 |
| 3.11801 | Safety | New shell | Summary of Waist to Height Ratio and Waist to Hip Ratio by Visit - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | W196<br>(including<br>W200) |
| 3.11803 | LS-Safety | New shell | Summary of Change from LS Baseline in Waist to Height Ratio and Waist to Hip Ratio at Week 196 - TBR arm – Late Switch Phase | | W196<br>(including<br>W200) |

| Safety: T | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.119 | Safety | New shell | Proportion of Subjects with Metabolic Syndrome at Week 144 | Refer Table 1.025 in RE<br>postcsr_2020_03 for shell<br>(overall only)<br>Not repeated | 144 |
| 3.11901 | Safety | New shell | Proportion of Subjects with Metabolic Syndrome at Week 196 - DTG <u>+ 3TC</u> arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | Refer Table 1.025 in RE postcsr_2020_03 for shell (overall only) | W196<br>(including<br>W200) |
| 3.120 | Safety | LB1 | Summary of Change from Baseline in Framingham Risk<br>Score at Week 144 | Not repeated | 144 |
| 3.12001 | Safety | LB1 | Summary of Change from Baseline in Framingham Risk<br>Score at Week 196 - DTG <u>+ 3TC</u> arm (Early and Late<br>Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | W196 |
| 3.121 | Safety | LB1 | Summary of Change from Baseline in Systolic Blood Pressure and Diastolic Blood Pressure at week 144 | Not repeated | 144 |
| 3.12101 | Safety | LB1 | Summary of Change from Baseline in Systolic Blood Pressure and Diastolic Blood Pressure at week 196 - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | LS Baseline for TBR arm | W196(includin<br>g W200 |

# 13.15.8. Safety Figures

| Safety: I | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Adverse | Events | | | | |
| 3.1. | Safety | AE10 | Plot of Common (>=2%) Adverse Events and Relative Risk- Early Switch Phase | Not repeated | Weeks 24, 48,<br>96, 144 |
| Laborat | ory | | | | |
| 3.2. | Safety | LIVER14 | Scatter Plot of Maximum vs. Baseline for ALT - Early Switch Phase | Not required | Weeks 24, 48,<br>96 |
| 3.3. | Safety | LIVER9 | Scatter Plot of Maximum ALT vs. Maximum Total Bilirubin - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 3.301 | Safety | LIVER9 | Scatter Plot of Maximum ALT vs. Maximum Total Bilirubin - DTG + 3TC arm - Early and Late Switch Phase | | W196<br>(including<br>W200) |
| 3.302 | LS-Safety | LIVER9 | Scatter Plot of Maximum ALT vs. Maximum Total Bilirubin - TBR arm - Late Switch Phase | | W196<br>(including<br>W200) |

| Safety: | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Other | | | | | |
| 3.4. | Safety | SAFE_F1 | Heatmap plot of Triglycerides, LDL Cholesterol, Total Cholesterol (mmol/L) NCEP Categories and Total Cholesterol/HDL Ratio at Week X vs. Baseline –Lipid LOCF - Early Switch Phase | Not repeated | Weeks 24, 48,<br>96 and 144 |
| 3.401 | Safety | SAFE_F1 | Heatmap plot of Triglycerides, LDL Cholesterol, Total Cholesterol (mmol/L) NCEP Categories and Total Cholesterol/HDL Ratio at Week X vs. Baseline – DTG + 3TC arm - Early and Late Switch Phase | | W196 |
| 3.402 | LS-Safety | SAFE_F1 | Heatmap plot of Triglycerides, LDL Cholesterol, Total<br>Cholesterol (mmol/L) NCEP Categories and Total<br>Cholesterol/HDL Ratio at Week X vs. LS Baseline - TBR<br>arm - Late Switch Phase | | W196 |
| 3.5. | | | | No longer required | |
| 3.6. | | | | No longer required | |
| 3.7. | Safety | SAFE_F2 | Line Plot of Adjusted Mean (95% CI) Change from Baseline in Renal Biomarkers Over Time — MMRM - Early Switch Phase | No longer required | Weeks 24, 48,<br>96 and 144 |
| 3.8. | Safety | SAFE_F3 | Line Plot of Ratio of Geometric Means (95% CI) in Renal<br>Biomarkers Over Time - Loge Transformed Data –<br>MMRM - Early Switch Phase | No longer required | Weeks 24, 48,<br>96 and 144 |

| Safety: | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.9. | Safety | SAFE_F2 | Line Plot of Adjusted Mean (95% CI) of Change from Baseline in Bone Biomarkers Over Time — MMRM - Early Switch Phase | No longer required | Weeks 24, 48,<br>96, 144 |
| 3.10. | Safety | SAFE_F5 | Line Plot of Adjusted Mean (95% CI) of Change from Baseline in Weight (kg) Over Time — MMRM - Early Switch Phase | No longer required | Weeks 24, 48,<br>96, 144 |
| 3.11. | Safety | SAFE_F5 | Line Plot of Adjusted Mean (95% CI) of Change from Baseline in BMI (kg/m2) Over Time — MMRM - Early Switch Phase | No longer required | Weeks 24, 48,<br>96, 144 |
| 3.12. | Safety | SAFE_F1 | Bar Chart of Total Cholesterol/HDL Ratio Categories at Week X vs. Baseline –Lipid LOCF | No longer required | Weeks 24, 48, |
| 3.13. | | | | No longer required | |
| 3.14. | | | | No longer required | |
| 3.15. | | | | No longer required | |
| 3.16. | Safety | SAFE_F2 | Line Plot of Ratio of Geometric Means (95% of CI) in HOMA-IR Over Time - Loge Transformed Data - MMRM - Early Switch Phase | No longer required | 48, 96, 144 |
| 3.17. | | | | No longer required | |
| 3.18. | | | | No longer required | |

| Safety: | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.19. | | | | No longer required | |
| 3.20. | | | | No longer required | |
| 3.21. | | | | No longer required | |
| 3.22. | Safety | SAFE_F2 | Line Plot of Ratio of Geometric Means (95% of CI) in Inflammatory Biomarkers Over Time - Loge Transformed – MMRM - Early Switch Phase | No longer required | 48, 96, 144 |
| 3.23. | Safety | SAFE_F2 | Line Plot of Ratio of Geometric Means (95% CI) in Fasting Lipids Over Time - MMRM - Lipid LOCF - Loge Transformed Data - Early Switch Phase | No longer required | 96, 144 |
| 3.24. | Safety | SAFE_F2 | Line Plot of Adjusted Mean (95% of CI) of Change from Baseline in Weight (kg) Over Time-MMRM-by Baseline BMI - Early Switch Phase | No longer required | 96, 144 |
| 3.25. | Safety | SAFE_T14 | Heatmap plot of BMI at Week X vs. Baseline - Early Switch Phase | Not repeated | 144 |
| 3.2501 | Safety | SAFE_T14 | Heatmap plot of BMI at Week X vs. Baseline - DTG <u>+</u> <u>3TC</u> arm - Early and Late Switch Phase | | W196<br>(including<br>W200) |
| 3.2502 | LS-Safety | SAFE_T14 | Heatmap plot of BMI at Week X vs. LS Baseline - TBR arm - Late Switch Phase | | W196<br>(including<br>W200) |

# 13.15.9. Virology tables

| Virolog | Virology: Tables | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.1. | CWW | VIR_T1 | Summary of INSTI Mutations and Major Mutations of NRTI, NNRTI and PI Classes by region at Baseline and Time of CWV at or prior to Week X - Early Switch Phase | Combine 4.1 and 4.2 | Weeks 24,<br>48, 96 and<br>144 |
| 4.101 | CW | VIR_T1 | Summaryof INSTI Mutations and Major Mutations of NRTI, NNRTI and PI Classes by region at Baseline and Time of CWW at or prior to Week X - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | Combine 4.1 and 4.2 | W196 |
| 4.2. | CW | VIR_T2 | Summary of Major Mutations of NRTI, NNRTI and PI<br>Classes by region at Baseline and Time of CWV at or<br>prior to Week X - Early Switch Phase | Not Required (Combine with 4.1) | Weeks 24,<br>48, 96 |

| Virolog | Virology: Tables | | | | |
|---|---|---|---|---|---|
| 4.3. | CWV | VIR_T3 | Summary of Genotypi c Susceptibility Score at Baseline and Time of CWW by Genotypic Cut-Off at or prior to Week X - Early Switch Phase | Not Required | All |
| 4.4. | CW | VIR_T4 | Summary of Phenotype at Baseline and Time of CWW by Phenotypic Cut-off at or prior to Week X - Early Switch Phase | Not repeated | Weeks 24,<br>48, 96 and<br>144 |
| 4.401 | CW | VIR_T4 | Summary of Phenotype at Baseline and Time of CVW by Phenotypic Cut-off at or prior to Week X - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | W196 |
| 4.5. | CW | VIR_T5 | Summary of Phenotype at time of CVW by Number of Drugs to Which Subject are Resistant at or prior to Week X - Early Switch Phase | Not repeated | Weeks 24,<br>48, 96 and<br>144 |
| 4.501 | CW | VIR_T5 | Summary of Phenotype at time of CWW by Number of Drugs to Which Subject are Resistant at or prior to Week X - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | W196 |
| 4.6. | CW | VIR_T6 | Summary of Fold Change to DTG, 3TC, TDF and FTC at - Time of CVW at or prior to Week X - Early Switch Phase | Not repeated | Weeks 24,<br>48, 96 and<br>144 |
| 4.601 | CW | VIR_T6 | Summary of Fold Change to DTG, 3TC, TDF and FTC at - Time of CWV at or prior to Week X - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | W196 |

| Virolog | Virology: Tables | | | | |
|---|---|---|---|---|---|
| 4.7. | Viral<br>Genotypic | VIR_T7 | Summary of Subject Accountability: Genotypes Available at or prior to Week X - Early Switch Phase | Not repeated | Weeks 24,<br>48, 96 and<br>144 |
| 4.701 | Viral<br>Genotypic | VIR_T7 | Summary of Subject Accountability: Genotypes Available at or prior to Week X - DTG <u>+ 3TC</u> arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | W196 |
| 4.8. | Viral<br>Phenotypic | VIR_T8 | Summary of Subject Accountability: Phenotypes Available at or prior to Week X - Early Switch Phase | Not repeated | Weeks 24,<br>48, 96 and<br>144 |
| 4.801 | Viral<br>Phenotypic | VIR_T8 | Summary of Subject Accountability: Phenotypes Available at or prior to Week X - DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | | W196 |

#### 13.15.10. Pharmacokinetic Tables

| Pharm | acokinetic : Tab | oles | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Intens | ive PK - PK Con | centration Da | ıta | | |
| 5. | | | | No longer required | |
| 5.2 | | | | No longer required | |
| Intens | ive PK Derived I | Parameters | | | - |
| 5.3. | | | | No longer required | |
| 5.4. | | | | No longer required | |
| Sparse | PK - PK Conce | entration Data | | · | |
| 5.5. | | | | No longer required | |
| 5.6. | | | | No longer required | |
| 5.7. | | | | No longer required | |
| 5.8. | | | | No longer required | |

# 13.15.11. Pharmacokinetic Figures

| Pharmaco | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Intensive | PK - PK Cond | centration Da | ta | | |
| 5.1. | | | | No longer required | |
| 5.2. | | | | No longer required | |
| 5.3. | | | | No longer required | |
| 5.4. | | | | No longer required | |
| 5.5. | | | | No longer required | |
| 5.6. | | | | No longer required | |
#### 13.15.12. Health Outcomes Tables

| Health | Health Outcomes : Tables | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| EQ-5D | -5L | | | | |
| 6.1. | ITT(E) | HO_T1 | Summary of EQ-5D Category Scores by visit – LOCF - Early Switch Phase | No longer required | Weeks 24, 48,<br>96 |
| 6.2. | ITT(E) | HO_T2 | Summary of EQ-5D Utility and Thermometer Scores by visit – LOCF - Early Switch Phase | Not repeated | Weeks 24, 48, 96 and 144 |
| 6.201 | ITT(E) | HO_T2 | Summary of EQ-5D Utility and Thermometer Scores by visit – DTG + 3TC arm (Early and Late Switch Phase) and TBR arm (Late Switch Phase) | Summary on Observed data<br>For LS DTG+3TC group, label<br>W144 as LS Baseline | W196 |
| 6.3. | ITT(E) | HO_T2 | Summary of Change from Baseline in EQ-5D Utility and Thermometer Scores – LOCF - Early Switch Phase | No longer required | Weeks 24, 48,<br>96 |
| 6.4. | ITT(E) | HO_T3 | Statistical Analysis of Change from Baseline in EQ-5D Utility Scores – MMRM – LOCF - Early Switch Phase | No longer required | Weeks 24, 48, 96 and 144 |
| 6.5. | ITT(E) | HO_T3 | Statistical analysis of Change from Baseline in EQ-5D Thermometer Scores – MMRM – LOCF - Early Switch Phase | No longer required | Weeks 24, 48,<br>96 and 144 |
| Willing | Willingness to switch | | | | |
| 6.6. | ITT(E) | HO_T4 | Summary of Reasons for Willingness to Switch – Early Switch Phase | Not repeated | All |

# 13.15.13. Health Outcomes Figures

| Health | Health Outcomes : Figures | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| EQ-5D | -5L | | | | |
| 6.1. | ITT(E) | HO_F1 | Line Plot of Adjusted Mean (95% CI) Change from Baseline in EQ-5D Utility Score Over Time – MMRM - LOCF - Early Switch Phase | No longer required | Weeks 24,<br>48, 96 and<br>144 |
| 6.2. | ITT(E) | HO_F1 | Line Plot of Adjusted Mean (95% CI) Change from Baseline in EQ-5D Thermometer Score Over Time – MMRM – LOCF - Early Switch Phase | No longer required | Weeks 24,<br>48, 96 and<br>144 |

# 13.15.14. ICH Listings

| ICH: L | CH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | ct Disposition | | | | |
| 1. | All<br>Subjects<br>Screened | ES7 | Listing of Reasons for Screen Failure | Not repeated | Weeks 24, 48,<br>96, 144 |
| 2. | ITT-E | ES2 | Listing of Reasons for Study Withdrawal | Include period (Early switch phase/Late switch phase) in the output Include "Day Since Switch" in Study day column and provide for TBR arm | All |
| 3. | ITT-E | SD3 | Listing of Reasons for Study Treatment Discontinuation | Include "Day Since Switch" in Study day column and provide for TBR arm | All |
| 4. | ITT | TA1 | Listing of Planned Randomised and Actual Strata and Treatment Assignments | Not repeated | Weeks 24, 48,<br>96 |
| 5. | ITT | POP_L1 | Listing of Subjects Randomised but not Treated | Not repeated | Weeks 24, 48,<br>96 |

| ICH: L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Protoc | col Deviations | 3 | | | |
| 6. | ITT-E | DV2 | Listing of Important Protocol Deviations | Include period (Early switch phase/Late switch phase) in the output Include "Day Since Switch" in Study day column and provide for TBR arm | All |
| 7. | ITT-E | IE4 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | Not repeated | Weeks 24, 48,<br>96 |
| Popul | ations Analys | ed | | | |
| 8. | ITT-E | SP3a | Listing of Protocol Deviations Leading to Exclusion from the Per Protocol Population | No longer required | Weeks 24, 48,<br>96, 144 |
| Demo | graphic and B | aseline Charac | teristics | | |
| 9. | ITT-E | DM4 | Listing of Demographic Characteristics | Not repeated | Weeks 24, 48,<br>96, 144 |
| 10. | ITT-E | DM10 | Listing of Race | Not repeated | Weeks 24, 48,<br>96, 144 |
| Effica | су | | | | |
| 11. | ITTE | EFF_L1 | Listing of Study Outcome (>= / < 50 c/mL) at Week X – Snapshot Analysis | Please add COVID-19<br>Relatedness column (Yes or blank) | All |
| 12. | ITTE | EFF_L2 | Listing of Quantitative and Qualitative Plasma HIV-1 RNA Data | Include study phase (Early switch phase/Late switch phase) in the output | All |

| ICH: L | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Expos | ure and Treat | ment Complian | ce | | |
| 13. | Safety | EX3 | Listing of Exposure Data | Include study phase (Early switch phase/Late switch phase) in the output | All |
| Adver | se Events | | | | |
| 14. | Safety | AE8 | Listing of All Adverse Events | Include study phase (Early switch phase/Late switch phase) in the output Include "Time Since Switch" in 'Time since 1st dose/Time since last dose' column and provide for TBR arm | All |
| 15. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | | All |
| 16. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | | All |
| 17. | Safety | PSRAE1 | Listing of Possible Suicidality-Related Adverse Event Data: Event and Description (Section 1 and Section 2) | Include study phase (Early switch phase/Late switch phase) in the output Include 'Time since switch' in output | All |
| 18. | Safety | PSRAE3 | Listing of Possible Suicidality-Related Adverse Event Data: Possible Cause(s) (Section 3) | Include study phase (Early switch phase/Late switch phase) in the output Include 'Time since switch' in output | All |

| ICH: L | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 19. | Safety | PSRAE4 | Listing of Possible Suicidality-Related Adverse Event Data (Section 4) | Include study phase (Early switch phase/Late switch phase) in the output Include 'Time since switch' in output | All |
| 20. | Safety | PSRAE5 | Listing of Possible Suicidality-Related Adverse Event Data (Section 5 and Section 8) | Include study phase (Early switch phase/Late switch phase) in the output Include 'Time since switch' in output | All |
| Seriou | s and Other S | ignificant Adve | erse Events | | |
| 21. | Safety | AE8 | Listing of Fatal Adverse Events | Include study phase (Early switch phase/Late switch phase) in the output Include 'Time since switch' in output | All |
| 22. | Safety | AE8 | Listing of Non-Fatal Serious Adverse Events | Include study phase (Early switch phase/Late switch phase) in the output Include 'Time since switch' in output | All |
| 23. | Safety | AE14 | Listing of Reasons for Considering as a Serious<br>Adverse Event | Include study phase (Early switch phase/Late switch phase) in the output | All |
| 24. | Safety | AE8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | Include study phase (Early switch phase/Late switch phase) in the output Include 'Time since switch' in output | All |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 25. | | | | No longer required | |
| Hepate | obiliary (Liver | ) | | | |
| 26. | Safety | MH2 | Listing of Medical Conditions for Subjects with Liver Stopping Events | | All |
| 27. | Safety | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events | | All |
| All Lal | ooratory | | | | |
| 28. | Safety | LB5 | Listing of Clinical ChemistryLaboratory Data for Subjects with Any Value of Potential Clinical Importance | | All |
| 29. | Safety | LB14 | Listing of Laboratory Data with Character Results | | All |
| 30. | Safety | LB5 | Listing of Urinalysis Data for Subjects with Any Value of Potential Clinical Importance | | All |
| Vital S | igns | | | | |
| 31. | Safety | VS4 | Listing of Vital Signs | Add waist to height ratio and waist to hip ratio also in the listing | All |

## 13.15.15. Non-ICH Listings

| Non-ICI | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Study P | opulation | | | | |
| 32. | All<br>Subjects<br>Screened | POP_L2 | Listing of Subject Recruitment by Country and Site Number | Not repeated | Weeks 24,<br>48, 96, 144 |
| 33. | All<br>Subjects<br>Screened | ES9 | Listing of Subjects Who Were Rescreened | Not repeated | Weeks 24,<br>48, 96, 144 |
| 34. | ITT(E) | POP_L3 | Listing of Visit Dates | | All |
| 35. | All<br>Subjects<br>Screened | POP_L4 | Listing of Study Populations | | All |
| 36. | ITT(E) | POP_L5 | Listing of Hepatitis Test Results at Entry | Not repeated | Weeks 24,<br>48, 96, 144 |
| 37. | ITT(E) | CDC3 | Listing of CDC Classification of HIV Infection at Baseline | Not repeated | Weeks 24,<br>48, 96 |
| 38. | ITT(E) | RF2 | Listing of HIV Risk Factors | Not repeated | Weeks 24,<br>48, 96 |
| 39. | ITT(E) | POP_L6 | Listing of Screening Cardiovascular Risk Assessment Data | Not repeated | Weeks 24,<br>48, 96 |

| Non-ICI | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 40. | ITT(E) | MH2 | Listing of Current and Past Medical Conditions at Baseline | Not repeated | Weeks 24,<br>48, 96, 144 |
| 41. | ITT(E) | POP_L7 | Listing of Relationship Between Concomitant AT C Level 1, Ingredient and Verbatim Text | | All |
| 42. | ITT(E) | CM2 | Listing of Concomitant Medications | Include 'Day since switch' in the output | All |
| 43. | ITT(E) | CM2 | Listing of Antiretroval Therapy Stopped Prior to Screening | Not repeated | Weeks 24,<br>48, 96, 144 |
| 44. | ITT(E) | CM2 | Listing of Antiretroval Therapy Received at Screening | Not repeated | Weeks 24,<br>48, 96, 144 |
| 45. | ITT(E) | POP_L8 | Listing of Relationship Between Concomitant ATC Level 4, Ingredient and Verbatim Text | | All |
| Efficacy | 1 | | | | |
| 46. | ITT(E) | EFF_L3 | Listing of Plasma HIV-1 RNA data for subjects with Confirmed Virologic Withdrawal | Include study phase (Early switch phase/Late switch phase) in the output Include 'Day since switch' in the output | All |
| 47. | ITT(E) | EFF_L4 | Listing of CD4+ Cell Count Data | Include study phase study<br>phase (Early switch phase/Late<br>switch phase) in the output | All |
| 48. | ITT(E) | EFF_L5 | Listing of CD8+ and CD4+/CD8+ Cell Count Ratio Data | | All |

| Non-ICI | H: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 49. | ITT(E) | HIV4 | Listing of Stage 3 HIV-1 Associated Conditions | Include study phase (Early switch phase/Late switch phase) in the output Include 'Day since switch' in the output | All |
| 50. | ITT(E) | EFF_L6 | Listing of Subjects Treatment-related discontinuation = Failure (TRDF) and Efficacy-related discontinuation = Failure (ERDF) | No longer required | Week 24, 48,<br>96, 144 |
| 51. | | | | No longer required | |
| Safety | | | | | |
| 52. | Safety | EG3 | Listing of ECG Findings | | All |
| 53. | Safety | SAFE_L1 | Listing of Post Baseline Maximum AL, Maximum AST and Maximum Bilirubin | | All |
| 54. | Safety | SAFE_L2 | Listing of Subjects Meeting Hepatobiliary Abnormality Criteria - Post-Baseline Emergent | | All |
| 55. | Safety | SAFE_L3 | Listing of C-SSRS Suicidal Ideation and Behaviour Data Alerts (4-9) | Include 'Day since switch' in output | All |
| 56. | Safety | SAFE_L4 | Listing of C-SSRS Suicidal Ideation and Behaviour Data | Include 'Day since switch' in output | All |
| 57. | Safety | SAFE_L5 | Listing of C-SSRS False Positive Alerts with Corresponding Reasons | Include 'Day since switch' in output | All |
| 58. | Safety | SAFE_L5 | Listing of all C-SSRS True Positives, with Corresponding Reasons and AE or SAE status | Include 'Day since switch' in output | All |

| Non-ICH | l: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 59. | Safety | SAFE_L6 | Listing of Subjects Who Became Pregnant During the Study | Include study phase (Early switch phase/Late switch phase) in the output | All |
| 60. | Safety | SAFE_L7 | Patient Profiles for Subjects Meeting Protocol Defined Liver Stopping Criteria | | All |
| 61. | Safety | SAFE_L7 | Patient Profiles for Subjects Meeting Confirmed Virologic Withdrawal Criteria | | All |
| 62. | Safety | SAFE_L8 | Listing of Cardiovascular Events | | All |
| Intensiv | e PK - PK Con | centration Dat | a | | |
| 63. | | | | No longer required | |
| 64. | | | | No longer required | |
| Intensiv | e PK Derived I | Parameters | | | |
| 65. | | | | No longer required | |
| 66. | | | | No longer required | |
| Sparse F | PK - PK Conce | entration Data | | | |
| 67. | | | | No longer required | |
| 68. | | | | No longer required | |
| Virology | <i></i> | | | | |
| 69. | Viral<br>Genotypic | VIR_L1 | Listing of All Genotypic Data | | All |
| 70. | | | | No longer required | |

| Non-ICH | l: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 71. | CW | VIR_L2 | Listing of Genotype by Genotypic Cut-Off – CVWs | Add 'Baseline S-GSS Score' before 'S-GSS Score' | All |
| 72. | | | | No longer required | |
| 73. | Viral<br>Phenotypic | VIR_L3 | Listing of All Phenotypic Data | | All |
| 74. | | | | No longer required | |
| 75. | | | | No longer required | |
| 76. | | | | No longer required | |
| 77. | | | | No longer required | |
| 78. | | | | No longer required | |
| 79. | | | | No longer required | |
| 80. | | | | No longer required | |
| 81. | CWW | VIR_L7 | Listing of Genotypic and Phenotypic Data for Subjects with Confirmed Virologic Withdrawal Criteria | | All |
| 82. | | | | No longer required | |
| Health C | Outcomes | | | • | |
| 83. | ITT(E) | HO_L1 | Listing of EQ-5D Category, Utility and Thermometer Scores | Not required | Weeks 24,<br>48, 96 |
| Other | | | | | |
| 84. | Safety | SAFE_L9 | Listing of Renal Biomarker Data | Not required | Weeks 24,<br>48, 96 |

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 85. | Safety | SAFE_L9 | Listing of Bone Biomarker Data | Not required | Weeks 24,<br>48, 96 |
| 86. | | | | | |
| 87. | Safety | SAFE_L9 | Listing of HOMA-Insulin Resistance Data | | All |
| 88. | ITT-E | VIR_L7 | Listing of Genotypic and Phenotypic Data for subjects Last on study VL>400 c/ml with resistance testing | For non-CWW and on-treatment patients | All |
| 89. | ITT(E) | EFF_L3 | Listing of Plasma HIV-1 RNA data for subjects with Potential Precautionary Virologic Withdrawal | Include study phase (Early switch phase/Late switch phase) in the output | All |
| 90. | Safety | LB5 | Listing of Hematology Laboratory Data for Subjects with Any Value of Potential Clinical Importance | | All |
| Study Po | opulation and | Safety | | • | |
| 91. | ITT(E) | POP_L9 | Listing of History of Cardiac Therapeutic Procedures | Not required | Weeks 24,<br>48, 96 |
| 92. | ITT(E) | POP_L10 | Listing of Investigational Product Accountability | | All |
| 93. | | | | No longer required | |
| 94. | Safety | | Listing of Inflammatory Biomarker Data | | 48,96,144,<br>196 |
| 95. | ITT(E) | POP_L11 | Listing of On-Treatment Antiretroviral Therapy Starting after Day 1 | Include "Day Since Switch" in<br>Study day column and provide for<br>TBR arm | 48,96,144,<br>196 |
| 96. | ITT(E) | POP_L11 | Listing of Antiretroviral Therapy Starting after Treatment Discontinuation | Include "Day Since Switch" in Study day column and provide for TBR arm | 48,96,144,<br>196 |

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 97. | ITT(E) | | Listing of non-Important COVID-19 Protocol Deviations | Not required | 96 |
| 98. | Safety | | Listing of All COVID-19 Adverse Events | Mock shell - Refer Listing 98 in RE internal 04 | 96, 144, 196 |
| 99. | Safety | PAN12 | Listing of COVID-19 Assessments and Symptom Assessments for Subjects with COVID-19 Adverse Events | | 96, 144, 196 |
| 100. | Safety | | Listing of Local Laboratory Data | Mock shell - Refer Listing 100 in RE internal 04 | 96, 144, 196 |
| 101. | ITT(E) | PAN7 | Listing of All Subjects with Visits and Assessments Impacted by the Pandemic | | 144, 196 |

### 13.16. Appendix 16: Example Mock Shells for Data Displays

No mock shells were produced.